

#### CLINICAL PROTOCOL

# CONTINUING ACCESS TO THE TYROSINE KINASE INHIBITOR OF VEGFR-2, AG-013736 (A406) FOR PATIENTS PREVIOUSLY RECEIVING AG-013736 IN CLINICAL TRIALS

Compound: Axitinib (AG-013736)

Compound Name: Inlyta®

US IND Number: 63,662

European Clinical Trial Database (EudraCT) 2005-000051-15

Number:

Protocol Number: A4061008

Phase: N/A

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not to disclose it to others (except where required by applicable law) or to use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer should be promptly notified.

# **Document History**

| Document | Version Date | Summary of Changes |
|---|---|---|
| Amendment 7 | 08 November 2018 | <ol> <li>Main changes include:* <ol></ol></li></ol> |
| Amendment 6 | 05 December 2012 | <ul> <li>Main changes include:</li> <li>Update of safety information to align with most recent version of Investigator Brochure (IB).</li> <li>Update AE and safety wording, including pregnancy and Hy's law, to align with current Pfizer SOP (Standard Operating Procedures).</li> <li>Review and simplification of wording and procedures where possible.</li> </ul> |
| Amendment 5 | 15 December 2008 | • See Amendment 5, Appendix D for details. |
| Amendment 4 | 06 February 2008 | See Amendment 5, Appendix C for details. |
| Amendment 3 | 17 October 2006 | See Amendment 5, Appendix B for details. |
| Amendment 2 | 04 November 2004 | • See Amendment 5, Appendix A for details. |

| Document | Version Date | Summary of Changes |
|----------------------|-------------------|-------------------------------|
| Amendment 1 | 19 December 2002 | See Amendment 1, for details. |
| Original<br>Protocol | 23 September 2002 | N/A |

This amendment incorporates all revisions to date, including amendments made at the request of country Health Authorities, IRB/ERB, ECs etc.

#### **SUMMARY**

#### **Indication:**

Patients who have been treated in previous Pfizer sponsored oncology studies, with axitinib either as monotherapy or in combination with another anticancer drug.

#### Rationale:

Some patients in axitinib clinical trials may be experiencing clinical benefit from axitinib treatment either as monotherapy or in combination with another anticancer drug and may wish to continue treatment following completion of the trial. Such patients, after a written re consent, may continue to receive axitinib and the combination study drug (if applicable) at the same dose and schedule as specified in their prior axitinib protocol with the consensus of the principal investigator and the approval of the sponsor company until patients no longer experience clinical benefit, develop unacceptable toxicity or withdraw consent. Complete information for the study drug(s) may be found in the Single Reference Safety Documents, which for this study are the current Investigator Brochures (IBs).

# **Objectives:**

The objective of the trial is to provide continued access to axitinib tablets and study drug(s) given in combination (if applicable) to patients who have completed their participation in a prior axitinib monotherapy or combination study and who have documented stable or responding disease at the time they discontinued in the trial. Continuing access will be provided to patients who have Progressive Disease (PD) but continue to experience clinical benefit from previous study treatment; in this case, clinical benefit is defined as the Sum of Longest Diameters (SLD) of measurable lesions remaining less than or equal to the baseline SLD in the previous axitinib trial (either monotherapy or combination). These patients must not be eligible for treatment with other available approved therapy for the disease under study.

# **Trial Design:**

Axitinib trials (either monotherapy or combination) have been designed with a maximum number of treatment cycles or length of treatment time. However, some patients may be deriving clinical benefit from the drug(s) and want to continue treatment with the investigational agent(s) but are unable to continue in their present trial.

This protocol will provide continued access to axitinib tablets and the combination study drug(s) if applicable for patients who were assigned to an axitinib-containing treatment arm in an axitinib clinical trial. For patients in combination treatment, if axitinib is interrupted due to toxicity, the continuation of the combination drug will be evaluated on a case by case analysis after discussion with the Sponsor (based on the benefit risk assessment and other available options).

To be eligible for this protocol, patients must have been receiving axitinib tablets (either monotherapy or combination) at the time their previous trial ended and have had Stable Disease (SD) or responding disease (PR or CR) according to the disease response criteria in the previous axitinib trial. Patients who have Progressive Disease (PD) but continue to experience clinical benefit in previous axitinib study will be eligible for enrollment; in this case, clinical benefit is defined as the Sum of Longest Diameters (SLD) of measurable lesions remaining less than or equal to the baseline SLD in the previous axitinib trial. These patients must not be eligible for treatment with other available approved therapy for the disease under study. These patients will be allowed to continue receiving study treatment(s) until the SLD of measurable lesions becomes greater than the baseline SLD in the previous trial.

During treatment on this protocol, all patients will be evaluated for safety per local standard clinical practice. Axitinib dosing or combination therapy (if applicable) and concomitant treatments will be monitored. Follow up information on alive/death status will be collected every 2 months starting from last study visit. Efficacy parameters will not be evaluated as part of this protocol. Pending drug availability, patients may continue to receive axitinib tablets or the combination drug(s) (if applicable) until the axitinib development program is terminated or when they are no longer receiving benefit (defined as no longer having stable or responding disease according to institutional standards), or clinical benefit for eligible patients with PD as previously defined.

# **Endpoints:**

All patients will be assessed for safety by monitoring adverse events and laboratory values per local standard clinical practice. Response to therapy will not be collected as part of this protocol.

#### **Trial Treatments – Axitinib:**

Axitinib will be supplied as 1-mg and 5-mg film-coated tablets for oral administration.

#### **Trial Treatments – Combination Drug (if applicable):**

The study drug(s) given in combination with axitinib will be supplied according to the indications reported in the parent study protocol included in the Appendix 1.

#### **Statistical Methods:**

Safety data will be summarized for all treated patients using appropriate tabulations and descriptive statistics (see Section 9.2).

# **SCHEDULE OF ACTIVITIES:**

| Assessments | Schedule |
|---|---|
| Written Informed Consent. | Before receiving axitinib tablets (either monotherapy or combination) in this protocol. |
| Safety Assessments (eg, physical exams, | According to local clinical practice. |
| blood pressure assessments, hematology, clinical chemistry, urinalysis). | If not performed within the last 8 weeks as part of previous axitinib study serum or plasma thyroid function tests (Free T4 and TSH) should be performed at screening/baseline and repeated subsequently as clinically indicated, and according to local clinical practice (but not less than every 12 weeks (±2 weeks). |
| | Pregnancy test and contraceptive check are to be performed at screening/baseline if clinically indicated, and repeated if indicated or required by EC/IRB or by local law. |
| | The following assessments should be added only for patients previously enrolled in the parent protocol A4061068: |
| | • Liver function test (Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST), Alkaline phosphatase, Bilirubin): to be performed every 4 weeks; |
| | ECG: to be performed at the time of<br>End of Treatment, and as clinically<br>indicated; |
| | Ophthalmologic examination: at the first occurrence of any vision changes and as clinically indicated. |
| Adverse Events. | According to local clinical practice. <sup>a</sup> |
| Concomitant Treatments. | According to local clinical practice. |
| Axitinib (as monotherapy) Dosing. | As per the patient's previous protocol. |

| Assessments | Schedule |
|---|---|
| Axitinib and the other anticancer drug (as combination therapy) Dosing. | As per the patient's previous protocol. |
| 28-day Safety Follow Up. | <sup>a</sup> Patients should be followed for safety including thyroid testing at least 28 days after last dose and according to standard clinical practice. |
| Follow up information on survival. | After follow up visit attempts should be made, where possible, to collect information every 2 months on alive/death status via phone call or routine visit. |

a. Adverse events should be collected throughout the trial, starting at the time written consent is given through to at least 28 days after the last dose of axitinib or combination drug(s) (if applicable). Adverse events that are serious, suspected to be related to axitinib or study drug(s) given in combination (if applicable) or considered significant by the investigator or Pfizer medical monitor must be followed after therapy discontinuation until the event or its sequelae resolve or stabilize at a level acceptable to the investigator and the Pfizer medical monitor or his/her designated representative. Following the active safety reporting period, other SAEs of which the investigator becomes aware should be reported to Pfizer, unless the SAE is attributed by the investigator to complications of either the underlying malignancy or any subsequent anti-cancer therapy or to the patient's participation in a subsequent clinical study. Refer to Section 8 for more details.

# **TABLE OF CONTENTS**

| LIST OF TABLES | 10 |
|---|---|
| APPENDICES | 11 |
| 1. INTRODUCTION | 12 |
| 1.1. Indication | 12 |
| 1.2. Background | 12 |
| 1.2.1. Molecular Formula and Molecular Activity | 12 |
| 1.2.2. Scope of Axitinib Clinical Program | 13 |
| 1.2.2.1. Overall Clinical Safety of Axitinib | 13 |
| 1.2.2.2. Overall Clinical Safety of Combination Drug (if applicable) | 14 |
| 1.3. Rationale | 14 |
| 2. TRIAL OBJECTIVES | 14 |
| 3. TRIAL DESIGN | 14 |
| 4. PATIENT SELECTION | 15 |
| 4.1. Inclusion Criteria | 15 |
| 4.2. Exclusion Criteria | 16 |
| 4.3. Life Style Guidelines. | 16 |
| 4.4. Sponsor Qualified Medical Personnel | 17 |
| 5. TRIAL TREATMENTS | 17 |
| 5.1. Allocation to Treatment (Axitinib and Combination Drug, if applicable) | 17 |
| 5.2. Drug Supplies (Axitinib and Combination Drug, if applicable) | 18 |
| 5.2.1. Preparation and Dispensing (Axitinib and Combination Drug, if applicable) | 18 |
| 5.2.2. Formulation and Packaging | 18 |
| 5.2.2.1. Formulation and Packaging (Axitinib Monotherapy) | 18 |
| 5.2.2.2. Formulation and Packaging (Combination Therapy, if applicable) | 18 |
| 5.2.3. Administration | 18 |
| 5.2.3.1. Administration (Axitinib Monotherapy) | 18 |
| 5.2.3.2. Administration (Combination Therapy, if applicable) | 19 |
| 5.2.4. Dose Interruption and Reductions | 19 |
| 5.2.4.1. Dose interruption and reductions (Axitinib Monotherapy) | 19 |

| 5.2.4.2. Dose Interruption and Reductions (Combination Therapy, if applicable) | |
|---|---|
| 5.3. Drug Storage and Drug Accountability (Axitinib and Combination Drug, if applicable) | 22 |
| 5.4. Concomitant Medication(s) | 23 |
| 5.4.1. Concomitant Medication(s) (Axitinib Monotherapy) | 23 |
| 5.4.2. Concomitant Medication(s) (Combination Therapy, if applicable) | 25 |
| 5.5. Rescue Therapy | 25 |
| 6. TRIAL PROCEDURES | 25 |
| 6.1. Patient Enrollment | 25 |
| 6.2. Trial Procedures | 25 |
| 6.3. Follow-up Visit | 26 |
| 6.4. Patient Withdrawal | 26 |
| 7. SAFETY ASSESSMENTS | 27 |
| 8. ADVERSE EVENT REPORTING | 27 |
| 8.1. Adverse Events | 27 |
| 8.2. Reporting Period | 28 |
| 8.3. Definition of an Adverse Event | 28 |
| 8.4. Medication Errors | 29 |
| 8.5. Abnormal Test Findings | 30 |
| 8.6. Serious Adverse Events | 30 |
| 8.6.1. Protocol-Specified Serious Adverse Events | 31 |
| 8.6.2. Potential Cases of Drug-Induced Liver Injury | 31 |
| 8.7. Hospitalization | 32 |
| 8.8. Severity Assessment | 33 |
| 8.9. Causality Assessment | 34 |
| 8.10. Exposure During Pregnancy | 34 |
| 8.11. Occupational Exposure | 35 |
| 8.12. Withdrawal Due to Adverse Events (See also Patient Withdrawal, Section 6.4) | 36 |
| 8.13. Eliciting Adverse Event Information | |
| 8.14. Reporting Requirements | |
| 8.14.1. Serious Adverse Event Reporting Requirements | |

| | 8.14.2. Non-Serious Adverse Event Reporting Requirements | 37 |
|---|---|---|
| | 8.14.3. Sponsor Reporting Requirements to Regulatory Authorities | 37 |
| 9. DATA | ANALYSIS/STATISTICAL METHODS | 37 |
| 9.1. | Sample Size Determination | 37 |
| 9.2. | Safety Analysis | 37 |
| 9.3. | Efficacy Analysis | 37 |
| 9.4. | Data Monitoring Committee | 37 |
| 10. QUAI | LITY CONTROL AND QUALITY ASSURANCE | 38 |
| 11. <b>DAT</b> / | A HANDLING AND RECORD KEEPING | 38 |
| 11.1 | 1. Case Report Forms/Electronic Data Record | 38 |
| 11.2 | 2. Record Retention | 39 |
| 12. ETHI | CS | 39 |
| 12.1 | I. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 39 |
| 12.2 | 2. Ethical Conduct of the Trial | 39 |
| 12.3 | 3. Patient Information and Consent | 40 |
| | 4. Reporting Of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 40 |
| 13. DEFI | NITION OF END OF TRIAL | 40 |
| 13.1 | 1. End of Trial in all Participating Countries | 40 |
| 14. SPON | ISOR DISCONTINUATION CRITERIA | 41 |
| 15. PUBL | ICATION OF TRIAL RESULTS | 41 |
| 15.1 | 1. Communication of Results by Pfizer | 41 |
| 15.2 | 2. Publications by Investigators | 42 |
| 16. APPE | NDICES | 44 |
| | LIST OF TABLES | |
| Table 1. | Available Axitinib as Monotherapy Dose Levels | 10 |
| | | 10 |
| Table 2. | Criteria for Dose Modification for Axitinib Monotherapy Related Adverse Events other than Hypertension, Hemoptysis or Proteinuria | 19 |
| Table 3. | Hypertension Management Plan for Axitinib Monotherapy | |

# **APPENDICES**

| Appendix 1. Study Protocol A4061068 | 44 |
|-------------------------------------|----|
|-------------------------------------|----|

#### 1. INTRODUCTION

#### 1.1. Indication

Patients who have been treated in previous Pfizer sponsored oncology studies, with axitinib either as monotherapy or in combination with another anticancer drug.

# 1.2. Background

Axitinib is a substituted indazole derivative that has a direct antiangiogenic effect mediated by the potent inhibition of vascular endothelial growth factor receptor 2 (VEGF-2; KDR) kinase activity. Axitinib is also a potent inhibitor of VEGFR-1 (flt-1) and VEGFR-3. Axitinib is currently being investigated as an anticancer agent in a series of clinical trials. Axitinib studies have been designed with a maximum number of cycles or time that a patient can be on the trial. Some patients may be deriving benefit from the drug and want to have continued access to this investigational agent. This protocol will provide continued access to axitinib tablets to patients who were assigned to an axitinib-containing treatment arm in an axitinib clinical trial.

The background relevant to the study drug(s) given in combination with axitinib, if applicable, is described in the parent protocol(s) attached in the Appendix 1.

# 1.2.1. Molecular Formula and Molecular Activity

Axitinib is a substituted indazole derivative that was discovered using structure-based drug design. The molecular formula is  $C_{22}H_{18}N_4OS$  with molecular weight of 386.47. The chemical name is

N-Methyl-2-[3-((E)-2-pyridin-2-yl-vinyl)-1H-indazol-6-ylsulfanyl]-benzamide:

The mechanism of action of axitinib is a direct anti-angiogenic effect mediated by the potent inhibition of vascular endothelial growth factor receptor 2 (VEGFR-2; KDR) kinase activity. Axitinib is also a potent inhibitor of VEGFR-1 (flt-1) and VEGFR-3.

# 1.2.2. Scope of Axitinib Clinical Program

Clinical trials with axitinib in cancer patients were initiated in April 2002. The ongoing clinical program is designed to test the safety and efficacy of axitinib, either as a single-agent or in combination with other anti-tumor agents, in a variety of advanced solid tumors.

Tumor types under study include, but are not limited to, advanced RCC, advanced NSCLC, HCC, advanced gastric cancer, and other solid tumors. Refer to the most recent version of IB for complete list of closed and ongoing studies, and the most updated information on the clinical program.

# 1.2.2.1. Overall Clinical Safety of Axitinib

As of 01 June 2012, a total of 4372 patients were enrolled into clinical studies in the axitinib clinical program and included in the safety (serious adverse event) database. Of these, 3075 patients received axitinib. In total, 2543 patients with cancer received either single-agent axitinib or axitinib in combination with chemotherapy. In addition, 516 healthy volunteers and 16 patients with hepatic impairment received single agent axitinib.

A complete overview of safety and additional information on axitinib can be found in the most current version of the Investigator's Brochure (IB).

Overall, the adverse events reported in axitinib clinical studies are considered manageable and were generally reversible and expected for this class of agents. For single-agent axitinib, the most common adverse events reported from 699 cancer patients regardless of causality included diarrhea (397 patients, 56.8%), fatigue (368 patients, 52.6%), hypertension (318 patients, 45.5%), decrease appetite (286 patients, 40.9%), nausea (264 patients, 37.8%), dysphonia (242 patients, 34.6%), palmar-plantar erythrodysaesthesia syndrome (202 patients, 28.9%), weight decreased (197 patients, 28.2%), vomiting (166 patients, 23.7%), constipation (165 patients, 23.6%), headache (151 patients, 21.6%), cough (149 patients, 21.3%), arthralgia and dyspnea (140 patients, 20%). Additionally, hypothyroidism and proteinuria were reported as adverse events in 122 patients (17.5%) and 117 patients (16.7 %), respectively. Grade 3+ events occurred most frequently for hypertension (134 patients, 19.2%), fatigue (90 patients, 12.9%), and diarrhea (65 patients, 9.3%).

In patients with solid tumors who received single-agent axitinib from completed studies, the majority of the hematological test abnormalities were Grade 1 and 2, however 53 patients (7.9%) reported Grade 3 lymphocytopenia, and the following Grade 3 or 4 events were reported: 9 patients (1.3%) hemoglobin decreased, 9 patients (1.3%) neutrophils decreased, 3 patients (0.4%) white blood cells decreased, 2 patients (0.3%) platelets decreased. As per clinical chemistry, Grade 3 or 4 lipase abnormalities were reported in 26 patients (7%), hyponatremia in 34 patients (5%), hyperglycemia in 23 patients (3.3%), hyperkalemia in 22 patients (3.2%), elevations in serum glutamic oxaloacetic transaminase (SGOT), aspartate aminotransferase (AST) and alkaline phosphatase in 13 patients (1.9%), total bilirubin increase in 5 patients (0.7%), and creatinine increased in 4 patients (0.6%). For urinalysis, Grade 3 proteinuria was reported in 24 patients (3.4%).

In Phase 3 study A4061032, hypothyroidism was reported in 69/359 patients (19%) receiving axitinib. Hyperthyroidism was reported in 4/359 patients (1%). In patients who had thyroid stimulating hormone (TSH) <5  $\mu$ U/mL before treatment, elevations of TSH to  $\geq$ 10  $\mu$ U/mL occurred in 79/245 patients (32%) receiving axitinib. Monitoring thyroid function before initiation of, and periodically throughout, treatment with axitinib is recommended. Hypothyroidism and hyperthyroidism should be treated according to standard medical practice to maintain euthyroid state.

# 1.2.2.2. Overall Clinical Safety of Combination Drug (if applicable)

An overview of safety and information on study drug(s) given in combination with the Axitinib is available in the parent protocol(s) in the Appendix 1.

Additional information for the study drug(s) may be found in the Single Reference Safety Document, which for this study are the current Investigator Brochure (IBs).

#### 1.3. Rationale

Some patients in axitinib clinical trials may be experiencing clinical benefit from axitinib either as monotherapy or in combination with another anticancer drug and may wish to continue treatment following completion of the trial. Such patients, after a written re-consent, may continue to receive axitinib and the combination study drug (if applicable) at the same dose and schedule as specified in their prior axitinib protocol, with the consensus of the principal investigator and the approval of the sponsor company until patients no longer experience clinical benefit, develop unacceptable toxicity or withdraw consent.

Complete information for the study drug(s) may be found in the Single Reference Safety Documents, which for this study are the current Investigator Brochures.

#### 2. TRIAL OBJECTIVES

The objective of the trial is to provide continued access to axitinib tablets and to the study drug(s) given in combination (if applicable) to patients who have completed their participation in a prioraxitinib monotherapy or combination study and who have documented stable disease, responding disease or clinical benefit as described below at the time they discontinued from the previous trial.

#### 3. TRIAL DESIGN

Axitinib trials (either monotherapy or combination) have been designed with a maximum number of treatment cycles. However, some patients may be deriving clinical benefit from the drug(s) and want to continue treatment with the investigational agent(s) but are unable to continue in their present trial.

This protocol will provide continued access to axitinib tablets and the combination study drug(s) if applicable for patients who were assigned to an axitinib-containing treatment arm in an axitinib clinical trial. For patients in combination treatment, if axitinib is interrupted due to toxicity, the continuation of the combination drug will be evaluated on a case by case analysis after discussion with the Sponsor (based on the benefit risk assessment and other available options).

To be eligible for this trial, patients must have been receiving axitinib tablets (as either monotherapy or combination as applicable) at the time their previous trial ended and have had Stable Disease (SD) or responding disease (PR or CR) according to the disease response criteria in the previous axitinib trial. Patients who have Progressive Disease (PD) but continue to experience clinical benefit in previous axitinib study will be eligible for enrollment; in this case, clinical benefit is defined as the Sum of Longest Diameters (SLD) of measurable lesions remaining less than or equal to the baseline SLD in the previous axitinib trial. These patients must not be eligible for treatment with other available approved therapy for the disease under study. These patients will be allowed to continue receiving study treatment(s) until the SLD of measurable lesions becomes greater than the baseline SLD in the previous trial.

During treatment on this protocol, all patients will be evaluated for safety and monitored per local standard clinical practice. Axitinib dosing or combination therapy, if applicable) and concomitant treatments will be monitored. Follow up information on alive/death status will be collected every two months starting from last study visit. Efficacy parameters will not be evaluated as part of this protocol. Pending drug availability, patients may continue to receive axitinib tablets or combination therapy (if applicable) until the axitinib development program is terminated or when they are no longer receiving benefit (defined as no longer having stable or responding disease according to institutional standards), or clinical benefit for eligible patients with PD as previously defined.

#### 4. PATIENT SELECTION

This clinical trial can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular patient.

#### 4.1. Inclusion Criteria

Patient eligibility should be reviewed and documented by an appropriately qualified member of the investigator's study team before patients are included in the study.

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

- Patients who were assigned to an axitinib-containing treatment arm in a previous clinical trial.
- Patients who were receiving axitinib tablets at the time their previous trial ended.
- Patients who have stable (SD) or responding disease (PR or CR) documented by the appropriate radiological, clinical, or laboratory assessments within 12 weeks before enrollment (Note: response criteria from the previous axitinib protocol should be used to determine stable or responding disease).

- Patients who have Progressive Disease (PD) but have experienced clinical benefit from previous axitinib treatment will be eligible for enrollment; in this case, clinical benefit is defined as the Sum of Longest Diameters (SLD) of measurable lesions remaining less than or equal to the baseline SLD in the previous axitinib trial. These patients must not be eligible for treatment with other available approved therapy for the disease under study. The Pfizer clinician must approve the enrollment prior to treatment start.
- Patients who are informed of, and willing and able to comply with the investigational nature of the trial, and have signed a written informed consent in accordance with institutional and ICH GCP guidelines.

#### 4.2. Exclusion Criteria

Patients presenting with any of the following will not be included in the trial:

• Patients may not participate in this trial if the conditions for continuing treatment in the previous axitinib protocol are not met.

#### 4.3. Life Style Guidelines

All male and female patients who, in the opinion of the investigator, are biologically capable of having children and are sexually active, must agree to use a highly effective method of contraception consistently and correctly for the duration of the active treatment period and for 90 days after the last dose of investigational product. The investigator, in consultation with the patient, will select the most appropriate method of contraception for the individual patient from the permitted list of contraception methods, and instruct the patient in its consistent and correct use. The investigator, at each study visit, will confirm and document consistent and correct use. In addition, the investigator will instruct the patient to call immediately if the selected birth control method is discontinued or if pregnancy is known or suspected.

Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (ie, perfect use) and include:

- 1. Established use of oral, injected or implanted hormonal methods of contraception.
- 2. Correctly placed intrauterine device (IUD) or intrauterine system (IUS).
- 3. Male condom or female condom used WITH a spermicide (ie, foam, gel, film, cream, suppository).
- 4. Male sterilization with appropriately confirmed absence of sperm in the post-vasectomy ejaculate.

5. Bilateral tubal ligation or bilateral salpingectomy.

Only for patients previously enrolled in the parent protocol A4061068 and under treatment with axitinib and crizotinib the following additional guideline is to be followed:

# **Sunlight Exposure**

Patients will be advised to report any reaction to sun exposed skin. In addition, special precaution will be taken to limit any potential photo irritation effect, by minimizing the patients' exposure to light including high intensity ultraviolet B light (UVB) sources such as tanning beds, tanning booths and sunlumps. Patients should be encouraged to apply sunscreen/sunblock daily.

# 4.4. Sponsor Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the "Study Team on Demand" (SToD).

To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, participants are provided with a contact card. The contact card contains, at a minimum, protocol and investigational product identifiers, participant numbers, contact information for the investigator site, and contact details for a contact center in the event that the investigator site staff cannot be reached to provide advice on a medical question or problem originating from another healthcare professional not involved in the participant's participation in the study. The contact number can also be used by investigator staff if they are seeking advice on medical questions or problems; however, it should be used only in the event that the established communication pathways between the investigator site and the study team are not available. It is therefore intended to augment, but not replace, the established communication pathways between the investigator site and the study team for advice on medical questions or problems that may arise during the study. The contact number is not intended for use by the participant directly, and if a participant calls that number, he or she will be directed back to the investigator site.

#### 5. TRIAL TREATMENTS

# 5.1. Allocation to Treatment (Axitinib and Combination Drug, if applicable)

This trial is open label. All patients will receive axitinib either as monotherapy or in combination with other study drug(s) according to the indications reported in the parent protocol (Appendix 1). The dose and the schedule of axitinib and of the study drug(s) given in combination (if applicable) will be the same as they were taking in the previous trial.

# 5.2. Drug Supplies (Axitinib and Combination Drug, if applicable)

The Global Supply Chain, Pfizer Global Research and Development will supply axitinib and the combination drug(s) (if applicable) for the trial. Clinical Trial Material (CTM) will be shipped to the study sites with an Investigational Drug Receipt Confirmation form. This form should be completed and returned as directed on the form.

#### 5.2.1. Preparation and Dispensing (Axitinib and Combination Drug, if applicable)

The investigator, or an approved representative (eg, pharmacist), will ensure that all study drug is stored in a secured area, under recommended storage conditions and in accordance with applicable regulatory requirements.

# 5.2.2. Formulation and Packaging

# 5.2.2.1. Formulation and Packaging (Axitinib Monotherapy)

Axitinib will be supplied as 1-mg and 5-mg film coated tablets for oral administration in HDPE (High density polyethylene) bottles with desiccant.

# 5.2.2.2. Formulation and Packaging (Combination Therapy, if applicable)

The combination therapy will be supplied according to the indications reported in the parent protocol (Appendix 1).

#### 5.2.3. Administration

# **5.2.3.1.** Administration (Axitinib Monotherapy)

Axitinib will be administered orally. Tablets should be taken with food, at approximately the same time each day. Patients should be instructed that if they vomit any time after taking a dose, that they must not "make it up" with an extra dose, but instead resume subsequent doses as prescribed. Missed doses may be taken late, up to 3 hours before the next scheduled dose, otherwise should be skipped. Patient must be instructed to record all doses (and missed or vomited doses) in a dosing diary supplied by the site. If doses are missed or vomited, this must be indicated in the source documents and CRFs.

Patients experiencing drug reaction greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 should undergo dose modification as recommended in Section 5.2.4.

| Table 1. | . Avai | lable A | xitinib | as Mo | onotherapy | Dose 1 | Levels |
|----------|--------|---------|---------|-------|------------|--------|--------|

| Dose | Dispensed As |
|-----------|--------------------------------------|
| 10 mg BID | 2 X 5 mg Tablets BID |
| 7 mg BID | 1 X 5 mg Tablet +2 X 1mg Tablets BID |
| 5 mg BID* | 1 X 5 mg Tablet BID |
| 3 mg BID | 3 X 1 mg Tablets BID |
| 2 mg BID | 2 X 1 mg Tablets BID |

<sup>\*</sup> Dosing regimen other than twice a day dosing (BID) is allowed ONLY with discussion and concurrence of Sponsor.

Once a patient has a dose reduction for study drug related toxicity, the dose normally will not be re-escalated. However, patients who tolerate the lower dose without toxicities above Grade 1 for at least 8 weeks may be considered for re-escalation. The investigator and sponsor's medical monitor will discuss the case and decide if re-escalation is appropriate.

#### 5.2.3.2. Administration (Combination Therapy, if applicable)

Patients receiving axitinib in combination with other study drug(s) should be treated according to administration rules showed in the relevant parent protocol (Appendix 1).

# 5.2.4. Dose Interruption and Reductions

# **5.2.4.1.** Dose interruption and reductions (Axitinib Monotherapy)

Adverse events and other symptoms will be graded according to the current Common Terminology for Adverse Events version 4.03 (CTCAE) (See URL: http://ctep.cancer.gov/reporting/ctc.html).

This section contains management of adverse events except hypertension, hemoptysis and proteinuria which are discussed in subsequent sections.

Patients developing a treatment-related CTCAE Grade 1 or 2 adverse event will have their dose continued at the same dose level.

If any patient requires doses lower than 2 mg BID, contact the sponsor for discussion.

The criteria for dose modification for study drug related adverse events are summarized in Table 2 below.

Table 2. Criteria for Dose Modification for Axitinib Monotherapy Related Adverse Events other than Hypertension, Hemoptysis or Proteinuria

| Related Adverse Events | Intervention |
|---|---|
| Grade 1. | Continue at same dose level. |
| Grade 2. | Continue at same dose level. |
| Grade 3 nonhematologic treatment-related | Decrease dose to one lower dose level. |
| toxicity. | |
| Grade 4 nonhematologic treatment-related | Interrupt dosing; re-start at one lower dose |
| toxicity or Grade 4 hematologic toxicity.* | level as soon as improvement to CTCAE |
| | Grade ≤2. If patient requires dose reduction |
| | below 2 mg BID, contact sponsor for |
| | discussion. |

<sup>\*</sup> Patients who develop grade 4 lymphopenia may continue study treatment without interruption.

Guidelines for dose reductions for specific adverse events are provided in the following sections.

# **5.2.4.1.1.** Dose Reduction for Hypertension (Axitinib Monotherapy)

Patients treated with axitinib will be issued blood pressure cuffs (provided by Pfizer) for home monitoring and instructed to measure their blood pressure (BP) twice daily, prior to taking each dose. All blood pressure measurements will be recorded in a diary and brought to the nurse or study coordinator at each clinic visit for review. Patients should be instructed by the study staff to contact their physician immediately for guidance if their systolic blood pressure rises above 150 mm Hg, diastolic blood pressure rises above 100 mm Hg, or if they develop symptoms perceived to be related to elevated BP (eg, headache, visual disturbance). See below for dose modifications for hypertension.

New or additional antihypertensive therapy (See Section 5.4, Concomitant Medication(s) for guidance) should be started if 2 blood pressure readings, taken in the clinic and separated by at least 1 hour, show the following: 2 systolic blood pressure readings greater than 150 or 2 diastolic blood pressure readings greater than 100 mm Hg. Alternately, the dose of existing antihypertensive medication(s) may be increased. Note: the early introduction of antihypertensive agents for Grade 1 and Grade 2 hypertension in order to minimize the occurrence of more severe or persistent hypertension while undergoing treatment with axitinib will not constitute a Grade 3 toxicity.

If the patient is already on maximal antihypertensive treatment, the study drug should be reduced by 1 dose level.

Patients on maximal antihypertensive treatment (to be defined on an individual patient basis according to the judgment of the investigator, but may include up to 4 anti-hypertensive medications given for 2 weeks) who have 2 systolic blood pressure readings, separated by at least 1 hour, greater than 160 mm Hg, or 2 diastolic blood pressure readings, separated by at least 1 hour, greater than 105 mm Hg, will have treatment with axitinib held. (Note: if study drug is held, patients receiving antihypertensive medications should monitor closely for hypotension).

Blood pressure may decrease within 24 hours of stopping therapy. Blood pressure measurements used to decide to discontinue or interrupt axitinib dosing or to adjust antihypertensive medications should be done in the clinic. Plasma half-life of axitinib is 2-4 hours and BP usually decreases within 1-2 days following dose interruption.

Treatment with axitinib should be restarted at 1 lower dose level, rounded down to accommodate dosage form availability, after the systolic blood pressure reduces to less than 150 mm Hg and the diastolic blood pressure reduces to less than 100 mm Hg.

Patients who develop recurrent systolic hypertension (2 BP readings separated by at least 1 hour show systolic pressure >150 mm Hg) or recurrent diastolic BP >100 mm Hg following previous study drug dose reduction should undergo another dose reduction by one dose level. If a patient requires dose reduction below 2 mg BID, contact Sponsor for discussion. Blood pressure measurements used for axitinib-discontinuation decision-making should be done in the clinic.

Guidance on dose interruption and reduction for hypertension is summarized in Table 3 below.

Table 3. Hypertension Management Plan for Axitinib Monotherapy

| Degree of Blood Pressure Elevation | | | Management |
|---|---|---|---|
| Systolic Pressure | | Diastolic Pressure | |
| 2 BP readings separated by at<br>least 1 hour show systolic<br>pressure >150 mm Hg | OR | 2 BP readings separated by at<br>least 1 hour show diastolic<br>pressure >100 mm Hg | If not on maximal antihypertensive treatment, institute new or additional antihypertensive medication and maintain dose of study drug. |
| | | | If on maximal antihypertensive treatment, reduce study drug to one lower dose level. |
| 2 BP readings separated by at<br>least 1 hour show systolic<br>pressure >160 mm Hg | OR | 2 BP readings separated by at<br>least 1 hour show diastolic<br>pressure >105 mm Hg | Interrupt dosing;* adjust<br>antihypertensive medication; as<br>soon as BP is less than<br>150/100 mm Hg, restart study<br>drug at one lower dose level. |
| Recurrent hypertension<br>following previous dose<br>reduction (2 BP readings<br>separated by at least 1 hour<br>show systolic pressure<br>>150 mm Hg) | OR | Recurrent diastolic BP<br>>100 mm Hg (2 BP readings<br>separated by at least 1 hour)<br>following previous dose<br>reduction | Repeat study drug dose reduction<br>by one lower dose level. If a<br>patient requires dose reduction<br>below 2 mg BID, contact Sponsor<br>for discussion |

<sup>\*</sup> If study drug is held, patients receiving antihypertensive medications should monitor closely for hypotension. Plasma half-life of axitinib is 2 – 4 hours and BP usually decreases within 1-2 days following dose interruption.

#### 5.2.4.1.2. Dose Reduction for Hemoptysis (Axitinib Monotherapy)

Bleeding from the lungs as evidenced by hemoptysis will be graded according to the Hemorrhage category of CTCAE.

Treatment with axitinib will be discontinued for hemoptysis of  $>\frac{1}{2}$  tsp of bright red blood per day. In addition, a radiologic assessment (eg, chest x-ray) should be considered for patients who have hemoptysis  $>\frac{1}{2}$  tsp of bright red blood per day. If the hemoptysis resolves to baseline within 1 week and there is no evidence of disease cavitation, treatment with axitinib may continue at the current dose level. Patients who experience hemoptysis without resolution to baseline within 1 week, or with evidence of disease cavitation should discontinue from treatment with axitinib.

# **5.2.4.1.3.** Dose Reduction for Proteinuria (Axitinib Monotherapy)

Monitoring for proteinuria before initiation of and periodically throughout treatment with axitinib is recommended, as per clinical judgment. For patients who develop moderate to severe proteinuria, monitoring, and dose reduction or temporary interruption of axitinib given in monotherapy should be considered.

General guidelines are reported below. Medical judgment, and the patient's clinical conditions, should always be considered to determine the most appropriate monitoring of proteinuria. Safeguard of the patient's safety and a positive risk-benefit assessment should always be evaluated when less restrictive monitoring is adopted.

Perform dipstick proteinuria (or equivalent semi-quantitative test) at regular frequency. At documentation of >2+ or equivalent proteinuria by dipstick, patients should have a 24-hour urine collection for total protein. Axitinib dosing may continue while waiting for test results.

If <2 g proteinuria/24-hour is reported, treatment with axitinib may continue without dose reduction.

If  $\geq 2$  g proteinuria/24-hour is reported, treatment with axitinib should be interrupted. A 24-hour urine collection for total protein and creatinine clearance should be performed weekly until results show  $\leq 2$  g proteinuria/24-hour, at which time treatment with axitinib may be restarted at one lower dose level. Patients, once restarted on axitinib, will have weekly monitoring for proteinuria by semiquantitative testing (eg, dipstick) as long as the proteinuria reading is 2+ or higher, or, alternatively, by quantitative methods as long as proteinuria is  $\geq 1$  g/24-hour. The 24-hour urine collection to monitor the degree of proteinuria should be repeated every 4 weeks until it has decreased to  $\leq 500$  mg/24-hour.

If recurrent ≥2 g proteinuria/24-hour is reported, treatment with axitinib should be interrupted again. 24-hour urine collection for total protein and creatinine clearance should be performed weekly until results show <2 g proteinuria/24-hour, at which time treatment with axitinib may be restarted at one lower dose level. If a patient requires dose reduction below 2 mg BID, contact the Sponsor for discussion.

# 5.2.4.2. Dose Interruption and Reductions (Combination Therapy, if applicable)

The recommended dose modifications of the combination therapy with axitinib and other anticancer study drug(s) are detailed in the relevant parent protocol (Appendix 1).

In case the patient withdraws the drug given in combination with axitinib, and continue on axitinib alone, the dose interruptions and modifications will follow the study A4061008 axitinib monotherapy dose modification rules.

# 5.3. Drug Storage and Drug Accountability (Axitinib and Combination Drug, if applicable)

The investigator or an approved representative (eg, pharmacist) will ensure that all trial drugs are stored in a secure area, under recommended storage conditions and in accordance with applicable regulatory requirements.

Axitinib and the other anticancer drug(s) given in combination should be stored at controlled room temperature (15-30°C), in provided packaging.

Investigators and site staff are reminded to check temperatures daily and ensure that thermometers are working correctly as required for proper storage of investigational products. These include thermometers for both the room storage and refrigerator storage. Any temperature excursions should be reported immediately.

To ensure adequate records, all study drug will be accounted for in the drug accountability inventory forms as instructed by Pfizer. Unless otherwise authorized by Pfizer, at the end of the clinical trial all drug supplies unallocated or unused by the patients must be destroyed by procedures approved by Pfizer or returned to Pfizer or its appointed agent (eg, a contract research organization).

Axitinib is a hazardous drug (due to possible reproductive toxicity), and should be handled according to the recommended procedures described in the current edition of the American Society of Hospital Pharmacists (ASHP), Technical Assistance Bulletin on Handling Cytotoxic and Hazardous Drugs, American Hospital Formulary Service (AHFS) Drug Information (1999) and its references. Procedures described in each institution's pharmacy or hospital standard operating procedure manual should be followed when handling hazardous drugs. Only qualified personnel who are familiar with procedures should undertake the handling, and safe disposal of study drug.

## 5.4. Concomitant Medication(s)

# 5.4.1. Concomitant Medication(s) (Axitinib Monotherapy)

Palliative and supportive care for disease-related symptoms will be offered to all patients on this trial. Low-dose oral steroids (defined as ≤5 mg per day prednisone or equivalent) or topical or inhaled steroids at any dose may be taken during the study. The therapeutic use of colony-stimulating factors is a matter of clinical judgment. Prophylactic use is permitted in patients who have experienced infection or grade 4 neutropenia during the previous cycle. If colony stimulating factors are given, use should be consistent with product labeling and should be documented in the patient's medical record.

In vitro studies with human liver microenzymes and recombinant CYP450 enzymes indicated that axitinib metabolism was primarily mediated by the drug-metabolizing enzyme CYP3A, and to a lesser extent by CYP1A2, CYP2C19 and UGT1A1. Clinically, there is likelihood that axitinib plasma concentrations may be increased in the presence of co-administered strong inhibitors of CYP3A. The potential exists for drug-drug interactions with CYP3A inhibitors such as grapefruit juice, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, verapamil, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, and delavirdine. Caution should be exercised in patients receiving axitinib in combination with these and other strong CYP3A inhibitors Axitinib metabolism may be induced in patients taking CYP3A4 inducers (carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, primidone, rifabutin, rifampin, and *St John's wort*) and this may reduce axitinib plasma concentrations. Patients who require concomitant treatment with strong CYP3A inducers are not eligible for the trial. Since CYP1A2 is also known to be induced in chronic smokers, there is likelihood that axitinib plasma concentrations may be reduced in these individuals.

The ability of axitinib to increase concentrations of co-administered drugs was also investigated in studies with human liver microsomes. At expected therapeutic plasma concentrations (0.01 to 1.0  $\mu g/mL$ ), axitinib appears most likely to inhibit the drug metabolizing enzymes CYP1A2 and CYP2C8, 2 enzymes not frequently observed as predominant drug metabolizing enzymes. However co-administration of axitinib with paclitaxel, a CYP2C8 substrate did not increase plasma concentrations of paclitaxel in patients, indicating lack of clinical CYP2C8 inhibition. Axitinib is highly bound to proteins in human plasma (99.5% bound at concentrations of 0.2 to 20  $\mu g/mL$ ). Therefore, drug interactions with other agents that are also highly bound to plasma proteins are a possibility.

Patients who need to be on chronic antacid therapy with histamine H<sub>2</sub> antagonists (eg, cimetidine [Tagamet<sup>®</sup>], famotidine [Pepcid<sup>®</sup>], nizatidine [Axid<sup>®</sup>], ranitidine [Zantac<sup>®</sup>]) or proton-pump inhibitors (eg, lansoprazole [Prevacid<sup>®</sup>], rabeprazole [Aciphex<sup>®</sup>], pantoprazole [Protonix<sup>®</sup>], and esomeprazole [Nexium<sup>®</sup>]) or locally acting antacids (eg, Maalox<sup>®</sup>, Milk of Magnesia<sup>®</sup>, Amphojel<sup>®</sup>) should stagger the timing of their axitinib and antacid dosing. Patients should avoid use of antacids for 2 hours before through 2 hours after taking axitinib tablets.

Axitinib is not likely to have drug-drug interactions with commonly used antihypertensive agents belonging to the class of ACE inhibitors including angiotensin II receptor antagonists (enalapril, captopril, losartan, vasartan), beta-blockers (atenolol, metoprolol, labetalol), or diuretics (hydrochlorothiazide, furosemide). Within the class of calcium channel blockers, verapamil, and to a lesser extent nifedipine, nicardipine, and diltiazem have a potential for increasing axitinib plasma concentrations, due to CYP3A inhibition and should not be used as first choice in antihypertensive treatment. Other calcium channel blockers (amlodipine, bepridil, felodipine) are less likely to raise axitinib plasma levels. The above information is based on preclinical data from studies using human and animal metabolizing enzyme systems.

Patients who need to be on anticoagulant therapy during treatment with axitinib should be treated with low molecular weight heparin as the preferred therapy.

All concomitant medications and blood products, as well as interventions (eg, analgesic use or paracentesis) received by patients from the first dose of study drug until the end of study visit will be recorded on the case report form (eCRF).

Regarding the concomitant surgery, no formal studies of the effect of axitinib on wound healing have been conducted, however caution is advise based on the mechanism of action.

If a major surgery or an interventional procedure (eg, endoscopy) is required, treatment with axitinib must be interrupted at least 24 hours before the procedure.

Patients may resume the treatment with axitinib according to the opinion of the investigator, when wound has completely healed and there are no wound healing complications (eg, delayed healing, wound infection or fistula).

# 5.4.2. Concomitant Medication(s) (Combination Therapy, if applicable)

Details regarding allowed concomitant medications, surgery and/or radiotherapy with the combination therapy are described in the parent protocol (Appendix 1).

# 5.5. Rescue Therapy

No mechanistically specific antagonists for axitinib are available and standard supportive measures should be used in the case of excessive pharmacological effects or adverse reaction.

#### 6. TRIAL PROCEDURES

#### **6.1. Patient Enrollment**

To enroll patients the investigator must send a completed registration form to the appropriate Clinical representative. The investigator should be prepared to answer questions concerning the patient's eligibility. Once eligibility is verified the clinical representative will confirm by facsimile that the patient has been accepted into the trial. If the patient fails to start treatment within 14 days of registration the clinical representative should be contacted before the start of treatment.

#### **6.2. Trial Procedures**

During treatment on this protocol, all patients will be followed and monitored according to local clinical practice.

Safety monitoring and laboratory analyses are to be performed as clinically indicated.

TSH, T3 (or free T3) and/or free T4 should be performed as clinically indicated. If thyroid function tests were not performed during the 8 weeks before enrollment in this study, serum or plasma thyroid function tests (Free T4 and TSH) should be performed at screening/baseline visit, and subsequently as clinically indicated, and not less than every 12 weeks (±2 weeks).

Pregnancy tests and contraceptive check should be performed at screening/baseline visit (when clinically indicated), and repeated if clinically indicated, and/or required by IRB/IECs, or local regulations.

Tumor assessments should be performed per standard clinical practice and results should be recorded in the patient's clinic chart (but will not be collected in the study eCRF).

Only for patients previously enrolled in the parent protocol A4061068 and treated with axitinib and crizotinib the following assessments should be added:

• Liver function test ((alanine aminotransferase (ALT) and aspartate aminotransferase (AST), alkaline phosphatase, bilirubin): to be performed every 4 weeks. The tests should be performed preferably at the clinical site's local laboratory and, when not possible, patients will provide the results copy (from the nonclinical site laboratory), eg, by telephone, and bring a copy of the laboratory test results at the visit.

- Electrocardiogram (ECG): to be performed at the time of End of Treatment, and as clinically indicated;
- Ophthalmologic examination: at the first occurrence of any vision changes and as clinically indicated.

# 6.3. Follow-up Visit

If the patient discontinues the treatment (as monotherapy or combination therapy), a final safety evaluation including thyroid testing will be performed at least 28 days after the last dose of study drug(s) and documented in the source documents.

Only for patients previously enrolled in the parent protocol A4061068 and treated with axitinib and crizotinib, the following assessments should be added in the final evaluation:

- Liver function test (ALT and AST, Alkaline phosphatase, Bilirubin);
- ECG;
- Ophthalmologic examination (as clinically indicated).

Reported adverse events that are ongoing at the time of study discontinuation and serious, or ≥ grade 3 or suspected to be related to the study drug(s), or clinically significant by the investigator or Pfizer medical monitor must be followed after the time of therapy discontinuation until the event or its sequelae resolve/stabilize at a level acceptable to the investigator and the Pfizer medical monitor or his/her designated representative. Following the active safety reporting period, other serious adverse events (SAEs) of which the investigator becomes aware should be reported to Pfizer, unless the SAE is attributed by the investigator to complications of either the underlying malignancy or any subsequent anti-cancer therapy or to the patient's participation in a subsequent clinical study.

Concomitant medications/treatments, AE and thyroid lab CRF shall be updated accordingly.

After the follow up visit, attempts should be made, where possible, to collect information every 2 months on patient alive/death status via phone call or routine visit.

### 6.4. Patient Withdrawal

A patient may withdraw from the trial at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator or sponsor for safety or behavioral reasons, or the inability of the patient to comply with the protocol required schedule of study visits or procedures at a given study site. If a patient does not return for a scheduled visit, every effort should be made to contact the patient. In any circumstance, every effort should be made to document patient outcome, if possible. The investigator should inquire about the reason for withdrawal, request the patient to return all unused investigational product(s), request the patient to return for a final visit, if applicable, and follow-up with the patient regarding any unresolved adverse events (AEs).

If the patient withdraws consent, no further evaluations should be performed and no attempts should be made to collect additional data. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

#### 7. SAFETY ASSESSMENTS

The safety of axitinib and the study drug(s) given in combination should be evaluated using the local standard clinical practice.

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However it is anticipated that from time to time there may be circumstances, outside of the control of the investigator that may make it unfeasible to perform the test. In these cases the investigator will take all steps necessary to ensure the safety and well being of the patient. When a protocol required test cannot be performed, the investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. The study team will be informed of these incidents in a timely manner.

Patients receiving axitinib (either as monotherapy or in combination therapy) should be monitored for signs and symptoms of hypothyroidism, such as fatigue, deepening of voice, cold intolerance, constipation, anorexia, periorbital edema, myxedema, or changes in skin or hair. Hypothyroidism should be treated per standard medical practice to maintain euthyroid state.

In case of combination therapy, additional texts or examination might be required in accordance with the parent protocol(s) (see Section 6.2 and 6.3 above and, for more details, see relevant sections in parent protocol Appendix 1).

# **Pregnancy Test**

For female patients of child bearing potential (ie, who in the opinion of the investigator are biologically capable of having children and sexually active), a serum or urine pregnancy test will be performed at screening/baseline visit. Pregnancy tests will also be done whenever one menstrual cycle is missed during the active treatment period (or when potential pregnancy is otherwise suspected). Tests may also be repeated as per request of IRB/IECs or if required by local regulations.

#### 8. ADVERSE EVENT REPORTING

#### 8.1. Adverse Events

All observed or volunteered adverse events regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported as described in the following sections.

For all adverse events the investigator must pursue and obtain information adequate both to determine the outcome of the adverse event and to assess whether it meets the criteria for classification as a serious adverse event (See Section 8.6) requiring immediate notification to

Pfizer or its designated representative. For all adverse events sufficient information should be obtained by the investigator to determine the causality of the adverse event. The investigator is required to assess causality. Follow-up by the investigator may be required until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

As part of ongoing safety reviews conducted by the Sponsor, any non-serious adverse event that is determined by the Sponsor to be serious will be reported by the Sponsor as an SAE. To assist in the determination of case seriousness further information may be requested from the investigator to provide clarity and understanding of the event in the context of the clinical study.

# 8.2. Reporting Period

For serious adverse events, the active reporting period to Pfizer or its designated representative begins from the time that the patient provides informed consent, which is obtained prior to the patient's participation in the study, ie, prior to undergoing any study-related procedure and/or receiving investigational product, through and including 28 calendar days (longer follow up period might need to be adopted based on the combination drug characteristics) after the last administration of the investigational product. SAEs occurring to a subject after the active reporting period has ended should be reported to the sponsor if the investigator becomes aware of them; at a minimum, all SAEs that the investigator believes have at least a reasonable possibility of being related to investigational product are to be reported to the Sponsor. Adverse events (serious and non-serious) should be recorded on the CRF from the time the patient has taken at least one dose of investigational product through last patient's last visit.

If a patient begins a new anticancer therapy, the adverse event reporting period for non-serious adverse events ends at the time the new treatment is started.

Death must be reported if it occurs during the serious adverse event reporting period after the last dose of investigational product, irrespective of any intervening treatment.

#### 8.3. Definition of an Adverse Event

An adverse event is any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Examples of adverse events include but are not limited to:

- Abnormal test findings;
- Clinically significant symptoms and signs;
- Changes in physical examination findings;
- Hypersensitivity;

- Drug abuse;
- Drug dependency.

Additionally, they may include the signs or symptoms resulting from:

- Drug overdose;
- Drug withdrawal;
- Drug misuse;
- Drug interactions;
- Extravasation;
- Exposure during pregnancy;
- Exposure via breastfeeding;
- Medication error;
- Occupational exposure;
- Worsening of signs and symptoms of the malignancy under trial should be reported as adverse events in the appropriate section of the CRF. Disease progression assessed by measurement of malignant lesions on radiographs or other methods should not be reported as adverse events.

#### 8.4. Medication Errors

Medication errors may result, in this study, from the administration or consumption of the wrong product, by the wrong subject, at the wrong time, or at the wrong dosage strength. Such medication errors occurring to a study participant are to be captured on the medication error CRF, which is a specific version of the Adverse Event (AE) page, and on the SAE form when appropriate. In the event of medication dosing error, the sponsor should be notified immediately.

Medication errors are reportable irrespective of the presence of an associated AE/SAE, including:

- Medication errors involving subject exposure to the investigational product;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the participating subject.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is captured on the medication error version of the AE page and, if applicable, any associated AE(s) are captured on an AE CRF page.

#### 8.5. Abnormal Test Findings

The criteria for determining whether an abnormal objective test finding should be reported as an adverse event are as follows:

- Test result is associated with accompanying symptoms; and/or
- Test result requires additional diagnostic testing or medical/surgical intervention; and/or
- Test result leads to a change in trial dosing outside of protocol-stipulated dose adjustments or discontinuation from the trial, significant additional concomitant drug treatment, or other therapy; and/or
- Test result is considered to be an adverse event by the investigator or sponsor.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an adverse event. Any abnormal test result that is determined to be an error does not require reporting as an adverse event.

#### 8.6. Serious Adverse Events

A serious adverse event is any untoward medical occurrence at any dose that:

- Results in death;
- Is life-threatening (immediate risk of death);
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability/incapacity; (substantial disruption of the ability to conduct normal life functions);
- Results in congenital anomaly/birth defect.

Progression of the malignancy under study (including signs and symptoms of progression) should not be reported as an SAE unless the outcome is fatal within the safety reporting period. Hospitalization due to signs and symptoms of disease progression should not be reported as an SAE. If the malignancy has a fatal outcome during the study or within the safety reporting period, then the event leading to death must be recorded as an AE and as an SAE with CTCAE Grade 5 (see the Section 8.8 Severity Assessment).

Medical and scientific judgment should be exercised in determining whether an event is an important medical event. An important medical event may not be immediately life threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the patient or may require intervention to prevent one of the other AE outcomes, the important medical event should be reported as serious.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

# 8.6.1. Protocol-Specified Serious Adverse Events

There are no protocol-specified SAEs in this study. All SAEs will be reported by the investigator as described in previous sections, and will be handled as SAEs in the safety database (see the section on Serious Adverse Event Reporting Requirements).

# 8.6.2. Potential Cases of Drug-Induced Liver Injury

Abnormal values in AST and/or ALT concurrent with abnormal elevations in total bilirubin that meet the criteria outlined below in the absence of other causes of liver injury are considered potential cases of drug-induced liver injury (potential Hy's Law cases) and should always be considered important medical events.

The threshold of laboratory abnormalities for a potential case of drug-induced liver injury depends on the patient's individual baseline values and underlying conditions. Patients who present with the following laboratory abnormalities should be evaluated further to definitively determine the etiology of the abnormal laboratory values:

- Patients with AST or ALT and total bilirubin baseline values within the normal range who subsequently present with AST or ALT values ≥3 times the upper limit of normal (X ULN) concurrent with a total bilirubin value ≥2 X ULN with no evidence of hemolysis and an alkaline phosphatase value ≤2 X ULN or not available.
- For patients with preexisting ALT **OR** AST **OR** total bilirubin values above the upper limit of normal, the following threshold values should be used in the definition mentioned above:
  - For patients with pre-existing AST or ALT baseline values above the normal range: AST or ALT values ≥2 times the baseline values and ≥3 X ULN, or ≥8 X ULN (whichever is smaller).

#### • Concurrent with:

• For patients with pre-existing values of total bilirubin above the normal range: Total bilirubin increased by one time the upper limit of normal  $\mathbf{or} \ge 3$  times the upper limit of normal (whichever is smaller).

The patient should return to the investigational site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history and physical assessment. The possibility of hepatic neoplasia (primary or secondary) should be also considered. In addition to repeating AST and ALT, laboratory tests should include albumin, creatine kinase, total bilirubin, direct and indirect bilirubin, gamma-glutamyl transferase, prothrombin time (PT)/INR, and alkaline phosphatase. A detailed history, including relevant information, such as review of ethanol, acetaminophen, recreational drug and supplement consumption, family history, occupational exposure, sexual history, travel history, history of contact with a jaundiced patient, surgery, blood transfusion, history of liver or allergic disease, and work exposure, should be collected. Further testing for acute hepatitis A, B, or C infection and liver imaging (eg, biliary tract) may be warranted. All cases confirmed on repeat testing as meeting the laboratory criteria defined above, with no other cause for LFT abnormalities identified at the time should be considered potential Hy's Law cases irrespective of availability of all the results of the investigations performed to determine etiology of the abnormal LFTs. Such potential Hy's Law cases should be reported as SAEs.

# 8.7. Hospitalization

Hospitalization is defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility or any prolongation of an existing admission. Admission also includes transfer within the hospital to an acute/intensive care unit (eg, from the psychiatric wing to a medical floor, medical floor to a coronary care unit, neurological floor to a tuberculosis unit).

An emergency room visit does not necessarily constitute a hospitalization; however, the event leading to the emergency room visit should be assessed for medical importance.

Hospitalization does not include the following:

- Rehabilitation facilities;
- Hospice facilities;
- Respite care (eg, caregiver relief);
- Skilled nursing facilities;
- Nursing homes;
- Same day surgeries (as outpatient/same day/ambulatory procedures).

Hospitalization or prolongation of hospitalization in the absence of a precipitating, clinical adverse event is not in itself a serious adverse event. Examples include:

• Admission for treatment of a preexisting condition not associated with the development of a new adverse event or with a worsening of the preexisting condition (eg, for work-up of persistent pre-treatment lab abnormality);

- Social admission (eg, patient has no place to sleep);
- Administrative admission (eg, for yearly physical examination);
- Protocol-specified admission during a clinical trial (eg, for a procedure required by the trial protocol);
- Optional admission not associated with a precipitating clinical adverse event (eg, for elective cosmetic surgery);
- Hospitalization for observation without a medical AE;
- Pre-planned treatments or surgical procedures. These should be noted in the baseline documentation for the entire protocol and/or for the individual patient;
- Admission exclusively for the administration of blood products.

Diagnostic and therapeutic non-invasive and invasive procedures, such as surgery, should not be reported as adverse events. However, the medical condition for which the procedure was performed should be reported and it meets the definition of an adverse event. For example, an acute appendicitis that begins during the adverse event reporting period should be reported as the adverse event, and the resulting appendectomy should be recorded as treatment of the adverse event.

# 8.8. Severity Assessment

If required on the adverse event case report forms, the investigator will use the following definitions of severity in accordance with National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 to describe the maximum intensity of the adverse event. If the event is serious, the CTCAE grade reported in the adverse event CRF must be consistent with the description of CTCAE grade included in the narrative section of the serious adverse event report.

| GRADE | Clinical Description of Severity |
|---|---|
| 0 | No Change from Normal or Reference Range (This grade is not included in the Version 4.03 document but may be used in certain circumstances.) |
| 1 | MILD Adverse Event |
| 2 | MODERATE Adverse Event |
| 3 | SEVERE Adverse Event |
| 4 | LIFE-THREATENING OR DISABLING Adverse Event |
| 5 | DEATH RELATED TO Adverse Event |

Note the distinction between the severity and the seriousness of an adverse event. A severe event is not necessarily a serious event. For example, a headache may be severe (interferes significantly with patient's usual function) but would not be classified as serious unless it met one of the criteria for serious adverse events, listed above.

### 8.9. Causality Assessment

The investigator's assessment of causality must be provided for all adverse events (serious and non-serious), the investigator must record the causal relationship in the CRF, as appropriate, and report such an assessment in accordance with the serious adverse reporting requirements if applicable. An investigator's causality assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an adverse event; generally, the facts (evidence) or arguments to suggest a causal relationship should be provided. If the investigator does not know whether or not the investigational product caused the event, then the event will be handled as "related to investigational product" for reporting purposes, as defined by the Sponsor (See the Section on Reporting Requirements). If the investigator's causality assessment is "unknown but not related to investigational product," this should be clearly documented on trial records.

In addition, if the investigator determines a serious adverse event is associated with trial procedures, the investigator must record this causal relationship in the source documents and CRF, as appropriate, and report such an assessment in accordance with the serious adverse event reporting requirements, if applicable.

# 8.10. Exposure During Pregnancy

For both unapproved/unlicensed products and for marketed products, an exposure during pregnancy (EDP) occurs if:

- A female becomes, or is found to be, pregnant either while receiving or having been exposed (eg, because of treatment or environmental exposure) to the investigational product, or the female becomes or is found to be pregnant after discontinuing and/or being exposed to the investigational product;
- An example of environmental exposure would be a case involving direct contact with a Pfizer product in a pregnant woman (eg, a nurse reports that she is pregnant and has been exposed to chemotherapeutic products);
- A male has been exposed, (eg, because of treatment or environmental exposure), to the investigational product prior to or around the time of conception and/or is exposed during his partner's pregnancy.

If any study patient or study patient's partner becomes or is found to be pregnant during the study patient's treatment with the investigational product, the investigator must submit this information to Pfizer drug safety unit on an SAE Report Form and an EDP supplemental form, regardless whether an SAE has occurred. In addition, the investigator must submit information regarding environmental exposure to a Pfizer product in a pregnant woman (eg, a

subject reports that she is pregnant and has been exposed to a cytotoxic product by inhalation or spillage) using the EDP supplemental form. This must be done irrespective of whether an adverse event has occurred and within 24 hours of awareness of the exposure. The information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

Follow-up is conducted to obtain general information on the pregnancy and its outcome forall EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer of the outcome as a follow up to the initial EDP supplemental form.

In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for a serious adverse event (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise neonatal death, or congenital anomaly [in a live born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death], the investigator should follow the procedures for reporting serious adverse events.

Additional information about pregnancy outcomes that are reported as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as serious adverse events when the investigator assesses the neonatal death as related or possibly related to exposure to the investigational product.

Additional information regarding the EDP may be requested by the investigator. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the study patient with the Pregnant Partner Release of Information Form to deliver to his partner. The Investigator must document in the source documents that the patient was given the Pregnant Partner Release of Information Form to provide to his partner.

#### 8.11. Occupational Exposure

An occupational exposure occurs when, during the performance of job duties, a person (whether a healthcare professional or otherwise) gets in unplanned direct contact with the product, which may or may not lead to the occurrence of an AE.

An occupational exposure is reported to the drug safety unit within 24 hours of the investigator's awareness, using the SAE report form, regardless of whether there is an associated AE/SAE. Since the information does not pertain to a subject enrolled in the study, the information is not reported on a CRF; however, a copy of the completed SAE report form is maintained in the investigator site file.

# 8.12. Withdrawal Due to Adverse Events (See also Patient Withdrawal, Section 6.4)

Withdrawal due to adverse events should be distinguished from withdrawal due to other causes, according to the definition of adverse event noted earlier, and recorded on the appropriate adverse event CRF page.

When a patient withdraws because of a serious adverse event, the serious adverse event must be reported in accordance with the reporting requirements defined below.

## 8.13. Eliciting Adverse Event Information

The investigator is to report all directly observed adverse events and all adverse events spontaneously reported by the study patient. In addition, each study patient will be questioned about adverse events.

# 8.14. Reporting Requirements

Each adverse event is to be assessed to determine if it meets the criteria for serious adverse event. If a serious adverse event occurs, expedited reporting will follow local and international regulations, as appropriate.

#### 8.14.1. Serious Adverse Event Reporting Requirements

If a serious adverse event occurs, Pfizer is to be notified within 24 hours of investigator awareness of the event.

In particular, if the serious adverse event is fatal or life-threatening, notification to Pfizer must be made immediately, irrespective of the extent of available adverse event information. This timeframe also applies to additional new information (follow-up) on previously forwarded serious adverse event reports as well as to the initial and follow-up reporting of EDP and exposure via breastfeeding cases.

In the rare event that the investigator does not become aware of the occurrence of a serious adverse event immediately (eg, if an outpatient study patient initially seeks treatment elsewhere), the investigator is to report the event within 24 hours after learning of it and document the time of his/her first awareness of the adverse event.

For all serious adverse events, the investigator is obligated to pursue and provide information to Pfizer in accordance with the timeframes for reporting specified above. In addition, an investigator may be requested by Pfizer to obtain specific additional follow-up information in an expedited fashion. This information collected for SAEs is more detailed than that captured on the adverse event case report form. In general, this will include a description of the adverse event in sufficient detail to allow for a complete medical assessment of the case
and independent determination of possible causality. Information on other possible causes of the event, such as concomitant medications, vaccines, and/or illnesses must be provided. In the case of a patient death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer or its designated representative.

### 8.14.2. Non-Serious Adverse Event Reporting Requirements

All adverse events are to be reported on the adverse event page of the CRF. It should be noted that the form for collection of SAE information is not the same as the AE CRF. Where the same data are collected, the forms must be completed in a consistent manner. For example, the same AE term should be used on both forms. AEs should be reported using concise medical terminology on the CRFs as well as on the form for collection of SAE information.

# 8.14.3. Sponsor Reporting Requirements to Regulatory Authorities

Adverse event reporting, including suspected unexpected serious adverse reactions, will be carried out in accordance with applicable local regulations.

# 9. DATA ANALYSIS/STATISTICAL METHODS

## 9.1. Sample Size Determination

The sample size is not statistically driven and is dependent upon the number of patients included in the clinical trial program for axitinib (as monotherapy or in combination therapy) who are eligible for this extension study and wish to continue with the treatment.

### 9.2. Safety Analysis

All patients receiving at least 1 dose of axitinib (as monotherapy or combination therapy) under this protocol will be included in the safety analyses. Adverse events will be coded and grouped by body system. The incidence of each adverse event will be tabulated and displayed by starting dose level. Tabulations by maximum severity and relationship to Axitinib and/or with another anticancer drug(s) given in combination with axitinib, if applicable will also be included. Summary patient listings will be provided for SAEs, adverse events resulting in discontinuation of axitinib, and deaths within 28 days of drug discontinuation and possibly or probably related to axitinib or to the anticancer drug(s) given in combination with axitinib.

## 9.3. Efficacy Analysis

Efficacy will not be assessed in this protocol.

### 9.4. Data Monitoring Committee

This study will not use an external Data Monitoring Committee/Pfizer Safety Committee/Internal Oncology Business Unit-Safety Data Monitoring Committee.

For the purpose of this protocol, Pfizer procedures for periodic safety review will be applied by an internal safety review team with medical and statistical capabilities to review individual and summary data collected in the safety and clinical databases.

## 10. QUALITY CONTROL AND QUALITY ASSURANCE

During trial conduct, Pfizer or its agent will conduct periodic monitoring visits to ensure that the protocol and GCPs are being followed. The monitors may review source documents to confirm that the data recorded on CRFs is accurate. The investigator and institution will allow Pfizer monitors or its agents and appropriate regulatory authorities direct access to source documents to perform this verification.

The trial site may be subject to review by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC), and/or to quality assurance audits performed by Pfizer, or companies working with or on behalf of Pfizer, and/or to inspection by appropriate regulatory authorities.

It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

#### 11. DATA HANDLING AND RECORD KEEPING

# 11.1. Case Report Forms/Electronic Data Record

As used in this protocol, the term Case Report Form (CRF) should be understood to refer to either a paper form or an electronic data record or both, depending on the data collection method used in this trial.

A CRF is required and should be completed for each included patient. The completed original CRFs are the sole property of Pfizer and should not be made available in any form to third parties, except for authorized representatives of Pfizer or appropriate regulatory authorities, without written permission from Pfizer.

The investigator has ultimate responsibility for the collection and reporting of all clinical, safety and laboratory data entered on the CRFs and any other data collection forms (source documents) and ensuring that they are accurate, authentic/original, attributable, complete, consistent, legible, timely (contemporaneous), enduring and available when required. CRFs must be signed by the investigator or by an authorized staff member to attest that the data contained on the CRF is true. Any corrections to entries made in the CRFs, source documents must be dated, initialed and explained (if necessary) and should not obscure the original entry.

In most cases, the source documents will be the hospital's or the physician's chart. In cases where the source documents are the hospital or the physician's chart, the information collected on the CRFs must match those charts.

In some cases, the CRF, or part of the CRF, may also serve as the source document. In these cases, a document should be available at the investigator's site as well as at Pfizer and clearly identify those data that will be recorded in the CRF, and for which the CRF will stand as the source document.

### 11.2. Record Retention

To enable evaluations and/or audits from regulatory authorities or Pfizer, the investigator agrees to keep records, including the identity of all participating patients (sufficient information to link records, eg, CRFs and hospital records), all original signed informed consent documents, copies of all CRFs, serious adverse event forms, source documents, and detailed records of treatment disposition, and adequate documentation of relevant correspondence (eg, letters, meeting minutes, telephone calls reports). The records should be retained by the investigator according to International Conference on Harmonisation (ICH), local regulations, or as specified in the Clinical Study Agreement, whichever is longer.

If the investigator relocates, retires, or for any reason withdraws from the trial, Pfizer should be prospectively notified. The trial records must be transferred to a designee acceptable to Pfizer, such as another investigator, another institution, or to an independent third party arranged by Pfizer. Investigator records must be kept for a minimum of 15 years after completion or discontinuation of the study or for longer if required by applicable local regulations.

The investigator must obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

## 12. ETHICS

## 12.1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

It is the responsibility of the investigator to have prospective approval of the trial protocol, protocol amendments, informed consent forms, and other relevant documents, eg, recruitment advertisements, if applicable, from the IRB/IEC. All correspondence with the IRB/IEC should be retained in the Investigator File. Copies of IRB/IEC approvals should be forwarded to Pfizer.

The only circumstance in which an amendment may be initiated prior to IRB/IEC approval is where the change is necessary to eliminate apparent immediate hazards to the patients. In that event, the investigator must notify the IRB/IEC and Pfizer in writing immediately after the implementation.

## 12.2. Ethical Conduct of the Trial

The study will be conducted in accordance with legal and regulatory requirements, as well as the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects (Council for International Organizations of Medical Sciences 2002), Guidelines for GCP (ICH 1996), and the Declaration of Helsinki (World Medical Association 2008). Where mandated by local law, compliance with 1996 version of the Declaration of Helsinki applies.

In addition, the study will be conducted in accordance with the protocol, the ICH guideline on GCP, and applicable local regulatory requirements and laws.

#### 12.3. Patient Information and Consent

All parties will ensure protection of patient personal data and will not include patient names on any sponsor forms, reports, publications, or in any other disclosures, except where required by laws.

Patient names, address, birth date and other identifiable data will be replaced by a numerical code consisting of a numbering system provided by Pfizer in order to de-identify the trial patient. In case of data transfer, Pfizer will maintain high standards of confidentiality and protection of patient personal data.

The informed consent form must be in compliance with ICH GCP, local regulatory requirements, and legal requirements.

The informed consent form used in this study, and any changes made during the course of the study, must be prospectively approved by both the IRB/IEC and Pfizer before use.

The investigator must ensure that each study patient, or his/her legal representative, is fully informed about the nature and objectives of the study and possible risks associated with participation. The investigator, or a person designated by the investigator, will obtain written informed consent from each patient or the patient's legal representative before any study-specific activity is performed. The investigator will retain the original of each patient's signed consent form.

## 12.4. Reporting Of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable Competent Authority in any area of the World, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of the investigational product, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study patients against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the investigator becomes aware of.

### 13. DEFINITION OF END OF TRIAL

### 13.1. End of Trial in all Participating Countries

End of Trial in all participating countries is defined as the time at which all patients enrolled in the study have completed treatment on study.

#### 14. SPONSOR DISCONTINUATION CRITERIA

Premature termination of this clinical trial may occur because of a regulatory authority decision, change in opinion of the IRB/IEC, drug safety problems, or at the discretion of Pfizer. In addition, Pfizer retains the right to discontinue development of axitinib given as monotherapy or in combination at any time.

If a trial is prematurely terminated or discontinued, Pfizer will promptly notify the investigator. After notification, the investigator must contact all participating patients and the hospital pharmacy (if applicable) within a 4-week time period. As directed by Pfizer, all trial materials must be collected and all CRFs completed to the greatest extent possible.

### 15. PUBLICATION OF TRIAL RESULTS

Publication of study results is discussed in the CSA.

## 15.1. Communication of Results by Pfizer

Pfizer fulfills its commitment to publicly disclose clinical study results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the European Clinical Trials Database (EudraCT), and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations. In addition, Pfizer reports study results outside of the requirements of local laws/regulations pursuant to its standard operating procedures (SOPs).

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

www.clinicaltrials.gov

Pfizer posts clinical trial United Stated (US) Basic Results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a Pfizer product, regardless of the geographical location in which the study is conducted. US Basic Results are submitted for posting within 1 year of the primary completion date (PCD) for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

PCD is defined as the date that the final subject was examined or received an intervention for the purposes of final collection of data for the primary outcome, whether the clinical study concluded according to the prespecified protocol or was terminated.

### **EudraCT**

Pfizer posts European Union (EU) Basic Results on EudraCT for all Pfizer-sponsored interventional studies that are in scope of EU requirements. EU Basic Results are submitted for posting within 1 year of the PCD for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

www.pfizer.com

Pfizer posts Public Disclosure Synopses (clinical study report synopses in which any data that could be used to identify individual patients has been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the US Basic Results document is posted to www.clinicaltrials.gov.

### Documents within marketing authorization packages/submissions

Pfizer complies with the European Union Policy 0070, the proactive publication of clinical data to the European Medicines Agency (EMA) website. Clinical data, under Phase 1 of this policy, includes clinical overviews, clinical summaries, CSRs, and appendices containing the protocol and protocol amendments, sample CRFs, and statistical methods. Clinical data, under Phase 2 of this policy, includes the publishing of individual participant data. Policy 0070 applies to new marketing authorization applications submitted via the centralized procedure since 01 January 2015 and applications for line extensions and for new indications submitted via the centralized procedure since 01 July 2015.

### **Data Sharing**

Pfizer provides researchers secure access to patient-level data or full CSRs for the purposes of "bona-fide scientific research" that contribute to the scientific understanding of the disease, target, or compound class. Pfizer will make available data from these trials 24 months after study completion. Patient-level data will be anonymized in accordance with applicable privacy laws and regulations. CSRs will have personally identifiable information redacted.

Data requests are considered from qualified researchers with the appropriate competencies to perform the proposed analyses. Research teams must include a biostatistician. Data will not be provided to applicants with significant conflicts of interest, including individuals requesting access for commercial/competitive or legal purposes.

## 15.2. Publications by Investigators

Pfizer has no objection to publication by Investigator of any information collected or generated by Investigator, whether or not the results are favorable to the Investigational Drug. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Investigator will provide Pfizer an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.

Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to Pfizer at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

Investigator will, on request, remove any previously undisclosed Confidential Information (other than the study results themselves) before disclosure.

If the study is part of a multi-centre study, Investigator agrees that the first publication is to be a joint publication covering all centers. However, if a joint manuscript has not been submitted for publication within 12 months of completion or termination of the study at all participating sites, Investigator is free to publish separately, subject to the other requirements of this Section.

For all publications relating to the study, Institution will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, <a href="http://www.icmje.org/index.html#authorship">http://www.icmje.org/index.html#authorship</a>, established by the International Committee of Medical Journal Editors.

Publication of study results is also provided for in the Clinical Study Agreement between Pfizer and the institution. In this section entitled Publications by Investigators, the defined terms shall have the meanings given to them in the Clinical Study Agreement.

### 16. APPENDICES

**Appendix 1. Study Protocol A4061068** 

(reference document for patients under axitinib and crizotinib treatment)

# THIS APPENDIX ONLY APPLIES TO PATIENTS UNDER AXITINIB AND CRIZOTINIB TREATMENT COMBINATION

Note that sections of this document have been cross-linked within protocol A4061008 to facilitate retrieval of relevant information.

Please check what applies and refer to protocol A4061008 for all other study processes and schedule.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017



#### CLINICAL PROTOCOL

A PHASE 1B, OPEN LABEL, DOSE ESCALATION STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AXITINIB (AG-013736) IN COMBINATION WITH CRIZOTINIB (PF-02341066) IN PATIENTS WITH ADVANCED SOLID TUMORS

Investigational Product Numbers: AG-013736, PF-02341066

Investigational Product Names: axitinib, crizotinib

United States (US) Investigational New IND 63,662 Drug (IND) Numbers: IND 73,544

European Clinical Trials Database 2015-001724-31 (EudraCT) Number

Protocol Number: A4061068

Phase: 1b

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### **Document History**

| Document | Version Date | Summary of Changes and Rationale |
|---|---|---|
| Amendment 3 | ()9 June 2017 | Main changes include: Discontinuation of enrollment in Expansion phase Cohort 2 (at least one but no more than two prior systemic treatment regimens directed at advanced RCC). Revision and simplification of Schedule of Activities procedures where applicable. Update of safety information to align with the most recent versions of axitinib and crizotinib Investigator Brochure (IB). Update protocol wording where possible (in particular the safety wording) to align with current Pfizer SOP (Standard Operating Procedures). |
| Amendment 2 | 27 January 2016 | Added EudraCT number. SCHEDULE OF ACTIVITIES: - Contraception check added to align with the Sponsor's most recent protocol template. - Registration and Study Treatment: updated to clarify which patient subgroup will receive axitinib single agent during a 7-day Lead-In period and which subgroup will start with the combination without the Lead-In period. - Archival Tumor Tissue, De Novo Tumor Biopsy: footnotes updated to align with Patient Selection Section, Inclusion Criterion #1. Section 1. Introduction: literature updated; axitinib and crizotinib safety data updated according to the last version of the Investigator's Brochure. Section 4. Patient Selection: |
| | | <ul> <li>Inclusion Criterion #1, Dose Expansion<br/>Phase: language updated: 1, to make the<br/>selected patient population more in line<br/>with the actual 2<sup>nd</sup> and 3<sup>rd</sup> line advanced<br/>RCC population; 2, to include alternative<br/>option for the collection of biopsy in the</li> </ul> |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| | | Dose Expansion Cohort 2 patients |
|---|---|---|
| | - 1 | <ul> <li>Exclusion Criterion #8; language<br/>updated to align with the current<br/>standard language of crizotinib clinical<br/>protocols.</li> </ul> |
| | | PK wording; whenever needed, the wording was updated to clarify that PK samples will be collected in at least 8 evaluable patients in the Expansion Phase Cohort 1. |
| | | The protocol wording (including pregnancy, contraception, AE Reporting, and publication of study results) and sections numbering were updated according to the Sponsor's most recent protocol template. The protocol language (including renal cyst monitoring, overdose instructions, concomitant medications, ophthalmology examinations) was updated according to the current standard language of crizotinib and axitinib clinical protocols. |
| Amendment 1 | 11 March 2014 | SCHEDULE OF ACTIVITIES: - Frequency of hepatic laboratory test monitoring and relevant footnote modified in accordance with the Dear Investigator Letter dated 23Oct2013. - Follow Up for dosing compliance: added recommendation to follow up for dosing compliance also whenever there is a dose change. - Tumor Assessments: footnote updated to be consistent with Section 7.5. Tumor Response Assessments - Home blood pressure monitoring, pulse rate: frequency and relevant footnote updated to clarify it has to be monitored starting from patient registration. - Archived tumor tissue: footnote updated to be consistent with Section 4, Patient Selection. |
| | | Section 4. Patient Selection: - Inclusion Criteria #1: language updated to clarify the collection of archival tumor tissue in the Dose Escalation Phase Inclusion Criteria #10: language about legal representative deleted in |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| | | accordance with Western Institutional Review Board request Inclusion Criteria #8, Exclusion Criteria #2, and Exclusion Criteria #7: language updated to clarify the criteria. Section 5.3.2.2. Dose Modifications in Case of Drug-Related Toxicity — Table 5: - Management of bradycardia modified in accordance with the recently updated erizotinib Core Data Sheet. Section 5.3.5. Compliance: added recommendation to perform follow up by |
|---|---|---|
| | | telephone whenever there is a dose change. Section 5.5.4. Other Concomitant Medications: - Language on concomitant use of anticoagulants updated. - Language on concomitant use of bradycardia inducing agents updated. |
| | | Section 6.1.1. Archival Tumor Tissue:<br>language updated to be consistent with<br>Section 4. Patient Selection. |
| | | Section 7.1.6. Ophthalmologic<br>Examinations and Section 9.6.4.<br>Ophthalmologic Data: language updated<br>to clarify optional tests to be done based<br>on clinical judgement. |
| | | Section 7.5 Tumor Response<br>Assessments: language updated to be<br>consistent with the Schedule of<br>Activities |
| | | Section 12.3. Patient Information and<br>Consent: language about legal<br>representative deleted in accordance with<br>Western Institutional Review Board<br>request. |
| Original protocol | 10 July 2013 | Not Applicable (N/A) |

This amendment incorporates all revisions to date, including amendments made at the request of country health authorities and institutional review boards (IRBs)/ethics committees (ECs).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

# TABLE OF CONTENTS LIST OF FIGURES 10 APPENDICES 10 1.2.3.1, c-MET and Resistance to Antiangiogenic Therapy ................21 1.2.3.2. Hypothesis to be Tested .......23 1.2.4.1. Crizotinib (XALKORI®, PF-02341066) as a c-MET Inhibitor ......23 1.2.4.2. Axitinib (INLYTA®, AG-013736)......25 2. STUDY OBJECTIVES AND ENDPOINTS 28 3.1. Study Overview 29 3.1.1.1. Starting Doses for Axitinib and Crizotinib (Dose Level 1) ......31 3.1.2. DLT Definition 34 3.1.5. Dose Expansion Phase \_\_\_\_\_\_35

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| CONTRACTOR OF THE PROPERTY OF | |
|---|---|
| 4. PATIENT ELIGIBILITY CRITERIA | 35 |
| 4.1. Inclusion Criteria | 35 |
| 4.2. Exclusion Criteria | 38 |
| 4.3. Life Style Guidelines | 40 |
| 4.3.1. Sunlight Exposure | 40 |
| 4.3.2. Contraception | 40 |
| 4.4. Sponsor Qualified Medical Personnel | 41 |
| 5. STUDY TREATMENTS | 42 |
| 5.1, Allocation to Treatment | 42 |
| 5.2. Investigational Product Supplies | 43 |
| 5.2.1. Dosage Form(s) and Packaging | 43 |
| 5.2.1.1. Axitinib | 43 |
| 5.2.1.2. Crizotinib | 43 |
| 5.2.2 Preparation and Dispensing | 43 |
| 5.3. Administration | 43 |
| 5.3.1. Food Requirements | 44 |
| 5.3.2. Recommended Dose Modifications | 44 |
| 5.3.2.1. Axitinib Intra-Patient Dose Escalation | 44 |
| 5,3,2,2. Dose Modifications in Case of Drug-Related Toxicity, | 45 |
| 5.3.2.3. Management of Axitinib-Related Hypertension | 51 |
| 5.3.3. Crizotinib-Related Adverse Events Safety Monitoring | 51 |
| 5.3.3.1. Pneumonitis | 51 |
| 5.3.3.2. Renal Cyst | 52 |
| 5.3.4. Overdose Instructions | 52 |
| 5.3.5. Compliance | 52 |
| 5.4. Investigational Product Storage and Accountability | 53 |
| 5.5, Concomitant Medication(s) | 54 |
| 5.5.1. Inhibitors and Inducers of CYP Enzymes | 54 |
| 5.5,2. Hematopoietic Growth Factors | 55 |
| 5,5,3. Anti Diarrhea, Anti Emetic Therapy | 55 |
| 5,5,4. Other Concomitant Medications, | 55 |
| 5.5.5. Concomitant Surgery | 56 |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| 5.5.6, Concomitant Radiotherapy | 56 |
|---|---|
| 6. STUDY PROCEDURES | 57 |
| 6.1. Screening | 57 |
| 6.1.1. Archival Tumor Tissue | 57 |
| 6.1.2. De Novo Tumor Biopsy | 57 |
| 6.2. Study Period | 57 |
| 6.3. Follow-up Visit | 58 |
| 6.4. Patient Withdrawal | 58 |
| 7. ASSESSMENTS. | 59 |
| 7.1. Safety Assessment | 59 |
| 7.1.1. Pregnancy Testing | 59 |
| 7.1.2. Adverse Events | 60 |
| 7.1.3. Laboratory Safety Assessment | 60 |
| 7.1,4, Vital Signs and Physical Examination | 61 |
| 7.1.5. ECG Measurements | 61 |
| 7.1.6. Ophthalmology Examinations | 61 |
| 7.2. Pharmacokinetics Assessments | 63 |
| 7.2.1. Blood Sample Collection for Pharmacokinetic Analysis | 63 |
| 7.2.2. Collection of Crizotinib PK Samples | 64 |
| 7.2.3. Collection of Axitinib PK Samples | 64 |
| 7.2.4. Processing, Storage and Shipment of Crizotinib and Axitinib PK Samples | |
| 7.3. Pharmacodynamic Assessments | 65 |
| 7.3.1. Archived Tumor Tissue and De Novo Tumor Biopsies | 65 |
| 7.3.2. Peripheral Blood | 65 |
| 7.4. Banked Biospecimens | 66 |
| 7.4.1. Markers of Drug Response | 66 |
| 7.4.2. Additional Research | 67 |
| 7,5. Tumor Response Assessments | 67 |
| 8. ADVERSE EVENT REPORTING | 68 |
| 8.1. Requirements. | 68 |
| 8.1.1. Additional Details On Recording Adverse Events on the CRF | 69 |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| 8.1.2. Eliciting Adverse Event Information | 69 |
|---|---|
| 8.1.3. Withdrawal From the Study Due to Adverse Events (see also the Patient Withdrawal section) | 69 |
| 8.1.4. Time Period for Collecting AE/SAE Information | 70 |
| 8.1.4.1. Reporting SAEs to Pfizer Safety | 70 |
| 8.1.4.2. Recording Non-serious AEs and SAEs on the CRF | 70 |
| 8.1.5. Causality Assessment | 70 |
| 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities | 71 |
| 8.2. Definitions | 71 |
| 8.2.1. Adverse Events | 71 |
| 8.2.2. Abnormal Test Findings | 72 |
| 8.2.3. Serious Adverse Events | 72 |
| 8.2.4. Hospitalization | 73 |
| 8.3. Severity Assessment | 74 |
| 8.4. Special Situations | 75 |
| 8.4.1. Potential Cases of Drug-Induced Liver Injury | 75 |
| 8.4.2. Exposure to the Investigational Product During Pregnancy or<br>Breastfeeding, and Occupational Exposure | 76 |
| 8.4.2.1. Exposure During Pregnancy | 76 |
| 8.4.2.2. Exposure During Breastfeeding | 78 |
| 8.4,2.3. Occupational Exposure | 78 |
| 8.4.3. Medication Errors | 78 |
| 8.4.3.1. Medication Errors | 78 |
| 9. DATA ANALYSIS/STATISTICAL METHODS | 79 |
| 9.1. Analysis sets | 79 |
| 9.2. Statistical Methods and Properties | 80 |
| 9.2.1. Statistical Methods for Dose Escalation/De-Escalation: mTPI | 80 |
| 9.2.2. Statistical Method for Estimating the MTD | 81 |
| 9.3. Sample Size Determination | 82 |
| 9.4. Efficacy Analysis | 82 |
| 9.4.1. Analysis of Efficacy Endpoints (Dose Expansion Phase Cohorts) | 82 |
| 9.5, Analysis of Other Endpoints | 83 |
| 9.5.1. Analysis of Pharmacokinetics | 83 |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| 9.5.1.1. Pharmacokinetic Analysis of Crizotinib and Axitinib | 83 |
|---|---|
| 9.5.1.2. Effect of Crizotinib on Axitinib Pharmacokinetics | 84 |
| 9.5.1.3. Population Pharmacokinetic Analysis or PK/PD Modeling | g84 |
| 9.5.1.4. Statistical Analysis of Biomarker Endpoints | 84 |
| 9.6. Safety Analysis | 84 |
| 9.6.1. Analysis of Primary Safety Endpoint | 84 |
| 9.6.2. Analysis of Secondary Safety Endpoints | 85 |
| 9.6.2.1. Adverse Events | 85 |
| 9.6,2,2. Laboratory Tests Abnormalities | 85 |
| 9.6.2.3. ECG | 85 |
| 9.6.3, Concomitant Medications/Follow-up Systemic Therapy | 85 |
| 9.6.4. Ophthalmologic Data | 85 |
| 9.7. Data Monitoring Committee | 86 |
| 10. QUALITY CONTROL AND QUALITY ASSURANCE | 86 |
| 11. DATA HANDLING AND RECORD KEEPING | 87 |
| 11.1. Case Report Forms/Electronic Data Record | 87 |
| 11.2. Record Retention | 87 |
| 12. ÉTHICS | 88 |
| 12.1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 88 |
| 12.2. Ethical Conduct of the Study | 88 |
| 12.3. Patient Information and Consent | 88 |
| 12.4. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH | |
| GCP | |
| 13. DEFINITION OF END OF TRIAL | 89 |
| 13.1. End of Trial in a Member State | 89 |
| 13.2. End of Trial in all other Participating Countries | |
| 14. SPONSOR DISCONTINUATION CRITERIA | 90 |
| 15. PUBLICATION OF STUDY RESULTS | 90 |
| 15.1. Communication of Results by Pfizer | 90 |
| 15.2. Publications by Investigators | 91 |
| 16 DEFEDENCES | 02 |

AG-013736, PF-02341066

Figure 2.

# THIS APPENDIX ONLY APPLIES TO PATIENTS UNDER AXITINIB AND CRIZOTINIB TREATMENT COMBINATION

| | LIST OF TABLES | |
|---|---|---|
| Table 1. | Dose Levels in Dose Escalation Phase | 3 |
| Table 2. | Possible Dose-Finding Sequences | 32 |
| Table 3. | Axitinib Dose Levels | 44 |
| Table 4 | Crizotinib Dose Levels | 44 |
| Table 5. | Dose Modifications for Drug-Related Toxicity | 46 |
| Table 6. | Required Laboratory Tests | 60 |
| Table 7. | Intraocular Inflammation Grading Scale for Biomicroscopy | 62 |
| | LIST OF FIGURES | |
| Figure 1. | Pharmacokinetic Simulations Indicating the Predicted Increase in Exposure of Axitinib when Combined with Crizotinib | 27 |

### APPENDICES

| Appendix 3. National Cancer Institute (NCI) Common Terminology Criteria for | |
|---|---|
| Adverse Events (CTCAE) | 99 |
| Appendix 4. Abbreviations and Definitions of Term | 100 |
| Appendix 5. Detailed Dose Escalation/De-Escalation Scheme | 103 |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### PROTOCOL SUMMARY

#### **Background and Rationale:**

Until 2005, interferon-alpha (IFN-\alpha) and high dose interleukin (IL)-2 cytokine-based therapies were the conventional treatments for patients with advanced renal cell cancer (RCC), but efficacy was modest. Since then, multiple vascular endothelial growth factor (VEGF) inhibitors and mammalian target of rapamycin (mTOR) inhibitors have supplanted cytokines as the cornerstone of therapy. VEGF inhibitors include VEGF receptor (VEGFR) tyrosine kinase inhibitors (TKIs) axitinib, sunitinib, pazopinib, and sorafenib, and the monoclonal anti-VEGF antibody bevacizumab.

Despite the success of these anti-angiogenic therapies in multiple treatment settings including RCC, a fraction of patients are refractory to VEGF inhibitors, and the majority of patients will eventually develop evasive resistance and exhibit disease progression while on therapy. Nonclinical models suggest that at progression, the resistant tumor is aggressive both locally and at distant metastatic sites. Several mechanisms have been proposed to explain these phenomena. Recent data support a significant role for the membrane receptor tyrosine kinase mesenchymal-epithelial transition factor (c-MET) and its ligand hepatocyte growth factor (HGF) (or scatter factor) in tumor resistance to VEGF inhibitors.

It is therefore proposed that combining a c-MET inhibitor with a VEGF inhibitor will provide clinical benefit compared to treatment with a VEGF pathway directed therapy alone. This supports the testing of crizotinib, as c-MET inhibitor, in combination with the VEGFR inhibitor axitinib. Since this will be the first study of axitinib given in combination with crizotinib, the primary objective of the study will be the assessment of the safety and tolerability of the combination regimen. However, once the tolerability of the combination has been confirmed, its antitumor activity will be preliminarly assessed in advanced RCC expansion cohorts in both the first line setting, and second/third line setting following disease progression on a VEGF pathway inhibitor. This will explore the activity of the combination in both preempting the development of resistance to VEGF pathway inhibitor and in treating tumors already resistant to VEGF pathway inhibitor.

#### Rationale for Protocol Amendment #3

The patient enrollment was completed as per protocol in the Escalation Phase of the study, with axitinib 5 mg twice/day (BID) plus crizotinib 250 mg BID established as the maximum tolerated dose (MTD), and also in the Expansion Phase Cohort 1 (no prior systemic therapy directed at advanced RCC).

As for Expansion phase Cohort 2 (at least one but no more than two prior systemic treatment regimens directed at advanced RCC), it was decided to discontinue the enrollment in this cohort due to the competitive landscape, that made the identification of eligible patients extremely challenging (7 patients were enrolled in Cohort 2 in about 1.5 years). Due to the small patient population and the decision to discontinue enrollment in Cohort 2, biomarker analyses will be performed only on Cohort 1.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

As of 01 March 2017, 24 patients were enrolled (22 patients treated) in the dose Escalation Phase, at four dose levels: axitinib 3 mg BID + crizotinib 200 mg BID (n=5), axitinib 3 mg BID + crizotinib 250 mg BID (n=3), axitinib 5 mg BID + crizotinib 200 mg BID (n=4), and axitinib 5 mg BID + crizotinib 250 mg BID (n=10). There were no Cycle 1 dose-limiting toxicities and axitinib 5 mg BID + crizotinib 250 mg BID was established as the MTD. The most frequent all causalities adverse events (AEs) in the MTD group were fatigue (70%), nausea (70%), diarrhea (60%) and vomiting (50%), mainly of severity grade 1-2.

In the Expansion Phase, 27 patients with advanced RCC have been treated at the MTD; 21 patients in Cohort 1, and 6 patients in Cohort 2 (one additional patient was enrolled in Cohort 2 on 6<sup>th</sup> March 2017, for a total of 7 patients, then the enrolment was discontinued in that cohort). The regimen has shown manageable toxicities in the two expansion cohorts, with diarrhea (63%), nausea (59%), dysphonia (44%), fatigue (44%) and vomiting (44%) as most frequent all causalities AEs. The response evaluation (as per Response Evaluation Criteria in Solid Tumors [RECIST] v1.1) is ongoing, with 4 partial responses (PR) in Cohort 1, and 1 PR in Cohort 2.

Overall, there are 11 patients (10 male and 1 female) currently continuing treatment in study A4061068, and they have received at least 5 treatment cycles. The main purpose of this amendment is to simplify the study procedures, where possible, for the patients on active study treatment.

During treatment on this protocol amendment, the patients will be evaluated for safety and for efficacy per local clinical practice, but not less than every 12 weeks (±2 weeks), except for liver function tests to be done at least every month. Axitinib and crizotinib dosing and concomitant treatments will be monitored, too. Follow up information will be collected until follow up visit (Day 28 after the last study treatment dose). Pending drug availability, patients may continue to receive axitinib until they are no longer receiving clinical benefit according to the investigator's judgment.

#### Objectives and Primary Endpoint:

#### **Primary Objective**

To assess the safety and tolerability of axitinib in combination with crizotinib in
patients with solid tumors and advanced RCC in order to estimate the maximum
tolerated dose (MTD) (or Maximum Feasible Dose [MFD]) and select the
recommended Phase 2 dose (RP2D).

#### Secondary Objectives

- · To evaluate the overall safety profile.
- To characterize the pharmacokinetics (PK) of axitinib and crizotinib when administered in combination and to assess the effect of crizotinib on the PK of axitinib (Dose Escalation Phase and at least 8 PK-evaluable subjects in Expansion Phase Cohort 1 only).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- · To characterize the effects of axitinib in combination with crizotinib on QTc.
- To document the anti-tumor activity of axitinib in combination with crizotinib in advanced RCC patients.
- To explore the pharmacodynamic effect of axitinib in combination with crizotinib in blood.
- To characterize the alterations and/or expression profiles of genes, proteins, and RNAs relevant to angiogenesis (eg. Ang-2), drug targets (eg. c-MET) and sensitivity and/or resistance (eg. PBRM1) to axitinib in combination with crizotinib in tumor and/or blood.

The primary endpoint of the study is first-cycle dose limiting toxicities (DLTs).

#### Study Design:

This is a Phase 1b, open-label, multi-center, multiple-dose, safety, PK and pharmacodynamic study of axitinib in combination with crizotinib in adult patients with advanced solid tumors. This clinical study will be composed of a Dose Escalation Phase and a Dose Expansion Phase. The Dose Escalation Phase will estimate the MTD in dose escalation cohorts in patients with advanced solid tumors, using the modified toxicity probability interval (mTPI) method.

The Dose Escalation Phase will lead to the identification of an Expansion Test Dose for axitinib in combination with crizotinib in patients with solid tumors. The Expansion Test Dose will be either the MTD or the MFD, ie, the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor. Once the Expansion Test Dose is identified, the Dose Expansion Phase will be opened and axitinib in combination with crizotinib will be tested in patients with advanced RCC.

The Dose Expansion Phase is comprised of two patient populations, both with histologically or cytologically confirmed advanced RCC with a component of clear cell subtype and:

- Cohort 1: No prior systemic therapy directed at advanced RCC.
- Cohort 2: At least one but no more than two prior systemic treatment regimens
  directed at advanced RCC, with at least one prior therapy being a regimen containing
  an approved VEGF-pathway inhibitor, and resistance to the most recently received
  approved VEGF-pathway inhibitor. Resistance is defined as disease progression as
  per RECIST version 1.1 while on treatment with a VEGF-pathway inhibitor.

To understand the PK effects of crizotinib on axitinib, a 7-day lead-in period of single-agent axitinib directly preceding the administration of the crizotinib and axitinib combination will be included prior to Cycle 1 in the Dose Escalation Phase of the study. Axitinib is not expected to affect crizotinib exposure so there will be no PK study with a lead-in period of single-agent crizotinib. The Dose Expansion Phase Cohort 1 will be used to further study crizotinib and axitinib PK interactions in at least 8 evaluable patients; in this cohort, the PK profile for axitinib single agent during the 7-day lead-in period will be compared to that of

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

axitinib in combination with crizotinib during Cycle 1. No lead-in period will be included in the Dose Expansion Phase Cohort 2.

Given the safety profile of crizotinib, in addition to standard safety tests, ophthalmology examinations will be carried out to assess any vision changes. Based on the safety profile of axitinib, blood pressure will be monitored throughout the treatment period, as well as thyroid function.

Electrocardiogram (ECG) measurements will be taken throughout the treatment period in allpatients and in conjunction with PK sampling in patients from the Dose Escalation Phase and the Dose Expansion Phase Cohort 1. Archived tumor tissues will be collected for all patients. De novo tumor biopsy will be collected for the patients in the Dose Expansion Phase Cohort 2. Biomarker studies on tumor tissue and blood will be carried out to help understand the mechanism of action of the axitinib plus crizotinib combination, as well as potential mechanisms of resistance. Such results may help in the future development of this combination. These analyses may also result in the identification of potential biomarkers of response to the axitinib plus crizotinib combination, ultimately leading to development of a patient selection strategy for further clinical investigation.

Up to 65 patients are expected to be enrolled in the study.

#### Study Treatment:

Crizotinib and axitinib will be given orally (PO) twice daily (BID) on a continuous dosing schedule in 28-day cycles. Treatment with study drugs will continue until disease progression, patient refusal, patient lost to follow up, or unacceptable toxicity occurs, or the study is terminated by the Sponsor. Patients with unacceptable toxicity attributed to one of the two drugs may be eligible for continued treatment with the other drug (after discussion between the Investigator and the Sponsor). Patients with disease progression but who are still experiencing clinical benefit will be eligible for continued treatment with single agent axitinib or axitinib combined with crizotinib provided that the treating physician has determined that the benefit/risk for doing so is favorable.

#### Statistical Methods:

Up-and-Down Matrix Design with the mTPI Method

The escalation/de-escalation rules will follow the modified toxicity probability interval (mTPI) method<sup>38</sup> (see Section 9.2 and Appendix 5). Briefly, the mTPI method relies upon a statistical probability algorithm, calculated using all patients treated in prior and current cohorts at the same dose level) to determine where future cohorts should involve dose escalation, no change in dose, or dose de-escalation.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Rules for dose-finding, using the mTPI method, include the following:

- The target enrollment cohort size is 3 patients. The first 3 patients treated in Dose Level 1 cohort will initiate dosing sequentially, at least 2 days apart to allow for the initial evaluation of toxicities and tolerability. If there are no safety concerns, any additional patients enrolled to this dose cohort will not be required to initiate dosing sequentially.
- The next cohort can be enrolled when all patients at the current dose cohort have been
  evaluated for 28 days (ie, the first treatment cycle), or experience a dose limiting
  toxicity (DLT), whichever comes first.
- If a patient withdraws from the study before receiving at least 75% of the planned first-cycle dose of both axitinib and crizotinib for reasons other than study drug-related toxicity, another patient will be enrolled to replace that patient at the current dose level.
- The dose-finding component of the trial is completed when at least 10 evaluable
  patients have been treated at the highest dose associated with a DLT rate <0.33. It is
  estimated that approximately 25 DLT evaluable patients will need to be enrolled to
  reach 10 DLT-evaluable patients at the estimated MTD.</li>
- The proposed doses, schedule and PK timepoints may be reconsidered and amended during the study based on the emerging safety and PK data.
- The RP2D will be confirmed in the Dose Expansion Phase, taking into account the MTD/MFD determination from the Dose Escalation Phase, and other factors related to safety, efficacy, and PK/PD involving all available data from tests cohorts.

#### Sample Size Determination

Due to the dynamic nature of the cohort allocation procedure used in this study, the sample size of the Up-and-Down matrix design using the mTPI approach cannot be determined in advance. It is estimated that 25 DLT evaluable patients will be enrolled in the Dose Escalation Phase in order to have a reliable and accurate estimate of the MTD. The two expansion cohorts will enroll up to 20 response evaluable patients each at the estimated MTD or MFD.

Expansion phase Cohort 2 (at least one but no more than two prior systemic treatment regimens directed at advanced RCC): it was decided to discontinue the enrollment in this cohort due to the competitive landscape, that made the identification of eligible patients extremely challenging (7 patients were enrolled in Cohort 2 in about 1.5 years).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### SCHEDULE OF ACTIVITIES

The Schedule of Activities table (SOA) provides an <u>overview</u> of the protocol visits and procedures. Refer to ASSESSMENTS section of the protocol for detailed information on each assessment required for compliance with the protocol.

The Investigator may schedule visits (unplanned visits) in addition to those listed in the Schedule of Activities table in order to conduct evaluations or assessments required to protect the well-being of the patient.

AG-013736, PF-02341066-A4061068 Final Protocol Amendment 3, 09 June 2017

#### SCHEDULE OF ACTIVITIES

At the time of this protocol amendment, the 11 patients on active treatment have received at least 5 treatment cycles. The simplified Schedule of Activities below shows the activities applicable to those patients from Cycle 6 on.

Note: the 11 patients on active treatment are 10 male and 1 female in postmenopausal status for ≥ 2 years. Based on that, the pregnancy test is no longer required in the simplified Schedule of Activities. In addition, for patient benefit, biomarker samples will not be further collected at the end of treatment visit as enough samples have been obtained for required analyses.

| Protocol Activities[1] | Study Treatment (1 cycle = 28 days) | Post Treatment | |
|---|---|---|---|
| | Cycles ≥ 6 Frequency according to local clinical practice, but not less than every 12 weeks (±2 weeks) | End of Treatment<br>/Withdrawal<br>(±3 days) <sup>[2]</sup> | Follow-up<br>Day 28 (+7 days) after Las<br>Dose <sup>[7]</sup> |
| Documentation | | ****** | 3 |
| Physical Examination 111 | X | X | |
| ECOG Performance Status | X | X | |
| Blood Pressure, Pulse Ratel <sup>1</sup> | X | Х- | |
| Home Blood Pressure<br>Monitoring, Pulse Rate [6] | , | C | |
| Ophthalmologic<br>Examination 1 | At the first occurrence of any vision | n changes and as clinically | indicated |
| Laboratory Studies | | | The second |
| Hematology <sup>[8]</sup> | X | X | |
| Blood Chemistry <sup>[1]</sup> | (except liver function, to be monitored once per cycle) | X | |
| Congulation <sup>(11)</sup> | X | X | |
| Urmalysis <sup>19</sup> | X | X | |
| 12-lead ECG <sup>10)</sup> | | X | |
| Thyroid Function Tests [11] | X | | |
| Contraception check[12] | 3 | X | |
| Disease Assessments | | | |
| Tumor Assessments<br>(including scans)[13] | 3 | X. | |
| Other Clinical Assessments | | | |
| Adverse Events[14] | | ( | |

A(1-013736, PF-02341066-A4061068 Final Protocol Amendment 3, 09 June 2017.

| Protocol Activities[1] | Study Treatment (1 cycle = 28 days) | Post Treatment | |
|---|---|---|---|
| | Cycles ≥ 6 Frequency according to local clinical practice, but not less than every 12 weeks (±2 weeks) | End of Treatment<br>/Withdrawal<br>(±3 days) <sup>[2]</sup> | Follow-up<br>Day 28 (+7 days) after Last<br>Dose <sup>[5]</sup> |
| Concomitant<br>Medications/Treatments <sup>[15]</sup> | X X | X | X |
| Study Treatment [16] | | | |
| Crizotinib | X (twice daily) | | |
| Axitinib | X (twice daily) | | |

#### Footnotes for Schedule of Activities

- Protocol Activities: All assessments should be performed prior to dosing with study medications unless otherwise indicated. Acceptable time windows for performing each assessment are described in the column headings. Patients will visit site at Day 1 of each Cycle, End of Treatment and Follow-up
- End of Treatment/Withdrawal: Obtain these assessments ±3 days of End of Treatment/Withdrawal if not completed in the last week, except for
- tumor assessment which need not be repeated if performed within the prior 12 weeks.

  Follow-up Day 28 after last dose: To occur at least 28 days, and no more than 35 days, after discontinuation of treatment
- Physical Examination: Includes an examination of major body systems, assessment of ECOG performance status, and weight. During the treatment period, the frequency of physical exam will be according to local clinical practice, but not less than every 12 weeks (£2 weeks).

  Blood pressure, pulse rate: Blood pressure and pulse rate should be taken with the patient in the seated position after the patient has been sitting quietly for at least 5 minutes. Two blood pressure readings will be taken at least 1 hour apart at each clinic visit. During the treatment period, the equency of blood pressure collection will be according to local clinical practice, but not less than every 12 weeks (±2 weeks).
- Home blood pressure monitoring, pulse rate: when patients are registered, they will receive home blood pressure monitoring devices to monitor blood pressure and pulse at home. Patients taking axitinib will monitor their blood pressure at least twice daily (before taking each dose of axitinib) and blood pressure should be recorded in a patient diary. Patients should be instructed to contact the site immediately for goidance if their systolic blood pressure rases above 100 mm Hg, or if they develop symptoms perseved to be related to elevated blood pressure (e.g., headache, visual disturbance) although a different blood pressure threshold for contacting the site may be used according to the Investigator's clinical judgment (see Section 5.3.2.5). It's also important to counsel patients about the risk of bradyoardis and inform them of what symptoms and siters to be aware of and actions to take.
- symptoms and signs to be aware of and actions to take.

  Ophthalmologic Examination: Includes visual acuty fundoscopy, and slit lamp and should be performed by an ophthalmologist. The ophthalmologic examination should be repeated during the study when AE vision disorders are first observed or worsen from previous visit (see Section 71.6).

  Hematology, Blood Chemistry, and Coagulation: Required tests are listed in Table 6. During the treatment period, the frequency of hematology,
- blood chemistry and coagulation tests will be according to local clinical practice, but not less than every 12 weeks (±2 weeks). Liver function tests (LFTs) (including transaminases and total bilirubin) have to be monitored once per cycle and as clinically indicated. LFTs should be measured more frequently in the event of Grade 2-4 elevations or signs or symptoms consistent with hepatotoxicity.

AG-013736, PF-02341066-A4061068 Final Protocol Amendment 3, 09 June 2017

- Urinalysis (Table 6): If protein ≥2+ by semiquantitative method (eg. urine dipstick), protein will have to be quantified by 24 hour urine collection. Dose adjustment may be required (see Section 5.3 2.2). Urine reflex microscopy is required whenever urine multitest dipstick is positive for blood or protein. During the treatment period, the frequency of urine analysis will be according to local clinical practice, but not less than every 12 weeks
- 10 12-lead ECG: See Section 7.1.5 for details. Triplicate ECG measurements will be measured at the time of End of Treatment/Withdrawa
- approximately 2 minutes apart. If the mean QTc interval is prolonged (:501 msec), then the ECG should be read by a cardiologist at the site for confirmation. Additional ECGs will be performed as clinically indicated.

  11. Thyroid function tests: from Cycle 6 Day 1 TSH should be repeated as clinically indicated, and according to local clinical practice, but not less than every 12 weeks ( #2 weeks). Free T3 and free T4 should be performed when clinically indicated. Hypothyroidism should be treated per standard.
- medical practice to maintain cuthyroid state.

  1.2. Contraceptive Check: Male patients who are able to father children and female patients who are of childbearing potential will need to affirm that they meet the criteria for correct use of 2 of the selected methods of contraception. The investigator of his or her designee will discuss with the patient the need to use 2 highly effective contraception methods consistently and correctly and document such conversation in the patient's chart. In addition, the investigator or his or her designee will instruct the patient to call immediately if one or both selected contraception methods are disco
- investigator or his or her designee will instruct the patient to call immediately if one or both selected contraception methods are discontinued, or if pregnancy is known or suspected in the patient or partner.

  13. Tumor Assessments: Tumor assessments will include all known or suspected disease sites. Imaging may include chest, abdomen and pelvis CT or MRI seans, brain CT or MRI sean for patients with suspected brain metastases. The CT soans should be performed with contrast agents unless contramidicated for medical reasons. The same imaging technique used to characterize each identified and reported lesion at baseline will be employed in the following tumor assessments. Antitumor activity will be assessed through radiological tumor assessments conducted at baseline, and then according to local clinical practice, but not less than every 12 weeks (£2 weeks), whenever disease progression is suspected (eg. symptomatic deterioration), and at the time of End of Treatment/Withdrawal (if not done in the previous 12 weeks). For patients with known or suspected bone metastases as bone scan (bone scintigraphy) or "F-FDG-PET CT is required any if new bone metastases are suspected. Bone imaging is also required at the time of confirmation of response for patients who have bone metastases. Assessment of mead using RE/CTST version 1.

  14. Adverse Events: Adverse events should be documented and recorded at each visit using NCI CTCAE version 4.03. The AE reporting period begins from the time that the patient provides informed consent through and including 28 calendar days after the last investigational product administration. SAEs experienced by a patient after the active reporting period has ended should be reported to the Sponsor if the Investigation becomes aware of them;
- SAEs experienced by a patient after the active reporting period has ended should be reported to the Sponsor if the Investigator becomes aware of them, at a minimum, all SAEs that the Investigator believes have at least a reasonable possibility of being related to investigational product are to be reported to the Sponsor. AEs (serious and non serious) should be recorded on the Case Report Form (CRF) from the time the patient has taken at least one dose of study treatment through last patient visit (Day 28 after last dose). If a patient begins a new anticancer therapy, the AE reporting period for non
- serious AEs ends at the time the new treatment is started.

  15. Concomitant Medications/Treatments: Concomitant medications and treatments will be recorded from 28 days prior to the start of study treatment and up to 28 days after the last dose of study treatment. All concomitant medications should be recorded in the CRF including supportive care drugs (eg. anti-emetic treatment and prophylaxis), and the drugs used to treat adverse events or chronic diseases, and non-drug supportive interventions
- Study Treatment: Axitinib and crizotinib will be given twice daily PO on a continuous schedule Acutuib in combination with crizotinib will be given every 28 days (28 days = 1 cycle) (see Section 5)

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 1. INTRODUCTION

#### 1.1. Indication

Axitinib in combination with crizotinib is indicated for the treatment of advanced solid tumors (Dose Escalation Phase) and de novo or VEGF inhibitor pretreated advanced renal cell cancer (RCC) patients (Dose Expansion Phase).

#### 1.2. Background and Rationale

#### 1.2.1. Tumor Angiogenesis and VEGF-Pathway Inhibition

Tumor angiogenesis is a complex dynamic process necessary for the continued growth of solid tumors. VEGF is one of the most important angiogenic factors secreted by the tumor and other cells. Its production is enhanced by several stimuli, including hypoxia. VEGF and VEGF receptors (VEGFRs) are critical components of the processes leading to the branching, extension, and survival of endothelial cells which form new blood vessels during angiogenesis, and which is an absolute necessity for tumor growth beyond microscopic size. Inhibitors of angiogenesis are now widely used in the treatment of cancer and most of these agents inhibit the VEGF pathway. VEGF inhibitors include the VEGFR TKIs axitinib, sumitinib, pazopanib, and sorafenib, and the monoclonal anti-VEGF antibody bevacizumab. VEGF inhibitors have been approved in a number of indications, including the treatment of RCC. <sup>1,2</sup>

#### 1.2.2. Renal Cell Cancer

An estimated 65,150 new cases of kidney cancer are expected to be diagnosed in the United States of America (US) in 2013. This includes 93% RCC, 6% renal pelvis cancer and 1% Wilms tumor. An estimated 13,680 patients will die from kidney cancer in 2013.

RCC arises from the renal epithelium and 5 major subtypes are currently recognized. Approximately 70-80% of these are clear cell RCC tumors while other less common cell types include papillary (Type I and II), chromophobe, collecting duct and unclassified RCC. Four RCC predisposing genes have been identified – MET protooncogene, von Hippel-Lindau tumor suppressor gene (VHL), fumarate hydratase tumor suppressor gene (FH), and Birt-Hogg-Dubé tumor suppressor gene (BHD).

Patients with von Hippel-Lindau disease have a >70% risk of developing clear cell RCC. This hereditary form of RCC is caused by germline mutations in the VHL tumor suppressor gene on chromosome 3p. More than 90% of sporadic clear cell RCC involves somatic VHL gene mutations or methylation. VHL gene mutations lead to loss of function of the VHL protein, accumulation of hypoxia-inducible transcription factors (eg., HIF-1alpha and HIF-2 alpha) which translocate to the nucleus and increase transcription of angiogenesis factors (such as VEGF and platelet derived growth factor (PDGF)) which induce tumorgenesis. Clear cell RCC is a highly vascular tumor with high expression of VEGF. VEGFRs and PDGF receptor. §

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

About one-third of patients with clear cell RCC present with Stage IV disease. Systemic therapy is given to patients with advanced disease (relapsed or Stage IV) that is not amenable to complete resection. However, it is recommended that these patients undergo a cytoreductive nephrectomy where possible, prior to beginning systemic therapy, as per treatment guidelines.<sup>6</sup>

There are 10 targeted agents approved in the US as systemic therapy for advanced RCC that is predominantly clear cell. First line systemic therapy is usually one of the VEGFR TKIs (sunitinib, pazopanib, or sorafenib), or the monoclonal anti-VEGF antibody bevacizumab (given in combination with interferon alfa) or the mTOR inhibitor, temsirolimus. The same targeted agents, or axitinib (VEGFR TKI), everolimus (mTOR inhibitor), cabozantinib (inhibitor of VEGFRs, mesenchymal-epithelial transition factor [MET], and AXL), nivolumab (monoclonal antibody specific for programmed death-1 [PD-1]), or lenvatinib (VEGFR TKI) in combination with everolimus, are used individually in subsequent lines of therapy for advanced clear cell RCC. <sup>6,7,8,9</sup>

#### 1.2.3. Rationale

#### 1.2.3.1. c-MET and Resistance to Antiangiogenic Therapy

Despite the success of antiangiogenic therapy in multiple treatment settings including RCC, a fraction of patients are refractory to VEGF inhibitor treatment and the majority of patients will eventually develop resistance and exhibit disease progression while on therapeutic regimen. Nonclinical studies suggest that anti-angiogenic therapy may have induced the tumor to be more aggressive. And Models show VEGF inhibitor-resistant tumors to be more locally invasive and exhibit enhanced distant metastases. Several mechanisms have been proposed to explain resistance and this increase in tumor aggressiveness. These include activation of pathways that favor epithelial-mesenchymal transition (EMT) such as c-MET; a switch to vasculogenesis; co-option of normal organ vasculature; blood flow alterations due to tumor vessel pruning and normalization; and changes in the dominant VEGF isoform.

Another proposed tumor resistance mechanism involves a switch from VEGF to alternative proangiogenic mediators such as HGF and PDGF. According to this hypothesis, antiangiogenic therapies normalize and reduce tumor vascularization and increase tumor hypoxia. Hypoxia and the overexpression of HIF-1 leads not only to the accumulation of VEGF and PDGF, but also increases HGF expression in tumor and surrounding normal interstitial cells and increases c-MET receptor expression in endothelial and tumor cells. The HGF/c-MET pathway and VEGFR pathway can act synergistically to promote tumor survival. Additionally, HGF has its own role as an independent angiogenic factor and so may substitute, at least in part, for VEGF. Up-regulation of HGF/c-MET signaling increases tumor invasiveness and distant metastasis. <sup>15,16,17</sup>

Nonclinical models support a role for HGF/c-MET in VEGF inhibitor resistance.<sup>17,18</sup> In several tumor models resistant to the VEGF TKI sunitinib, a combination of sunitinib plus the c-MET inhibitor PF-04217903 inhibited tumor growth to a greater degree compared to either inhibitor alone.<sup>19</sup> A similar synergistic action was seen in a later study using sunitinib combined with the c-MET inhibitor crizotinib in both breast and colorectal orthotopic tumor

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

models resistant to sunitinib. Histological analysis suggested that combination treatment mainly targeted the vasculature in resistant tumors. Moreover, exogenous HGF conferred resistance to sunitinib. In a pancreatic neuroendocrine RIP-TAG-2 model, sunitinib increased hypoxia, expression of HIF-1alpha, c-MET, and markers of EMT. Importantly, invasion and metastasis were prevented when sunitinib was accompanied by concurrent administration of one of the c-MET inhibitors PF-4217903 or crizotinib. A similar benefit was found in orthotopic pancreatic carcinomas treated with cabozantinib (XL184), a receptor TKI that blocks both c-MET and VEGFR2. Cabozantinib prevented or reversed invasiveness, reduced the number and size of liver metastases, and prolonged survival.

There has been a report of axitinib in combination with crizotinib in two RCC nonclinical models. Human high cMET expressing 786-O and low cMET expressing RP-01 xenograft tumors were treated with vehicle, axitinib, crizotinib, or axitinib combined with crizotinib. Significant synergistic effects were found with crizotinib combined with axitinib with tumor inhibition reported as 17% with axitinib alone compared to 76% with the combination (P<0.05).<sup>23</sup>

Taken together, nonclinical data indicate that resistance to VEGF inhibitors is accompanied by intratumoral hypoxia, activation of HIF-1 alpha, an increase in c-MET activity, and EMT. Inhibition of cMET and VEGFR together has synergistic effects on tumor growth, angiogenesis, invasiveness, and metastasis in a number of models. <sup>17,18,19,20,21,22,23</sup> The recently reported synergistic effect between axitinib and crizotinib further suggests that dual targeting of c-MET and VEGF pathways may be effective in RCC. <sup>23</sup>

Further support for combining a VEGFR inhibitor with a c-MET inhibitor comes from the observed clinical activity of cabozantinib. Cabozantinib has demonstrated broad clinical activity in multiple tumor types including medullary thyroid cancer, breast, ovarian, prostate and lung cancers, melanoma, glioblastoma, hepatocellular carcinoma and RCC. A Phase 2 study in 171 patients with castration-resistant prostate cancer (CRPC) reported that 72% of evaluable patients had shrinkage of soft tissue lesions whereas 68% had an improvement on bone scan. The objective response rate (ORR) at 12 weeks was 5% and there was stable disease (SD) in 75% of patients. The observed effects on bone scan are unprecedented and not seen with single agent VEGF-pathway targeted therapy, this suggests that dual targeting of both VEGF and c-MET pathways may lead to improved outcome for patients with CRPC. 25

Clinical activity of cabozantinib in advanced pretreated RCC has been noted in a Phase I trial and confirmed in the METEOR trial, a randomized Phase 3 trial of cabozantinib versus everolimus in patients with renal cell carcinoma that had progressed after VEGFR-targeted therapy. <sup>26,42</sup> Progression-free survival (PFS) was longer with cabozantinib than with everolimus, with median PFS 7.4 months with cabozantinib and 3.8 months with everolimus. The risk of progression or death was 42% lower with cabozantinib than with everolimus (hazard ratio, 0.58; 95% confidence interval [CI] 0.45 to 0.75; P<0.001). The ORR was 21% with cabozantinib and 5% with everolimus (P<0.001). A planned interim analysis showed that overall survival (OS) was longer with cabozantinib than with everolimus (hazard

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

ratio for death, 0.67; 95% CI, 0.51 to 0.89; P = 0.005) but did not cross the significance boundary for the interim analysis.<sup>42</sup>

In conclusion, dual targeting of VEGF and c-MET pathways demonstrates significant clinical activity in a number of cancers including RCC. This is consistent with the nonclinical data supporting a role for c-MET in resistance to VEGFR targeted therapy and demonstration of synergy between VEGF pathway inhibition and c-MET inhibition in several models including axitinib in combination with crizotinib in RCC.

#### 1.2.3.2. Hypothesis to be Tested

The above clinical and nonclinical data support the hypothesis that c-MET signaling contributes significantly to VEGF inhibitor resistance such that combining a c-MET inhibitor with a VEGFR inhibitor will provide clinical benefit compared to treatment with a VEGF pathway directed therapy alone.

This supports the testing of crizotinib, as c-MET inhibitor, in combination with the VEGFR inhibitor axitinib. Since this will be the first study of axitinib given in combination with crizotinib, the primary objective of the study will be the assessment of the safety and tolerability of the combination regimen. However, once the tolerability of the combination has been confirmed, its antitumor activity will be preliminarly assessed in advanced RCC expansion cohorts in both the first line setting, and second/third line setting following disease progression on a VEGF pathway inhibitor. This will explore the activity of the combination in both preempting the development of resistance to VEGF pathway inhibitor and in treating tumors already resistant to VEGF pathway inhibitor.

### 1.2.4. Study Drugs

### 1.2.4.1. Crizotinib (XALKORI®, PF-02341066) as a c-MET Inhibitor

Crizotinib (XALKORI®, PF-02341066) is indicated for the treatment of anaplastic lymphoma kinase (ALK)-positive advanced non-small cell lung cancer (NSCLC), and for the treatment of ROS1-positive metastatic NSCLC (actual indication varies according to region/country).<sup>27</sup>

Although, crizotinib is a selective ATP-competitive small-molecule, oral ALK/ROS1 TK1 with proven clinical activity in ALK-positive NSCLC patients, it is also an inhibitor of c-MET and its oncogenic variants (eg. c-MET/HGFR mutations). <sup>28,29</sup> Crizotinib demonstrated potent (inhibition constant [K<sub>i</sub>] in nM range) concentration-dependent inhibition of c-MET phosphorylation in biochemical kinase assays and cell-based assays using tumor cell lines. <sup>29</sup> Crizotinib also demonstrated antitumor efficacy, including marked cytoreductive antitumor activity, in multiple tumor models implanted in athymic mice that expressed activated crizotinib targets including c-MET/HGF. In all assays, crizotinib was found to be at least as potent, if not more potent, an inhibitor of c-MET compared to ALK. Since clinical studies have demonstrated that crizotinib has activity against ALK, this implies that the level of drug attainable in human plasma would be sufficient enough to also inhibit c-MET.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Clinical evidence for crizotinib inhibition of c-MET comes from the Phase 1 clinical trial (A8081001).<sup>79</sup> Crizotinib has shown pharmacodynamic modulation (increase) of soluble MET (sMET), which is a c-MET pathway-specific plasma biomarker. The increase was time-dependent. These observations are consistent with the effects reported for other c-MET inhibitors including foretinib (XL880) and rilotumumab (AMG102).<sup>30</sup>

In addition, antitumor activity has been seen in a number of patients with amplification in the cMET gene locus detected by FISH (MET/CEP7  $\geq$ 2.2). Two of 4 patients having gastroesophageal cancer with MET amplification (MET/CEP7  $\geq$ 5) experienced tumor shrinkage of -30% (confirmed PR<sub>2</sub>) and -16% when treated with crizotinib and PFS was 3.7 and 3.5 months, respectively. A patient with ALK negative, c-MET amplified (MET/CEP7  $\geq$ 5) non-small cell lung cancer (NSCLC) experienced a tumor shrinkage of -54% (confirmed PR) and a durable response of 10+ months when treated with crizotinib. A patient with glioblastoma multiforme (MET/CEP7 = 2.8), previously treated with the pan-VEGF inhibitor cediranib, had SD for 6+ months associated with significant tumor shrinkage (-40% by MacDonald criteria) when treated with crizotinib. A

Taken together, the nonclinical and clinical data support crizotinib as a potent inhibitor of c-MET and further clinical investigation of this activity is warranted.

Among the 2071 patients with NSCLC treated with single-agent crizotinib 250 mg BID, the most commonly reported treatment-related adverse events (AEs) of any severity grade (reported by ≥20% of patients) in decreasing frequency were VISION DISORDER, Diarrhoea, Nausea, Vomiting, OEDEMA, ELEVATED TRANSAMINASES, Constipation, and NEUTROPENIA (event terms written in ALL CAPITALS represent CLUSTERED TERMS which included multiple preferred terms). Among the 172 patients with NSCLC treated with single-agent crizotinib 250 mg BID in the randomized Phase 3 study comparing crizotinib to standard of care chemotherapy (pemetrexed or docetaxel), the most common crizotinib-related AEs (reported in ≥20% of patients) of any severity in decreasing frequency were VISION DISORDER, Diarrhoea, Nausea, Vomiting, ELEVATED TRANSAMINASES, Constipation, OEDEMA, NEUTROPENIA, Dysgeusia, Decreased appetite, and LEUKOPENIA. Among the 275 patients with NSCLC treated with single-agent crizotinib 250 mg BID in the randomized Phase 3 studies comparing crizotinib to standard of care chemotherapy (pemetrexed/cisplatin or pemetrexed/carboplatin), the most common crizotinib-related AEs (reported in ≥20% of patients) of any severity in decreasing frequency were VISION DISORDER, Diarrhoea, ELEVATED TRANSAMINASES, Nausea, Vomiting, OEDEMA, NEUTROPENIA, Constipation, Decreased appetite, and LEUKOPENIA. The safety profile observed for 159 patients with tumor types other than NSCLC treated with single-agent crizotinib 250 mg BID was similar to that of patients with advanced NSCLC. The most common treatment-related AEs (reported in ≥20% of patients) of any severity grade in decreasing frequencies were Nausea, VISION DISORDER, Vomiting, Diarrhoea, and Fatigue.

Additional information for crizotinib may be found in the Single Reference Safety Document (SRSD), which for this study is the Investigator Brochure. <sup>29</sup> Further information may be found in the crizotinib United States Package Insert (USPI). <sup>34</sup>

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 1.2.4.2. Axitinib (INLYTA®, AG-013736)

Axitinib (INLYTA®, AG-013736) is an oral, small molecule, TKI selective for VEGFRs 1, 2 and 3 and is approved for the treatment of advanced RCC after failure of one prior systemic therapy (actual indication varies according to region/country).

Axitinib is an adenosine triphosphate (ATP)-competitive inhibitor that binds to the unphosphorylated (non-activated) "DFG-out" conformation of the catalytic domain of a receptor tyrosine kinase. In enzymatic assays, axitinib was found to be highly potent (K<sub>i</sub> = 28 picomolar) against the kinase activity of juxta-membrane (JM) domain containing human VEGFR 2 recombinant protein.<sup>35</sup> In additional kinase assays, axitinib showed potent and ATP-competitive inhibition of the VEGFRs 1, 2, and 3 and PDGFR-β, but not other closely-related family kinases. Receptor binding studies and cell-based assays, confirmed that axitinib is a potent and selective inhibitor of VEGFRs 1, 2, and 3. Axitinib was shown to have antiangiogenic activity in a number of models including spontaneous pancreatic islet-cell tumors of RIP-TAG-2 transgenic mice model and demonstrated antitumor efficacy including marked cytoreductive antitumor activity, in multiple tumor models implanted in athymic mice.

The safety and efficacy of axitinib were evaluated in a randomized, open-label, multi-center Phase 3 study. Patients with advanced RCC (99% clear cell) whose disease had progressed on or after treatment with 1 prior systemic therapy, including sunitinib-, bevacizumab-, temsirolimus-, or cytokine-containing regimens were randomized to receive axitinib (N=361) or sorafenib (N=362). There was a statistically significant advantage for axitinib over sorafenib for the primary PFS endpoint, 6.7 (95% CI: 6.3, 8.6) vs 4.7 (95% CI: 4.6, 5.6) months respectively (p <0.0001). There was no statistically significant difference between the treatment arms in the secondary overall survival (OS) endpoint, 20.1 (95% CI: 16.7, 23.4) vs 19.2 (95% CI: 17.5, 22.3). The objective response rate (ORR) was 19.4% (95% CI: 15.4, 23.9) for axitinib and 9.4% (95% CI: 6.6, 12.9) for sorafenib. The most common (≥20%) adverse reactions observed in this study following treatment with axitinib were diarrhea (55%), hypertension (40%), fatigue (39%), decreased appetite (34%), nausea (32%), dysphonia (31%), palmar-plantar crythrodysesthesia (hand-foot) syndrome (27%), weight decreased (25%), vomiting (24%), asthenia (21%), and constipation (20%).

Overall, the adverse events reported for axitinib in clinical studies are considered manageable, generally reversible and expected for this class of agents. For single-agent axitinib 98% (1445/1474) of subjects reported at least one AE. The most common treatment-emergent all-causality AEs reported were: diarrhoea 55.0%, hypertension 51,0%, fatigue 47.1%, decreased appetite 40.0%, nausea 32.6%, weight decreased 32.2%, dysphonia 31.1%, palmar-plantar erythrodysaesthesia syndrome 29.4%, hypothyroidism and vomiting 22.6%, constipation 20.3%, proteinuria 20.1%.

Additional information for axitinib may be found in the SRSD, which for this study is the Investigator Brochure. 35 Further information may be found in the axitinib USPL 36

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 1.2.5. Rationale for Starting Doses of Axitinib and Crizotinib

Nonclinical and clinical pharmacokinetic (PK) data for crizotinib are reported in the crizotinib Investigator's Brochure. <sup>29</sup> In nonclinical studies pharmacokinetic/pharmacodynamic (PK/PD) analyses for inhibition of c-MET/HGFR activity established a targeted efficacious concentration (C<sub>eff</sub>) range of 40 to 62 ng/mL (8.1 to 12.8 nM, free drug). In clinical studies, repeated oral administration of crizotinib at 250 mg BID for 15 days or longer resulted in a median trough plasma concentration of 274 ng/mL (57 nM, free drug). The RP2D and approved dose in ALK-positive patients is 250 mg BID. <sup>29,34</sup> Based on simulations, 250 mg every day (QD), 200 mg BID and 250 mg BID doses of crizotinib are expected to yield trough plasma concentrations exceeding crizotinib's Ceff for c-MET. In consideration of safety, the axitinib plus crizotinib combination will be first tested using a crizotinib starting dose of 200 mg BID (RP2D-1). The target crizotinib dose in the combination will be the currently approved dose of 250 mg BID. Dose de-escalation to crizotinib 250 mg QD will be allowed in the event of toxicity. Dose escalation and de-escalation will be based on DLTs.

The currently approved starting dose for axitinib is 5 mg PO BID. 35 Clinical PK data for crizotinib indicate that crizotinib is a moderate time-dependent cytochrome P450 (CYP) 3A4/5 inhibitor. 29 Axitinib is primarily metabolized by CYP3A4/5 as evidenced by a 2-fold increase in axitinib plasma exposures noted in the presence of the strong CYP3A4/5 inhibitor, ketoconazole. 35 Hence, there is a potential for increased axitinib exposure (by approximately 50%) in the presence of crizotinib. Considering this potential drug-drug interaction and the overlapping toxicities of axitinib and crizotinib (such as diarrhea, nausea, vomiting and fatigue), the starting dose of axitinib has been decreased to 3 mg PO BID for this study. Based on PK simulations, 3 mg PO BID axitinib in combination with crizotinib is predicted to provide similar plasma exposure to axitinib 5 mg PO BID alone (Figure 1). During the Dose Escalation Phase, the starting dose of axitinib may be increased to 5 mg BID or decreased to 2 mg BID in subsequent cohorts based on toxicity. Dose escalation and de-escalation will be based on DLTs. Axitinib is not expected to affect crizotinib exposure.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Figure 1. Pharmacokinetic Simulations Indicating the Predicted Increase in Exposure of Axitinib when Combined with Crizotinib



#### 1.3. Rationale for Protocol Amendment #3

The patient enrollment was completed as per protocol in the Escalation Phase of the study, with axitinib 5 mg twice/day (BID) plus crizotinib 250 mg BID established as the maximum tolerated dose (MTD), and also in the Expansion Phase Cohort 1 (no prior systemic therapy directed at advanced RCC).

As for Expansion phase Cohort 2 (at least one but no more than two prior systemic treatment regimens directed at advanced RCC), it was decided to discontinue the enrollment in this cohort due to the competitive landscape, that made the identification of eligible patients extremely challenging (7 patients were enrolled in Cohort 2 in about 1.5 years). Due to the small patient population and the decision to discontinue enrollment in Cohort 2, biomarker analyses will be performed only on Cohort 1.

As of 01 March 2017, 24 patients were enrolled (22 patients treated) in the dose Escalation Phase, at four dose levels: axitinib 3 mg BID + crizotinib 200 mg BID (n=5), axitinib 3 mg BID + crizotinib 250 mg BID (n=3), axitinib 5 mg BID + crizotinib 200 mg BID (n=4), and axitinib 5 mg BID + crizotinib 250 mg BID (n=10). There were no Cycle 1 dose-limiting toxicities and axitinib 5 mg BID + crizotinib 250 mg BID was established as the MTD. The most frequent all causalities adverse events (AEs) in the MTD group were fatigue (70%), nausea (70%), diarrhea (60%) and vomiting (50%), mainly of severity grade 1-2.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

In the Expansion Phase, 27 patients with advanced RCC have been treated at the MTD: 21 patients in Cohort 1, and 6 patients in Cohort 2 (one additional patient was enrolled in Cohort 2 on 6<sup>th</sup> March 2017, for a total of 7 patients, then the enrolment was discontinued in that cohort). The regimen has shown manageable toxicities in the two expansion cohorts, with diarrhea (63%), nausea (59%), dysphonia (44%), fatigue (44%) and vomiting (44%) as most frequent all causalities AEs. The response evaluation (as per Response Evaluation Criteria in Solid Tumors [RECIST] v1.1) is ongoing, with 4 partial responses (PR) in Cohort 1, and 1 PR in Cohort 2.

Overall, there are 11 patients (10 male and 1 female) currently continuing treatment in study a4061068, and they have received at least 5 treatment cycles. The main purpose of this amendment is to simplify the study procedures, where possible, for the patients on active study treatment.

During treatment on this protocol amendment, the patients will be evaluated for safety and for efficacy per local clinical practice, but not less than every 12 weeks (±2 weeks), except for liver function tests to be done at least every month. Axitinib and crizotinib dosing and concomitant treatments will be monitored, too. Follow up information will be collected until follow up visit (day 28 after the last study treatment dose). Pending drug availability, patients may continue to receive axitinib until they are no longer receiving clinical benefit according to the investigator's judgment.

#### 2. STUDY OBJECTIVES AND ENDPOINTS

### 2.1. Objectives

#### Primary Objective

To assess the safety and tolerability of axitinib in combination with crizotinib in
patients with solid tumors and advanced RCC in order to estimate the MTD (or MFD)
and select the RP2D.

### Secondary Objectives

- · To evaluate the overall safety profile.
- To characterize the PK of axitinib and crizotinib when administered in combination and to assess the effect of crizotinib on the PK of axitinib (Dose Escalation Phase and at least 8 PK-evaluable subjects in Dose Expansion Phase Cohort 1 only).
- · To characterize the effects of axitinib in combination with crizotinib on QTc.
- To document the anti-tumor activity of axitinib in combination with crizotinib in advanced RCC patients.
- To explore the pharmacodynamic effect of axitinib in combination with crizotinib in blood.
AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

> To characterize the alterations and/or expression profiles of genes, proteins, and RNAs relevant to angiogenesis (eg. Ang-2), drug targets (eg. c-MET) and sensitivity and/or resistance (eg. PBRM1) to axitinib in combination with crizotinib in tumor and/or blood.

### 2.2. Endpoints

### **Primary Endpoint**

· First-cycle DLTs,

### Secondary Endpoints

- Adverse events as characterized by type, frequency, severity (as graded by NCI Common Terminology Criteria for Adverse Events (CTCAE) v.4.03), timing, seriousness and relationship to study therapy.
- Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v.4.03) and timing.
- · Vital signs (blood pressure, pulse rate, weight, ECOG Performance Status [PS]).
- QTc interval.
- PK parameters of axitinib and crizotinib assuming steady state is achieved for both drugs: C<sub>max</sub>, T<sub>max</sub>, AUC<sub>0-12</sub>, CL/F and V<sub>z</sub>/F as data permit.
- Objective tumor response, as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.
- Time-to-event endpoints (Dose Expansion Phase Cohorts only): Duration of Response (DR) and PFS.
- Pre- and post-dose blood levels of plasma and serum biomarkers.
- Baseline and at progression plasma, serum and tumor tissue biomarkers (eg, c-MET, HGF).

### 3. STUDY DESIGN

#### 3.1. Study Overview

This is a Phase 1b, open-label, multi-center, multiple-dose, safety, PK and pharmacodynamic study of axitinib in combination with crizotinib in adult patients with advanced solid tumors.

This clinical study will be composed of two phases:

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Dose Escalation Phase: This phase will estimate the MTD in dose escalation cohorts in patients with advanced solid tumors. The modified toxicity probability interval (mTPI) method will be applied in the Dose Escalation.
- Dose Expansion Phase: This phase will confirm the safety and tolerability and explore the antitumor activity of axitinib in combination with crizotinib in two cohorts of patients with advanced RCC.

All patients will receive axitinib in combination with crizotinib in 28-day cycles.

To understand the PK effects of crizotinib on axitinib, a 7-day lead-in period of single-agent axitinib directly preceding the administration of the crizotinib and axitinib combination will be included prior to Cycle 1 in the Dose Escalation Phase of the study. Axitinib is not expected to affect crizotinib exposure so there will be no PK study with a lead-in period of single-agent crizotinib. The Dose Expansion Phase Cohort 1 will be used to further study crizotinib and axitinib pharmacokinetic interactions; in this cohort, the PK profile for axitinib single agent during the 7-day lead-in period will be compared to that of axitinib in combination with crizotinib during Cycle 1. Patients participating in serial PK sampling (all patients in the Dose Escalation Phase and at least 8 evaluable patients in Cohort 1 of the Dose Expansion Phase) need to receive at least 3 consecutive days of axitinib treatment prior to axitinib PK sample collection (on Lead-in Day 7 and Cycle 1 Day 15). If, for any reason, this is not feasible, the patient will be replaced. No lead-in period will be included in the Dose Expansion Cohort 2.

In all patients, treatment with investigational product will continue until either disease progression, patient refusal, patient lost to follow up, unacceptable toxicity, or the study is terminated by the Sponsor. Patients with unacceptable toxicity attributed to one of the two investigational products may be eligible for continued treatment with the other investigational product (after discussion between the Investigator and the Sponsor). Patients with disease progression but who are still experiencing clinical benefit will be eligible for continued treatment with single agent axitinib or axitinib combined with crizotinib provided that the treating physician has determined that the benefit/risk for doing so is favorable. Pending drug availability, patients may continue to receive axitinib until they are no longer receiving clinical benefit according to the investigator's judgment.

Given the safety profile of crizotinib, in addition to standard safety tests, ophthalmology examinations will be carried out to assess any vision changes. Based on the safety profile of axitinib, blood pressure will be monitored throughout the treatment period, as well as thyroid function.

ECG measurements will be taken throughout the treatment period in all patients and in conjunction with PK sampling in patients from the Dose Escalation Phase and the Dose Expansion Phase Cohort 1. Archived tumor tissues will be collected for all patients. De novo tumor biopsy will be collected for the patients in the Dose Expansion Phase Cohort 2. Biomarker studies on tumor tissue and blood will be carried out to help understand the mechanism of action of the axitinib plus crizotinib combination, as well as potential

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

mechanisms of resistance. Such results may help in the future development of this combination. These analyses may also result in the identification of potential biomarkers of response to the axitinib plus crizotinib combination, ultimately leading to development of a patient selection strategy for further clinical investigation.

Up to 65 patients are expected to be enrolled in the study.

#### 3.1.1. Dose Escalation Phase

### 3.1.1.1. Starting Doses for Axitinib and Crizotinib (Dose Level 1)

The rationale for the starting doses is given in Section 1.2.5. The starting doses (Dose Level 1) are axitinib 3 mg BID in combination with crizotinib 200 mg BID in 28-day cycles.

#### 3.1.1.2. DLT Observation Period

Patients will be monitored for the occurrence of DLTs. For dose escalation purposes, the DLT observation period is Cycle 1 (28 days).

Patients who discontinue treatment before completing the DLT observation period and who do not take at least 75% of the planned doses of both axitinib and crizotinib for reasons other than treatment related toxicity (for example, missed appointments, misplaced study drug supplies, development of rapidly progressing disease) will be replaced.

#### 3.1.1.3. Criteria for Dose Escalation

Dose escalation and de-escalation will follow a matrix. "Up-and-Down" design, using doses of crizotinib and axitinib as shown in Table 1.

Table 1. Dose Levels in Dose Escalation Phase

| Dose Level | Crizotinib | Axitinib |
|-----------------------|------------|----------|
| -1B | 250 mg QD | 3 mg BID |
| -1A | 200 mg BID | 2 mg BID |
| (Starting Dose Level) | 200 mg BID | 3 mg BID |
| 2A | 250 mg BID | 3 mg BID |
| 2B | 200 mg BID | 5 mg BID |
| 3 | 250 mg BID | 5 mg BID |

BID: twice daily; QD: once daily

The proposed doses, schedule(s) and PK timepoints may be reconsidered and amended during the study based on the emerging safety and pharmacokinetic data.

In this dosing algorithm there are up to 6 potential dose levels: (-1B) crizotinib 250 mg QD + axitinib 3 mg BID; (-1A) crizotinib 200 mg BID + axitinib 2 mg BID; (1) crizotinib 200 mg BID + axitinib 3 mg BID; (2A) crizotinib 250 mg BID + axitinib 3 mg BID; (2B) crizotinib 200 mg BID + axitinib 5 mg BID and (3) crizotinib 250 mg BID + axitinib 5 mg BID.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

The matrix approach allows for parallel dose cohorts exploration as escalations and de-escalations are called for based upon toxicity results. Possible dose escalation/de-escalation scenarios based on the starting (1) dose level tolerability are illustrated in Figure 2.

Figure 2. Possible Scenarios for Dose Escalation/De-escalation Based on Dose Level Tolerability



The arrows represent either dose de-escalation (red arrow) or dose escalation (green arrows).

During the course of the study, only 1 investigational product (crizotinib or axitinib, but not both) can be dose escalated or de-escalated in the next cohort.

There are several potential dosing sequences for escalation or de-escalation of crizotinib + axitinib. The specific sequence to be followed depends upon the number of patients enrolled in the study and the number of DLTs observed at each specific dose combination. The sequences are mutually exclusive, meaning only one of the sequences will be followed through the course of the study. Some possible sequences are listed below in Table 2.

Table 2. Possible Dose-Finding Sequences

| Dose 1 meets escalation criteria in the initially enrolled cohort | Dose 1 meets de-escalation criteria in the<br>initially enrolled cohort |
|---|---|
| $1 \rightarrow (2A, 2B) \rightarrow 3$ | $1 \rightarrow (-1A, -1B) \rightarrow 1 \rightarrow (2A, 2B) \rightarrow 3$ |
| $1 \rightarrow (2A, 2B)$ | $1 \rightarrow (-1A, -1B) \rightarrow 1 \rightarrow (2A, 2B)$ |
| $1 \rightarrow (2A, 2B) \rightarrow 3 \rightarrow (2A, 2B)$ | $1 \rightarrow (-1A, -1B) \rightarrow 1$ |
| $1 \rightarrow (2A, 2B) \rightarrow 3 \rightarrow (2A, 2B) \rightarrow 1$ | 1 → (-1A, -1B) |
| $1 \rightarrow (2A, 2B) \rightarrow 3 \rightarrow (2A, 2B) \rightarrow 1 \rightarrow (-1A, -1B)$ | |

Dosing will begin at Dose Level 1 and escalated or de-escalated according to Table 1. The escalation/de-escalation rules will follow the mTPI method<sup>38</sup> (see Section 9.2 and Appendix 5). Briefly, the mTPI method relies upon a statistical probability algorithm, calculated using all patients treated in prior and current cohorts at the same dose level to

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

determine where future cohorts should involve dose escalation, no change in dose, or dose de-escalation. As an example, if the total number of patients (cumulative in the study from prior and current cohorts) treated at the current dose combination is 3 the following dosing rules are applied:

- 0 DLT → escalate;
- 1 DLTs → remain at the same dose;
- 2 DLTs → de-escalate;
- 3 DLTs → de-escalate and consider current dose as intolerable.

Rules for dose-finding, using the mTPI method, include the following:

- The target enrollment cohort size is 3 patients. The first 3 patients treated in Dose Level 1 cohort will initiate dosing sequentially, at least 2 days apart to allow for the initial evaluation of toxicities and tolerability. If there are no safety concerns, any additional patients enrolled to this dose cohort will not be required to initiate dosing sequentially.
- The next cohort can be enrolled when all patients at the current dose cohort have been
  evaluated for 28 days of the first treatment cycle, or experience a dose limiting
  toxicity (DLT), whichever comes first.
- If a patient withdraws from the study before receiving at least 75% of the planned first-cycle dose of both axitinib and crizotinib for reasons other than study drug-related toxicity, another patient will be enrolled to replace that patient at the current dose level.
- The dose-finding component of the trial is completed when at least 10 evaluable
  patients have been treated at the highest dose associated with DLT rate <0.33. It is
  estimated that approximately 25 DLT evaluable patients will need to be enrolled to
  reach 10 DLT-evaluable patients at the estimated MTD.</li>
- The proposed doses, schedule, and PK timepoints may be reconsidered and amended during the study based on the emerging safety and pharmacokinetic data.
- The RP2D will be confirmed in the Dose Expansion Phase, taking into account the MTD/MFD determination from the Dose Escalation Phase, and other factors related to safety, efficacy, and PK/PD involving all available data from tests cohorts.

No intra-patient dose escalation will be permitted in the Dose Escalation Phase.

Once an MTD/MFD has been identified at the end of the Dose Escalation Phase, that dose level may be expanded with up to additional 10 patients patients to allow the collection of additional PK and/or safety data.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 3.1.2. DLT Definition

Severity of adverse events will be graded according to NCI CTCAE version 4.03 (See Appendix 3). For the purpose of Dose Escalation, any of the following adverse events occurring during the DLT observation period (Cycle 1), that are attributable to one, the other, or both agents in the combination will be classified as DLTs:

- · Hematologic;
  - Grade 4 neutropenia.
  - Febrile neutropenia, defined as absolute neutrophil count (ANC) <1000/mm<sup>3</sup> with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of ≥38 degrees C (100.4 degrees F) for more than one hour.
    - Grade ≥3 neutropenic infection.
  - Grade ≥3 thrombocytopenia with bleeding.
  - Grade 4 thrombocytopenia.
- Non-hematologic:
  - Grade ≥3 toxicities (except asymptomatic hypophosphatemia, hyperuricemia without signs and symptoms of gout, and tumor lysis syndrome).
  - Nausea, vomiting or diarrhea must persist at Grade 3 or 4 despite maximal medical therapy.
  - Grade 3 hypertension will be considered a DLT if the event is persistent despite
    use of anti-hypertensive medications.
- In an asymptomatic patient, Grade 3 QTc prolongation (QTc ≥501 msec) will first
  require immediate repeat testing, re-evaluation by a qualified person, and correction
  of reversible causes such as electrolyte abnormalities or hypoxia for confirmation. If,
  after correction of any reversible causes, the Grade 3 QTc prolongation persists, then
  the event should be considered a DLT.
- Failure to deliver at least 75% of dose of each investigational product due to toxicities attributable to one or both investigational products.

### 3.1.3. Maximum Tolerated Dose Definition

The MTD estimate is the highest dose of axitinib and crizotinib associated with the occurrence of DLTs in <33% of DLT-evaluable patients (see Section 9.1).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 3.1.4. Dose Expansion Phase Test Dose

The Expansion Test Dose will be either the MTD or the MFD, ie, the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor.

#### 3.1.5. Dose Expansion Phase

The Dose Expansion Phase will test axitinib in combination with crizotinib in patients with advanced RCC who are at their first diagnosis (Cohort 1) or have recurred during or after a VEGF-pathway inhibitor containing regimen (Cohort 2).

All patients in the Dose Expansion Phase may be enrolled simultaneously. A total of up to 20 patients will be enrolled into each Dose Expansion Phase Cohort. PK samples will be collected from at least 8 evaluable patients in Dose Expansion Phase Cohort 1.

Further experience in the Dose Expansion Phase Cohorts may result in the need to explore a lower Expansion Test Dose in one or both populations. Only doses declared safe in the Dose Escalation Phase will be considered.

For axitinib, intra-patient dose escalation to higher doses may be permitted in Cycle 2 and beyond (see Section 5.3.2.1).

#### 3.2. Recommended Phase 2 Dose

The RP2D is the dose of axitinib and crizotinib in combination chosen for further study based on Phase 1 study results. If the MTD/MFD proves to be clinically feasible for long term administration in a reasonable number of patients, then this dose usually becomes the RP2D. Further experience with the MTD/MFD may result in a RP2D dose lower than the MTD/MFD.

#### 4. PATIENT ELIGIBILITY CRITERIA

This study can fulfill its objectives only if appropriate patients are enrolled. The following eligibility criteria are designed to select patients for whom participation in the study is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a particular patient is suitable for this protocol.

#### 4.1. Inclusion Criteria

Patient eligibility should be reviewed and documented by an appropriate member of the Investigator's study team before patients are included in the study.

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

- 1. Diagnosis:
  - a. Dose Escalation Phase:

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Histologically or cytologically confirmed diagnosis of advanced solid tumor that is resistant to standard therapy or for which no standard therapy is available.
- Mandatory archival tumor tissue (formalin-fixed, paraffin-embedded [FFPE] tissue block(s) from either initial diagnosis or recurrence or metastatic site, or at least 12 unbaked, unstained slides). In cases where archival tumor tissue is not available, a de novo biopsy must be obtained for this purpose.
- b. Dose Expansion Phase:
  - Histologically or cytologically confirmed advanced RCC with a component of clear cell subtype, and:
    - · Cohort 1: no prior systemic therapy directed at advanced RCC; or
    - Cohort 2: at least one but no more than two prior systemic treatment regimens directed at advanced RCC, with at least one prior therapy being a regimen containing an approved VEGF-pathway inhibitor, and resistance to the most recently received approved VEGF-pathway inhibitor. Resistance is defined as disease progression as per RECIST version 1.1 while on treatment with a VEGF-pathway inhibitor.
  - Mandatory tumor tissue/biopsy collection:
    - Cohort 1 and Cohort 2: mandatory archival tumor tissue (FFPE tissue block(s) from initial diagnosis or at least 12 unbaked, unstained slides). In cases where archival tumor tissue is not available, a de novo biopsy must be obtained for this purpose.
    - Cohort 2 only: baseline de novo tumor biopsy collection. Alternatively, a recently obtained FFPE tumor tissue block from a resection or biopsy of a primary, recurrent or metastatic lesion can be provided if the following criteria are met: 1) the biopsy or resection was performed within 4 months of patient registration AND 2) the patient has not received any new intervening systemic anti-cancer treatment from the time the tissue was obtained and the patient registration.
  - At least one measureable lesion as defined by RECIST version 1.1.
- Age ≥18 years.
- 3. ECOG Performance Status 0 or 1 (see Appendix 1).
- 4. Adequate bone marrow function, including:
  - a. Absolute Neutrophil Count (ANC) ≥1,500/mm<sup>3</sup> or ≥1.5 x 10<sup>9</sup>/L;

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- b. Platelets  $\geq 100,000/\text{mm}^3$  or  $\geq 100 \times 10^9/\text{L}$ :
- e. Hemoglobin ≥9 g/dL.
- 5. Adequate renal function, including:
  - a. Serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥60 mL/min as calculated using the method standard for the institution and;
  - b. Urinary protein <2+ by urine dipstick. If dipstick is ≥2+, then a 24-hour urinary protein <2 g per 24 hours.</li>
- 6. Adequate liver function, including:
  - a. Total serum bilirubin ≤1.5 x ULN;
  - b. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (≤5.0 x ULN if there is tumor involvement in the liver);
- c. Alkaline phosphatase ≤2.5 x ULN; (≤5 x ULN in case of bone metastasis).
- 7. INR or prothrombin time (PT) <1.5 x ULN.
- If applicable, end of prior anticancer systemic treatment ≥2 weeks (≥4 weeks for bevacizumab + IFN) of patient registration, with resolution of all treatment-related toxicity to baseline severity or Grade ≤1 except for alopecia, hypothyroidism and other AEs not constituting a safety risk by Investigator judgment.
- No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure (BP) readings taken at least 1 hour apart. The baseline systolic BP readings must be ≤150 mm Hg, and the baseline diastolic BP readings must be ≤90 mm Hg.
- 10. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
- Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
- 12. Serum/urine pregnancy test (for females of childbearing potential) negative at screening and at the baseline visit (before the patient may receive the investigational product).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

13. Male patients able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use two highly effective methods of contraception throughout the study and for at least 90 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active.

#### 4.2. Exclusion Criteria

Patients presenting with any of the following will not be included in the study:

- Prior therapy with an agent that is known or proposed to be active by action on c-MET/HGF including but not limited to cabozantinib (XL184), foretinib (XL880), onartuzumab (MetMAb) and rilotumumab (AMG102).
- 2. Major surgery <4 weeks or radiation therapy <2 weeks of patient registration. Prior palliative radiotherapy (≤10 fractions) to metastatic lesion(s) is permitted, provided it has been completed 48 hours prior to the initiation of study medication and there is at least one measurable lesion that has not been irradiated (except patients in Dose Escalation Phase, who are not required to have any measurable lesion).</p>
- 3. Gastrointestinal abnormalities including:
  - · Inability to take oral medication;
  - · Requirement for intravenous alimentation;
  - Prior surgical procedures affecting absorption including total gastric resection;
  - · Treatment for active peptic ulcer disease in the past 6 months:
  - Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
  - Malabsorption syndromes.
- Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose
  anticoagulants for maintenance of patency of central venous access devise or
  prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular
  weight heparin is allowed.
- Evidence of inadequate wound healing, active bleeding disorder or other history of significant bleeding episodes within 30 days before study entry.
- Known, prior or suspected hypersensitivity to study drugs or any component in their formulations.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- History of or known active seizure disorder, brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
- 8. Any of the following within the 12 months prior to investigational product administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, or machine-read ECG with QTc interval ≥481 msec.
- Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
- 10. History of or known presence of extensive, disseminated/bilateral or Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, or pulmonary fibrosis, but not including a history of prior radiation pneumonitis.
- 11. Use of drugs or foods that are known strong CYP3A4/5 inhibitors within 7 days prior to the first dose of investigational product including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.
- 12. Use of drugs that are known strong CYP3A4/5 or CYP1A2 inducers within 12 days prior to the first dose of investigational product, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort.
- 13. Use of drugs that are CYP3A4/5 substrates with narrow therapeutic indices, including but not limited to dihydroergotamine, ergotamine, pimozide, astemizole\*, cisapride\*, and terfenadine\* (\* withdrawn from U.S. market).
- 14. Dose Expansion Phase only: diagnosis of any other malignancy within 2 years prior to registration, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix.
- 15. Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Pfizer employees directly involved in the conduct of the trial.
- 16. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- 17. Other severe acute or chronic medical (including severe gastrointestinal conditions such as diarrhea or ulcer) or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or end-stage renal disease on hemodialysis, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
- 18. Pregnant female patients, breastfeeding female patients, male patients with partners currently pregnant, male patients able to father children and female patients of childbearing potential who are unwilling or unable to use two highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after last dose of investigational product.

#### 4.3. Life Style Guidelines

#### 4.3.1. Sunlight Exposure

Patients will be advised to report any reaction to sun exposed skin. In addition, special precautions will be taken to limit any potential photo irritation effect, by minimizing the patients' exposure to light including high intensity ultraviolet B light (UVB) sources such as tanning beds, tanning booths and sunlamps. Patients should be encouraged to apply sunscreen/sunblock daily.

### 4.3.2. Contraception

In this study, male patients who are able to father children and female patients who are of childbearing potential will receive axitinib, which has been associated with teratogenic risk, in combination with crizotinib. Patients who are, in the opinion of the investigator, sexually active and at risk for pregnancy with their partner(s) must agree to use two (2) methods of highly effective contraception throughout the study and continue to do so for at least 90 days after the last dose of the investigational product. The Investigator or his or her designee, in consultation with the patient, will confirm that the patient has selected 2 appropriate methods of contraception for the individual patient and his or her partner(s) from the list of permitted contraception methods (see below) and will confirm that the patient has been instructed in their consistent and correct use. At time points indicated in the schedule of activities, the investigator or designee will inform the patient of the need to use 2 highly effective methods of contraception consistently and correctly and document the conversation, and the patient's affirmation, in the patient's chart. In addition, the Investigator or his or her designee will instruct the patient to call immediately if one or both selected contraception methods are discontinued or if pregnancy is known or suspected in the patient or partner.

Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (ie, perfect use) and include:

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Established use hormonal methods of contraception associated with inhibition of ovulation (eg, oral, inserted, injected, implanted or transdermal), provided the patient or male patient's female partner plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness.
- 2. Correctly placed copper containing intrauterine device (IUD).
- Male condom or female condom used WITH a spermicide (ic, foam, gel, film, cream, suppository). For countries where spermicide is not available or condom plus spermicide is not accepted as highly effective contraception, this option is not appropriate.
- 4. Male sterilization with absence of sperm in the post-vasectomy ejaculate.
- Bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed in accordance with the device's label).

Female subjects of non-childbearing potential must meet at least one of the following criteria:

- Have undergone a documented hysterectomy and/or bilateral oophorectomy;
- · Have medically confirmed ovarian failure; or
- Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state.

All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.

All sexually active male subjects must agree to prevent potential transfer to and exposure of partner(s) to drug through ejaculate by using a condom consistently and correctly, beginning with the first dose of investigational product and continuing for at least 90 days after the last dose of investigational product.

### 4.4. Sponsor Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the trial is documented in the study contact list located in the coordinator's manual.

To facilitate access to appropriately qualified medical personnel on study related medical questions or problems, patients are provided with a contact card. The contact card contains, at a minimum, protocol and investigational compound identifiers, patient study number, contact information for the investigational site and contact details for a help desk in the event that the investigational site staff cannot be reached to provide advice on a medical question

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

or problem originating from another healthcare professional not involved in the patients participation in the study. The help desk number can also be used by investigational staff if they are seeking advice on medical questions or problems, however it should only be used in the event that the established communication pathways between the investigational site and the study team are not available. It is therefore intended to augment, but not replace the established communication pathways between the investigational site and study team for advice on medical questions or problems that may arise during the study. The help desk number is not intended for use by the patient directly and if a patient calls that number they will be directed back to the investigational site.

#### 5. STUDY TREATMENTS

For the purposes of this study, and per International Conference on Harmonisation (ICH) guidelines investigational product is defined as a pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use (ICH E6 1.33).

For this study, the investigational product(s) are axitinib and crizotinib.

### 5.1. Allocation to Treatment

Dose level allocation will be performed by the Sponsor after patients have given their written informed consent and have completed the necessary baseline assessments.

The site staff will fax or e-mail a complete Registration Form to the designated Sponsor study team member(s) requesting approval for patient enrollment.

After review of patient's eligibility and concomitant medications, the Sponsor will approve patient's enrollment, if appropriate, and assign a patient identification number, which will be used on all Case Report Form (CRF) pages and other trial-related documentation or correspondence referencing that patient.

The Sponsor will fax or email the approved Registration Form reporting the patient identification number to the site.

No patient shall receive investigational product until the Investigator or designee has received the following information in writing from the Sponsor:

- · Confirmation of the patient's enrollment;
- · Specification of the dose level for that patient;
- Permission to proceed with dosing the patient.

The Sponsor or designee will notify the other sites of the inclusion of a new patient, and will inform study sites about the next possible enrollment date.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 5.2. Investigational Product Supplies

Axitinib (AG-013736) and crizotinib (PF-02341066) will be supplied for the study by the Global Clinical Supply, Worldwide Research and Development. Drug supplies will be shipped to the study sites with a Drug Shipment & Proof of Receipt form. This form should be completed, filed, and the shipment confirmed as directed on the bottom of the Drug Shipment & Proof of Receipt form.

### 5.2.1. Dosage Form(s) and Packaging

#### 5.2.1.1. Axitinib

Axitinib will be supplied for oral administration as 1 mg and 5 mg film-coated tablets in High Density Polyethylene (HDPE) bottles with desiccant.

#### 5.2.1.2. Crizotinib

Crizotinib will be supplied for oral administration as capsules containing 200 mg, or 250 mg of study medication and will be packaged in HDPE bottles.

#### 5.2.2. Preparation and Dispensing

Only qualified personnel who are familiar with procedures that minimize undue exposure to them and to the environment should undertake the preparation, handling, and safe disposal of chemotherapeutic agents.

Axitinib will be dispensed in opaque plastic bottles to protect the compounds from light. Axitinib is a hazardous drug (due to possible reproductive toxicity), and should be handled according to the recommended procedures described in the current edition of the American Society of Hospital Pharmacists (ASHP), Technical Assistance Bulletin on Handling Cytotoxic and Hazardous Drugs, American Hospital Formulary Service (AHFS) Drug Information (1999) and its references. Procedures described in each institution's pharmacy or hospital standard operating procedure manual should be followed when handling hazardous drugs.

Axitinib and crizotinib will be dispensed at the beginning of each treatment cycle (or as otherwise indicated). Patients should be instructed to keep their medication in the bottles provided and not transfer it to any other container. In the event of dose modification, a request should be made of the patient to return all previously dispensed medication to the clinic.

### 5.3. Administration

Axitinib and crizotinib will be each administered orally BID at approximately the same time in the morning and evening on a continuous daily dosing schedule, ie, without a break in dosing in the absence of drug-related toxicity (see Section 5.3.2.2). The two drugs can be taken together and the evening dose of each drug should be taken approximately 12 hours after the morning dose. Both drugs may be administered without regard to meals. Cycles are defined in 28-day periods to facilitate scheduling of visits and assessments. Capsules must not be opened or dissolved.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

A dosing card will be provided to the patients to provide guidance for the correct use of the two drugs.

Patients must be instructed that if they miss a dose or vomit anytime after taking a dose, they must not "make it up" with an extra dose, but instead resume subsequent doses as prescribed. Any missed dose may be taken late up to 3 hours for axitinib dose or up to 6 hours for crizotinib dose before the next scheduled dose, otherwise, it should be skipped and dosing resumed with subsequent doses as prescribed. Patient must be instructed to record all doses (and missed or vomited doses) in a dosing diary supplied by the site. If doses are missed or vomited, this must be indicated in the source documents and CRFs.

If a patient inadvertently takes 1 extra dose during a day, the patient should not take the next dose.

### 5.3.1. Food Requirements

Both axitinib and crizotinib can be taken with or without food. Avoid grapefruit or grapefruit juice which may increase plasma concentrations of axitinib and crizotinib.

#### 5.3.2. Recommended Dose Modifications

Axitinib and crizotinib dose levels for intra-patient dose modification are listed in Table 3 and Table 4, respectively.

Table 3. Axitinib Dose Levels

| Dose |
|-----------|
| 10 mg BID |
| 7 mg BID |
| 5 mg BID |
| 3 mg BID |
| 2 mg BID |

Table 4. Crizotinib Dose Levels

| Dose |
|------------|
| 250 mg BID |
| 200 mg BH) |
| 250 mg QD |

Intra-patient dose escalation is permitted in the Dose Expansion Phase only and for axitinib only.

### 5.3.2.1. Axitinib Intra-Patient Dose Escalation

Patients enrolled to either Dose Expansion Phase Cohort, who are in Cycle 2 or beyond, and who tolerate axitinib with no drug-related grade ≥3 adverse events for 2 consecutive weeks have the option to have their axitinib dose increased by one dose level in subsequent cycles as indicated in Table 3, up to a maximum dose of 10 mg BID (unless the patient's BP is >150/90 mm Hg or the patient is receiving antihypertensive medication). Since crizotinib may cause inhibition of axitinib metabolism, particular attention should be provided to a

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

patient's overall safety profile prior to implementing intra-patient dose escalation for axitinib. The Sponsor must be notified of the decision to increase the dose of axitinib.

#### 5.3.2.2. Dose Modifications in Case of Drug-Related Toxicity

Every effort should be made to administer investigational product on the planned dose and schedule.

In the event of significant toxicity dosing may be delayed and/or reduced as described below. In the event of multiple toxicities, dose modification should be based on the worst toxicity observed. Patients are to be instructed to notify Investigators at the first occurrence of any adverse symptom.

Dose modifications may occur in two ways:

- Within a cycle: dosing interruption until adequate recovery and dose reduction, if required, during a given treatment cycle.
- In the next cycle: dose reduction may be required in a subsequent cycle based on toxicity experienced in the previous cycle.

Investigators are encouraged to employ best supportive care according to local institutional clinical practices and according to the guidance for selected adverse events provided below.

Patients will be monitored closely for toxicity, and axitinib and/or crizotinib treatment may be adjusted by dosing interruption with or without dose reduction as indicated below. Dose modification can occur independently for the 2 drugs. Dosing interruption and/or intrapatient dose reduction by 1, and if needed, 2 doses will be allowed depending on the type and severity of toxicity encountered. If the patient is already at the lowest dose for one or the other study drug, the relevant study drug should be permanently discontinued. Management of patients requiring more than 2 dose reductions should be discussed with the Sponsor.

Dose modifications for toxicity can occur in both the Dose Escalation and Dose Expansion Phases. In the event of multiple toxicities, dose modification should be based on the worst toxicity observed. Toxicities should initially be attributed to either axitinib or crizotinib and managed accordingly.

Dosing CRFs should be utilized to document each time study medication is modified, started and stopped.

Recommended dose modifications in case of drug-related toxicity are shown in Table 5.

AG-013736, PF-02341066-A4061068 Final Protocol Amendment 3, 09 June 2017

### Table 5. Dose Modifications for Drug-Related Toxicity

| Toxicity | NCI CTCAE Severity Grade | Dose modifications |
|---|---|---|
| Hematologic | Grade 1 or Grade 2 | Axitinib: Continue at the same dose level. |
| Laboratory | | Crizotinih: Continue at the same dose level. |
| Investigations | Grade 3 | Axitinib. Continue at the same dose level. |
| | | Crizotinib: Withhold until recovery to Grade <2. Then, resume at the same dose level or reduce by 1 dose level as per Investigator judgement. Grade 3 lymphopenia not associated with clinical events, eg. opportunistic infection: study treatment may continue without interruption. |
| | Grade 4 | Axitinib: Withhold until recovery to Grade <2. Then, reduce by 1 dose level and resume treatment. Grade 4 lymphopenia not associated with clinical events, eg, opportunistic infection: study treatment may continue without interruption. |
| | | Crizolinib. Withhold until recovery to Grade ≤2. Then, reduce by 1 dose level and resume treatment as per Investigator judgement or after discussion with the Sponsor. Chade 4 lymphopenia not associated with clinical events, eg. opportunistic infection: study treatment may continue without interruption. |
| Non-hematologic | Grade 1 or Grade 2 | Axitinib: Continue at the same dose level. |
| Toxicites and or | The The Control of the Control of th | Crizotinib: Continue at the same dose level. |
| Laboratory<br>Abnormalities<br>(excluding exceptions<br>mentioned below) | Grade 3 | Axitinib: Reduce by 1 dose level. Grade 3 toxicities controlled with symptomatic medications, or Grade 3 asymptomatic biochemistry laboratory abnormalities, continue at the same dose level as per Investigator judgement. |
| | | Crizotinib: Withhold until recovery to Grade ≤1, or to baseline Grade. Then, resume at the same dose level or reduce by 1 dose level as per Investigator judgement. Grade 3 hypophosphatemis and/or hyperuricemia without clinical symptoms: study treatment may continue without interruption as per Investigator judgement. Persistent Grade 3 musea, vomiting or diarrhea despite maximal medical therapy reduce by 1 dose level. |
| | Grade 4 | Ashinib: Withhold current dose until recovery to Grade <2. Then, reduce by 1 dose level and resume freatment. Grade 4 asymptomatic blochemistry laboratory abnormality—study treatment continue without interruption. |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| Toxicity | NCI CTCAE Severity Grade | Dose modifications |
|---|---|---|
| | | Crizotinib: Withhold current dose until recovery to Grade ≤1, or to baseline Grade. Then, reduce by 1 dose level and resume treatment, or permanently discontinue as per Investigator judgement. Grade 4 hypophosphatemia and/or hyporuricemia without elimical symptoms: study treatment may continue without interruption as per Investigator judgement. Persistent Grade 4 vomiting or diarrhea despite maximal medical therapy reduce by 1 dose level. |
| Laboratory | Grade 1 | Axitinib. Continue at the same dose level. |
| Investigations: ALT | | Crizotinib: Continue at the same dose level |
| increase with total | Grade 2 | Axitinib: Continue at the same dose level. |
| bilirubin <2 X ULN (in | | Crizotinib Continue at the same dose level |
| absence of cholestasis | | Obtain repeat ALT and total bilirubin when symptomatic or within 7 days. |
| or hemolysis) | Gradé 3 | Axitinib: Reduce by 1 dose level. |
| | | Crizotinib: Withhold until recovery to Grade ≤1, or to baseline Grade. Then, reduce by 1 dose level and resume treatment. If Grade 3 ALT elevation recurs, then reduce further (at most by 2 dose levels from the initial dose level). If recurrence at dose level-2, then discuss with Sponsor whether or not to discontinue permanently. If ALT elevation does not recur after at least 4 weeks, then the dose may be escalated by single dose-level increments up to the initial dose level. |
| | Grade 4 | Axitinib: Withhold current dose until recovery to Grade \$2. Then, reduce by 1 dose level and resume treatment. |
| | | Crizotinib: Withhold until recovery to Grade \$1, or to baseline Grade. Then, reduce by 1 dose level and resume treatment. If Grade 4 ALT elevation recurs, then reduce further (at most by 2 dose levels from the initial dose level). If recurrence at dose level-2, then discuss with Sponsor whether or not to discontinue permanently. If ALT elevation does not recur after at least 4 weeks, then the dose may be escalated by single dose-level increments up to the initial dose level. |
| Laboratory | Grade 1 | Axitinib Continue at same dose level |
| Investigations: ALT<br>increase and bilirubin<br>increase >2 X ULN (in | | Crizotinib: Continue at the same dose level. Obtain repeat ALT and total bilirubin within 48-hours. |
| absence of cholestasis | Grade 2 | Axitinib: Continue at the same dose level |
| or hemolysis) | | Crizotinib: Permanently discontinue. |
| | Grade 3 | Axitinih: Reduce by 1 dose level. |
| | | Crizotinib: Permanently discontinue |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| Toxicity | NCI CTCAE Severity Grade | Dose modifications |
|---|---|---|
| | Grade 4 | Axitinib: Withhold current dose until recovery to Grade ≤2. Then, reduce by 1 dose level and resume treatment. |
| | | Crizotinib: Perminently discontinue |
| Pneumonitis (not<br>attributable to disease<br>progression, infection,<br>other pulmonary<br>disease, or radiation<br>effect. To confirm<br>diagnosis see Section<br>5.3.3.1) | Any Grade | Axitinib: Continue at same dose level * |
| | | Crizotinih: Permanently discentinue |
| Electrocardiogram QT prolongation | Grade I | Axitinib: Continue at the same dose level* |
| | 75.7. | Crizotinib: Continue at the same dose fevel |
| | Gride 2 | Axitinib: Continue at the same dose level* Assess and correct electrolytes (particularly Cn+, K+, and Mg+) and concomitant medications. |
| | | Crizotinib: Continue at the same dose level. Assess and correct electrolytes (particularly Ca+, K+, and Mg+) and concomitant medications. |
| | Grade 3 | Axitinib: Reduce by 1 dose level.* Assess and correct electrolytes (particularly Ca+, K+, Mg+) and concomitant medications. |
| | | Crizotinib: Withhold until recovery to Grade ≤1. Assess and correct electrolytes (particularly Ci+, K+, Mg+) and concomitant medications. Then, reduce by 1 dose level and resume treatment if no other cause for QTc prolongation is found, otherwise resume at the same dose level. |
| | Grade 4 | Axitinib: Withhold current dose until recovery to Grade \$2.* Then, reduce by 1 dose level and resume treatment. |
| | | Crizotinib: Permanently discontinue. |
| Bradysardia | Gride 1 | Axitinib: Continue at the same dose level.* |
| | 0-1-2-N-1-1 | Crizotinib: Continue at the same dose level. |
| | Grade 2 or Grade 3 | Axitinih: Continue at the same dose level.* |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

| Toxicity | NCI CTCAE Severity Grade | Dose modifications |
|---|---|---|
| | | Crizotinib: Withhold until recovery to Grade ≤1. Evaluate concomitant medications known to cause bindycardia, as well as anti-hypertensive medications. If contributing concomitant medication is identified and discontinued, or its dose is adjusted, resume treatment at previous dose. If no contributing concomitant medication is identified, or if contributing concomitant medication is identified, or if contributing concomitant medications are not discontinued or dose modified, then reduce by 1 dose level and resume treatment. |
| | Grade 4 | Axitinib: Continue at the same dose level.* |
| | | Crizotinib: Permanently discontinue if no contributing concomitant medication is identified. If contributing concomitant medication is identified and discontinued, or its dose is adjusted: withhold until recovery to Grade \$1, then reduce to 250 mg QD and resume treatment, with frequent monitoring. Permanently discontinue for recurrence. |
| Vision Disorder | Grade 1 or Grade 2 | Axitinib: Continue at the same dose level.* |
| | | Crizotinib: Continue at the same dose level 1 |
| | Grade 3 | Axitinib: Continue at the same dose level.* If due to a thrombotic event, reduce by 1 dose level. |
| | | Crizotinib: Withhold until recovery to Grade 51. ‡ Then, reduce by 1 dose level and resume treatment. |
| | Grade 4 | Axitinib Continue at the same dose level.* If due to a thrombous event, withhold current dose until recovery to Grade Then, reduce by 1 dose level and resume treatment. Crizotinib Permanently discontinue. † |
| | † Repeat ophthalmologic consultation. For details see Section 7.1.6. | |
| Proteinuna | Dipstick negative or shows 1= (Grade 1) | Axitinib: Continue at the same dose level. |
| Trondularia | 24,000 | Crizotinib Continue at the same dose level. § |
| | If dipatick shows > 1 +, perform 24 hour urine collection. Dosing may continue while waiting for test results | |
| | g proteinuria/24 hour | Axitinib: Continue at the same dose level |
| | | Crizotinib: Continue at the same dose level. § |
| | ≥2 g proteinuria/24 hours | Axifinib: Withhold until proteinura is ≤ g/24 hours. Repeat 24 hour urine collection for proteinuria and creatinine clearance (interval at Investigator discretion) until proteinuria is ≤ g/24 hours. Then, resume at the same dose level or reduce by 1 dose level as per Investigator judgement. |
| | | Judgement. Crizotinib: Continue at the same dose level. § |

AG-013736, PF-02341066-A4061068 Final Protocol Amendment 3, 09 June 2017

| Toxicity | NCI CTCAE Severity Grade | Dose modifications |
|---|---|---|
| les<br>s1.<br>An<br>2 d<br>les | 2 systolic BP readings separated by at<br>least 1 hour show systolic pressure | Axitinib: Continue at the same dose level See Section 5.3.2.3 for monitoring/management of axitinib-related hypertension |
| | ≈150 mm Hg (one or both readings) And 2 diastolic BP readings separated by at least 1 hour show diastolic pressure ≤100 mm Hg (one or both readings) | Crizotinib: Continue at the same dose level. § |
| | 2 systolic BP readings separated by at<br>least 1 hour show systolic pressure<br>>150 mm Hg | Axitinib: If not on maximal antihypertensive treatment, institute new or additional<br>antihypertensive medication and continue at the same dose level<br>If on maximal antihypertensive treatment, reduce by 1 dose level. |
| least I hour show diastolic pressure ≥100 mm Hg 2 systolic BP readings separated by least I hour show systolic pressure ≥160 mm Hg OR 2 diastolic BP readings separated by least I hour show diastolic pressure ≥105 mm Hg Recurrent hypertension following previous dose reduction (2 systolic) readings separated by at least I hour systolic pressure ≥150 mm Hg OR Recurrent diastolic BP ≥100 mm Hg (2 BP readings separated by at least | 2 diastolic BP readings separated by at<br>least 1 hour show diastolic pressure | See Section 5.3.2.3 for monitoring/management of axitinib-related hypertension. Crizotinib Continue at the same dose level § |
| | 2 systolic BP readings separated by at<br>least 1 hour show systolic pressure<br>>160 mm Hg<br>OR<br>2 diastolic BP readings separated by at<br>least 1 hour show diastolic pressure | Axitinib: Withhold until BP is less than 150/100 mm Hg <sup>1</sup> and adjust antihypertensive medication. Then, reduce by 1 dose level and resume treatment. Then, reduce by 1 dose level and resume treatment. If axitinib dosing is temporarily discontinued, patients receiving antihypertensive medications should monitor closely for hypotension. The plasma half-life of axitinib is 2-4 hours and BP usually decreases within 1-2 days following dose interruption. See Section 5.3.2.3 for monitoring/management of axitinib-related hypertension. Crizotinib: Continue at same dose level, 8. |
| | previous dose reduction (2 systolie BP readings separated by at least 1 hour show systolic pressure >150 mm (Ig) | Axitinib: Repeat dose reduction by one lower dose level. See Section 5.3.2.3 for monitoring management of axitinib-related hypertension. Crizotinib: Continue at same dose level § |

<sup>\*</sup> Toxicity not reported in the Investigator Brochure of astimib. Warning and Precautions section. 

Toxicity not reported in the Investigator Brochure of crizonimb, Adverse Drug Reaction section. 

Toxicity not reported in the Investigator Brochure of crizonimb, Adverse Drug Reaction section.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 5.3.2.3. Management of Axitinib-Related Hypertension

Patients will be issued BP cuffs (provided by the Sponsor) for home monitoring and instructed to measure their BP twice daily, prior to taking each dose. All BP measurements will be recorded in a diary and brought to the nurse or study coordinator at each clinic visit. Patients should contact the site for guidance if their systolic BP rises above 150 mm Hg, diastolic BP rises above 100 mm Hg, or if they develop symptoms perceived to be related to elevated BP (eg, headache, visual disturbance).

To treat an increase in BP, standard antihypertensives can be used (for example, thiazide or thiazide-like diuretics, angiotensin II receptor blockers, angiotensin converting-enzyme inhibitors, and dihydropyridine (DHP) calcium channel blockers) although bradycardic agents (such as beta adrenergic blockers with or without alpha-blocking properties, and non-DHP calcium channel blockers, clonidine, digoxin) should be avoided to the extent possible.<sup>37</sup>

### 5.3.3. Crizotinib-Related Adverse Events Safety Monitoring

#### 5.3.3.1. Pneumonitis

Investigators must evaluate thoroughly patients who demonstrate potential signs/symptoms of pneumonitis. If a patient has a potential diagnosis of pneumonitis or drug-related lung injury, then the following evaluations/procedures should be considered to confirm or exclude the diagnosis of pneumonitis during this period in the absence of disease progression, other pulmonary disease, infection, or radiation effects:

- Sputum gram stain and culture (induced sputum if needed) for bacterial, viral, fungal, protozoal, and mycobacterial pathogens.
- Blood culture should be performed in febrile patients. Consider appropriate serologies (mycoplasma, legionella, cytomegalovirus, other viruses, etc.).
- Thoracentesis if pleural fluid is present (culture, microbiology, cytology).
- Bronchoscopy with bronchoalveolar lavage (BAL) if appropriate the BAL fluid should be sent for culture, microbiology, and cytology.
- Lung biopsy (eg, open or thorascopic preferable, bronchoscopy with transbronchial biopsy) if appropriate.
- Plasma sample for BNP (B-type Natriuretic Peptide) to evaluate for evidence of congestive heart failure (CHF).

If clinically appropriate, high-dose corticosteroid treatment should be initiated. Should the event be fatal, an autopsy is highly recommended to confirm or exclude the diagnosis. See Table 5 for appropriate dose modifications.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 5.3.3.2. Renal Cyst

The development of complex renal cysts has been reported in some patients with NSCLC treated with crizotinib. These cysts may be symptomatic or asymptomatic, and have usually developed from 2 to 6 months after starting crizotinib. The precise nature and significance of these cysts is unclear, however, while no evidence of malignancy has been found based on aspiration of cyst fluid and biopsy in the reported cases, complex renal cysts may be associated with renal malignancy, and thus consultation with a urologist or suitable alternate medical expert is recommended.

Active surveillance with appropriate imaging (contrast-enhanced CT scanning or magnetic resonance imaging) should be performed at the time of the renal cysts diagnosis and as scheduled per protocol. Investigators should also review retrospectively all CT/MRIs for any prior occurrence of complex renal cysts.

#### 5.3.4. Overdose Instructions

In the event of an overdose, the Sponsor should be contacted to discuss the details of the overdose and formulate a clinical management plan.

No information regarding overdose of crizotinib in humans is available. In Phase 3 study with axitinib for the treatment of patients with RCC, 1 patient inadvertently received a dose of 20 mg twice daily for 4 days and experienced dizziness (Grade 1). In a clinical dose finding study with axitinib, subjects who received starting doses of 10 mg twice daily or 20 mg twice daily experienced adverse reactions which included hypertension, seizures associated with hypertension, and fatal hemoptysis.

No antidote exists for the treatment of crizotinib or axitinib overdose. In the event of an accidental overdose, the patient should be monitored for possible signs of toxicity as mentioned above, and general supportive care should be provided.

### 5.3.5. Compliance

An Investigational Product (IP) manual will be provided to the sites and will contain information about the drug supplies. A patient diary will be provided to the patients to aid in drug compliance. The diary will be maintained by the patient to include missed or changed doses.

Patients will be required to return all bottles of study medication at each visit. The number of tablets or capsules remaining will be documented and recorded at each clinic visit. The patient diary may also be used to support this part of the drug accountability process.

The site is to follow up (for example, via a telephone call) with each patient at Cycle 1 Day 3 (+ 3 days) to confirm that the patient understands and is in compliance with dosing instructions. The follow-up for dosing compliance by telephone is recommended also whenever there is a dose change.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 5.4. Investigational Product Storage and Accountability

The Investigator, or an approved representative (eg, pharmacist), will ensure that all investigational product is stored in a secured area, under specified storage conditions and in accordance with applicable regulatory requirements.

 Crizotinib and axitinib should be stored at controlled room temperature (between 15-30°C) in provided packaging.

Storage conditions stated in the SRSD (ie, Investigator Brochure) will be superseded by the label storage.

All study drug supplies must be kept in a locked, limited access room. The study drug must not be used outside the context of this protocol. Under no circumstances should the Investigator or other site personnel supply study drug to other Investigators, patients, or clinics, or allow supplies to be used other than directed by this protocol without prior authorization from the Sponsor. The Investigator and or site staff must report any unacceptable condition of the investigational product to the site monitor.

Investigators and site staff are reminded to check temperatures daily (ie, manually or by using alarm systems to alert of any excursions) and ensure that thermometers are working correctly as required for proper storage of investigational products. These include thermometers for both the room storage and refrigerator storage. Any temperature excursions should be reported to the sponsor.

The investigational product(s) must be stored as indicated. Deviations from the storage requirements, including any actions taken, must be documented and reported to the sponsor. Once a deviation is identified, the investigational product must be quarantined and not used until the sponsor provides documentation of permission to use the investigational product.

The Investigator must maintain adequate records documenting the receipt, use, loss, or other disposition of the investigational product. Pfizer may supply drug accountability forms that must be used or may approve use of standard institution forms. In either case, the forms must identify the investigational product, including batch or code numbers, and account for its disposition on a patient-by-patient basis, including specific dates and quantities.

The prescribed dose should be recorded in the patient's medical records. Drug dispensing needs to be verified and documented by a second individual and the forms must be signed by both the individual who dispensed the drug and the second individual who verified the dispensing. Copies must be provided to Pfizer.

All bottles of study drug must be returned to the Investigator by the patient. At the end of the trial, or at appropriate points during the trial, Pfizer will provide instructions as to disposition of any unused investigational product. If Pfizer authorizes destruction at the trial site, the Investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer. Destruction must be adequately documented. If drug destruction is not permitted locally, Pfizer should be contacted for further directions.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 5.5. Concomitant Medication(s)

Concomitant medications and treatments, including herbal supplements, will be recorded from 28 days prior to the start of study treatment and up to 28 days post the last dose of study treatment. All concomitant medications should be recorded in the CRF including supportive care drugs (eg., antiemetic treatment and prophylaxis), and the drugs used to treat adverse events or chronic diseases, and non drug supportive interventions (eg., transfusions).

Concurrent anticancer therapy with agents other than axitinib and crizotinib is not allowed. Medications intended solely for supportive care (ie, antiemetics, analgesics, megestrol acetate for anorexia) are allowed. Investigators are encouraged to employ best supportive care according to local institutional clinical practices and according to the guidance of selected adverse event provided in this protocol.

### 5.5.1. Inhibitors and Inducers of CYP Enzymes

The metabolism of crizotinib is predominantly mediated by the CYP3A4/5 isozymes in human liver microsomes and hepatocytes. Similarly, in vitro studies with human liver microsomes and recombinant CYP enzymes indicate that axitinib metabolism is primarily mediated by the drug-metabolizing enzyme CYP3A4/5, and to a lesser extent by CYP1A2, CYP2C19 and UGT1A1. Co-administration with drugs that are strong CYP3A4/5 inhibitors and inducers may change the plasma concentrations of crizotinib and axitinib.

The concurrent use of strong CYP3A4/5 inhibitors, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice, are not allowed in the study. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.

The concurrent use of strong CYP3A4/5 or CYP1A2 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort, are not allowed in this study.

Crizotinib showed time-dependent inhibition of CYP3A4/5 isozymes in human liver microsomes. In cancer patients, a mean 3.6-fold (90% CI: 2.7-4.9-fold) increase in the oral midazolam AUC was observed following 28 days of crizotinib dosing at 250 mg BID, suggesting that crizotinib is a moderate inhibitor of CYP3A4/5. Caution must be exercised in patients receiving crizotinib in combination with drugs that are predominantly metabolized by CYP3A4/5, such as alfentanil, cyclosporine, fentanyl, quinidine, sirolimus, and tacrolimus. In particular, co-administration of crizotinib with CYP3A4/5 substrates with narrow therapeutic indices including, but not limited to dihydroergotamine, ergotamine, pimozide, astemizole\*, cisapride\*, and terfenadine\* (\*withdrawn from U.S. market) must be avoided from the time of the first dose of crizotinib until treatment discontinuation.

Crizotinib has minimal potential to inhibit other human CYP isoforms such as CYP1A2, CYP2C8, CYP2C9, CYP2C19, and CYP2D6. In vitro studies indicated that axitinib does not inhibit CYP3A4/5, CYP2A6, CYP2C9, CYP2C19, CYP2D6, CYP2E1, or UGT1A1 at therapeutic plasma concentrations.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Additionally, the concurrent use of non-prescription drugs, complementary medicines (excluding vitamins) or herbal supplements is not recommended.

#### 5.5.2. Hematopoietic Growth Factors

Primary prophylactic use of granulocyte-colony stimulating factors is not permitted during the first cycle of treatment but they may be used to treat treatment emergent neutropenia as indicated by the current American Society of Clinical Oncology (ASCO) guidelines.<sup>41</sup>

In subsequent cycles, the use of hematopoietic growth factors is at the discretion of the treating physician in line with local guidelines. Patients who enter the study on stable doses of erythropoietin or darbepoietin may continue this treatment, and patients may start either drug during the study at the discretion of the treating physician.

### 5.5.3. Anti Diarrhea, Anti Emetic Therapy

Patients may receive prophylaxis of treatment-induced diarrhea. Symptomatic care such as loperamide (Imodium<sup>®</sup>) is recommended (4 mg at first onset, then 2 mg every 2-4 hours until symptom-free for 12 hours, for diarrhea Grade  $\geq$ 2). Other anti-diarrheal medications can be used per local standard of care.

Standard anti-emetics may be used for the treatment of nausea and/or vomiting. Taking the medication with food may reduce nausea. The use of anti-emetics for profilaxis may be considered.

#### 5.5.4. Other Concomitant Medications

- Palliative and supportive care for disease-related symptoms, including pain medications, will be allowed to all patients on this trial.
- Patients with fever or infection requiring treatment should be treated with antimicrobials that are not prohibited due to their action on CYP enzymes as noted above.
- Packed red blood cell and platelet transfusions should be administered as clinically indicated.
- Anti-inflammatory or narcotic analgesics may be offered as needed. Acetaminophen/paracetamol to a MAXIMUM total daily dose of 2 g is permitted. Daily intake over 2 g is prohibited.
- Patients who need to be on anticoagulant therapy during treatment should be treated
  with low molecular weight heparin. If low molecular weight heparin cannot be
  administered, the administration of coumadin, other coumarin derivatives, or other
  anticoagulants may be allowed; appropriate monitoring of prothrombin
  time/International normalized ratio (PT/INR) should be performed.
- Patients on this trial may be supported with appropriate hormone replacement therapy as clinically indicated.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Bisphosphonate therapy for metastatic bone disease is permitted. Bisphosphonate therapy should be given as per local medical practice.
- The concurrent use of crizotinib with other bradycardic agents (eg, beta-blockers, non-dihydropyridine calcium channel blockers such as verapamil and diltiazem, clonidine, digoxin) should be avoided to the extent possible due to the increased risk of symptomatic bradycardia. It is important to counsel patients about the risk of bradycardia and inform them of what symptoms and signs to be aware of and actions to take.
- Crizotinib should be used with caution when administered concomitantly with
  medicinal products that are known to prolong QT interval and/or antiarrhythmics, or
  when it is administered to patients who have a history of or predisposition for QTc
  prolongation. When using crizotinib in these patients, periodic monitoring with
  electrocardiograms and electrolytes should be considered.

### 5.5.5. Concomitant Surgery

No formal studies of the effect of axitinib on wound healing have been conducted, however caution is advised based on the mechanism of action. If a major surgery or an interventional procedure (eg., endoscopy) is required, treatment with axitinib must be interrupted at least 24 hours before the procedure and the patient BP should be monitored closely for hypotension. Patients may resume axitinib seven days after minor surgery and 2-3 weeks after major surgery, assuming wound has completely healed and there are no wound healing complications (eg., delayed healing, wound infection or fistula).

The effect of crizotinib on wound healing is not known and has not been investigated; therefore, caution is advised on theoretical grounds (potential antiangiogenic effect). In the event elective surgery is necessary during study participation, crizotinib dosing should be stopped 48 hours before surgery and resumed no sooner than 48 hours after surgery.

#### 5.5.6. Concomitant Radiotherapy

Palliative radiotherapy to specific sites of disease is permitted if considered medically necessary by the treating physician. All attempts should be made to rule out disease progression in the event of increased localized pain. Crizotinib treatment should be interrupted during palliative radiotherapy – stopping 1 day before and resuming treatment 1 day after.

If palliative radiotherapy is needed to control bone pain the sites of bone disease should be present at baseline.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 6. STUDY PROCEDURES

#### 6.1. Screening

Since at the time of this protocol amendment the 11 patients on active treatment have received at least 5 treatment cycles, the screening activities reported in the original Schedule of Activities (SOA) and Assessments section (Section 7) are no longer applicable. Based on that, the original Schedule of Activities has been replaced with a simplified one, not including the screening activities.

#### 6.1.1. Archival Tumor Tissue

All patients will provide a formalin-fixed paraffin embedded (FFPE) archival tumor specimen, or, if not available, a de novo tumor biopsy must be obtained for this purpose in accordance with local institutional practice for tumor biopsies. For patients in the Dose Escalation Phase, the archival tumor tissue can be from either initial diagnosis or recurrence or metastatic site. For patients in the Dose Expansion the archival tumor tissue must be from the initial diagnosis. Formalin fixed, paraffin embedded (FFPE) tissue block of archival tumor tissue that contains sufficient tissue to generate at least 12 unstained slides, each with tissue sections that are 5 microns thick, will be collected. If no FFPE block is available, then at least 12 unbaked and unstained slides containing FFPE tissue sections, that are 5 microns thick must be provided.

#### 6.1.2. De Novo Tumor Biopsy

A de novo tumor biopsy is mandatory for all patients enrolled in Dose Expansion Phase Cohort 2 and should be collected for this purpose in accordance with local institutional practice for tumor biopsies. This de novo biopsy must be taken no more than 28 days prior to registration. Alternatively, a recently obtained FFPE tumor tissue block from a resection or biopsy of a primary, recurrent or metastatic lesion can be provided if the following criteria are met: 1) the biopsy or resection was performed within 4 months of study start AND 2) the patient has not received any new intervening systemic anti-cancer treatment from the time the tissue was obtained and the study start.

Patients enrolled into the Dose Escalation Phase or into the Dose Expansion Phase Cohort 1 may provide a de novo biopsy on a voluntary basis. For those patients, this sample will be provided in addition to the archived tumor tissue that is required for enrollment, unless archived tumor tissue is not available in which case the de novo biopsy is mandatory.

The de novo biopsy will consist of an incisional or excisional biopsy, or a core needle biopsy, of a primary or metastatic lesion. Fine needle aspiration biopsies are not acceptable. The tumor tissue will be processed as specified in the Laboratory Manual.

### 6.2. Study Period

For treatment period procedures, see Schedule of Activities (SOA) and Assessments section (Section 7).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 6.3. Follow-up Visit

For follow-up procedures see Schedule of Activities (SOA) and Assessments section (Section 7).

#### 6.4. Patient Withdrawal

Patients may withdraw from treatment at any time at their own request, or they may be withdrawn at any time at the discretion of the Investigator or Sponsor for safety or behavioral reasons, or the inability of the patient to comply with the protocol required schedule of study visits or procedures at a given study site.

Reasons for discontinuation of study treatment may include:

- Objective disease progression according to RECIST version 1.1; however, patients
  with disease progression who are continuing to derive clinical benefit from the study
  treatment will be eligible to continue with single agent axitinib or axitinib plus
  crizotinib provided that the treating physician has determined that the benefit/risk for
  doing so is favorable;
- · Global deterioration of health status requiring discontinuation;
- Unacceptable toxicity. If the unacceptable toxicity is attributed to one of the two study drugs, the Investigator (in discussion with the Sponsor) can continue the study treatment with the other study drug;
- Pregnancy;
- Significant protocol violation (post study start; includes patient noncompliance);
- · Lost to follow-up:
- Patient refused further treatment (follow-up permitted by patient);
- · Study terminated by Sponsor;
- Death

Reasons for withdrawal from study follow-up may include:

- · Completed study follow-up:
- Study terminated by Sponsor;
- · Lost to follow-up;
- Refusal for further follow-up for survival;

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### Death.

If a patient does not return for a scheduled visit, every effort should be made to contact the patient. All attempts to contact the patient and information received during contact attempts must be documented in the patient's medical record. In any circumstance, every effort should be made to document patient outcome, if possible. The Investigator should inquire about the reason for withdrawal, request the patient to return all unused investigational product(s), request the patient to return for a final visit, if applicable, and follow up with the patient regarding any unresolved AEs.

If the patient withdraws from the study, and also withdraws consent for disclosure of future information, no further evaluations should be performed, and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

#### 7. ASSESSMENTS

Every effort should be made to ensure that the protocol required tests and procedures are completed as described. However it is anticipated that from time to time there may be circumstances, outside of the control of the Investigator, that may make it unfeasible to perform the test. In these cases the Investigator will take all steps necessary to ensure the safety and well being of the patient. When a protocol required test cannot be performed the Investigator will document the reason for this and any corrective and preventive actions which he/she has taken to ensure that normal processes are adhered to as soon as possible. The study team will be informed of these incidents in a timely fashion.

#### 7.1. Safety Assessment

Safety assessments will include collection of AEs, SAEs, vital signs and physical examination, ECG (12-lead), laboratory assessments, including pregnancy tests and verification of concurrent medications.

### 7.1.1. Pregnancy Testing

For female patients of childbearing potential, a serum or urine pregnancy test, with sensitivity of at least 25 mIU/mL, will be performed on two occasions prior to starting study treatment, once at the start of screening and once at the baseline visit, immediately before investigational product administration. Following a negative pregnancy test result at screening, appropriate contraception must be commenced and another negative pregnancy test result will then be required at the baseline visit before the patient may receive the investigational product. Pregnancy tests will also be routinely repeated at every treatment cycle during the active treatment period, at the end of studytreatment and additionally whenever one menstrual cycle is missed or when potential pregnancy is otherwise suspected. In the case of a positive hCG test, the patient will be withdrawn from administration of investigational product but may remain in the study.

Additional pregnancy tests may also be undertaken if requested by Institutional Review Board/Independent Ethics Committees (IRB/IECs) or if required by local regulations.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Note: the 11 patients on active treatment are 10 male and 1 female in postmenopausal status for  $\geq$  2 years. Based on that, the pregnancy test is no longer required in the simplified Schedule of Activities.

#### 7.1.2. Adverse Events

Assessment of adverse events will include the type, incidence, severity (graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CAE] version 4.03), timing, seriousness, and relatedness.

Adverse events that occur during the study, including baseline signs and symptoms, will be recorded on the adverse events CRF page.

### 7.1.3. Laboratory Safety Assessment

Haematology and blood chemistry will be drawn at the time points described in the Schedule of activities (SOA) and analyzed at local laboratories. The required laboratory tests are listed in Table 6.

Table 6. Required Laboratory Tests

| Hematology | Chemistry | Urinalysis | Coagulation<br>Tests | Pregnancy<br>Tests |
|---|---|---|---|---|
| Hemoglobin | ALT | Protein, glucose and<br>blood. | PT | For female<br>patients of<br>childbearing<br>potential, serum<br>or urine |
| Platelets | AST<br>Alk Phos<br>Sodium | | INR | |
| WBC | | | | |
| Absolute Neutrophils | | Urine dipstick for | | |
| Absolute Lymphocytes | Potassium | urine protein: If positive collect 24-hour and microscopic (Reflex Testing) | | |
| Absolute Monocytes | Magnesium | | | |
| Absolute Eosinophils | Chloride | | | |
| Absolute Basophils | Calcium | | | |
| | Total Bilirubin sales | | | |
| | BUN or Urca | Urine dipstick for<br>urine blood: If positive<br>collect a microscopic<br>(Reflex Testing) | | |
| | Creatinine | | | |
| | Une Acid | | | |
| | Glucose (non-fasted) | | | |
| | Albumin | | | |
| | Total Protein | | | |
| | Phosphorus or Phosphate | | | |
| | Thyroid Function Tests:<br>TSH, free T3, free T4 (as<br>indicated) | | | |

<sup>\*\*\*</sup> For potential Hy's law cases, in addition to repeating AST and ALT, laboratory tests should include albumin, creatine kinase, total bilirubin, direct and indirect bilirubin, gamma glutamyl transferase, prothrombin time (PT)/INR, alkaline phosphatase, total bile acids and acetaminophen drug and/or protein adduct levelss.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 7.1.4. Vital Signs and Physical Examination

Patients will have a physical exam to include weight, blood pressure, pulse rate, assessment of ECOG performance status and height; height will be measured at screening only. Blood pressure and pulse rate should be taken with the patient in the seated position after the patient has been sitting quietly for at least 5 minutes. Two blood pressure readings will be taken at least 1 hour apart at each clinic visit.

#### 7.1.5. ECG Measurements

A 12-lead (with a 10-second rhythm strip) tracing will be used for all ECGs. Triplicate ECG measurements will be obtained at all time points except for a single ECG measurement at screening. For triplicate measures, three consecutive 12-lead ECGS will be collected approximately 2 minutes apart. It is required that the machine used has a capacity to calculate the standard intervals automatically. ECG measurements will include PR interval, OT interval, RR interval, and ORS complex. Additional ECGs will be performed as clinically indicated. If the OTc is prolonged (≥501 msec), then the ECG should be read by a cardiologist at the site for confirmation. Any manual overread done at site must be entered into the CRF as an unplanned ECG result. In case of a QTc interval measurement ≥501 msec (Grade ≥3) dosing should be interrupted, and permanently discontinued for a Grade 4 QTc prolongation. For Grade 3 or 4 QTc prolongations continuous ECG monitoring will be done under physician supervision until the QTc recovers to Grade ≤1. Triplicate ECG surveillance will again be performed when crizotinib is restarted on a reduced dose due to Grade 3 QTc prolongation. The timing of the triplicate assessment of ECGs should be prior to (0 hour) and 2-6 hours after morning dosing of crizotinib on Day 1 of Cycles 1, 2, and 3, and on Day 15 of Cycle 1. Additional ECGs will be performed as clinically indicated.

### 7.1.6. Ophthalmology Examinations

Ophthalmologic examinations for both right and left eyes will be performed at screening and should be performed by an ophthalmologist.

Ophthalmologic examinations should be repeated during the course of the study whenever a vision disorder AE is observed or CTCAE grade change occurs from a previous visit.

### **Best Corrected Visual Acuity and Refraction**

Best corrected visual acuity will be assessed using a standard wall or projection chart (Snellen) before implementing any procedures that can affect vision (eg, pupil dilation). The same chart will be used throughout the study for a specific patient, and the right eye should be tested first. The refractive error also will be determined. The examiner should ensure that patients are seated comfortably and that they do not move their head forward or backward during testing. Patients will be told that the chart contains only letters.

The line read with 2 or fewer errors will be recorded. If 3 of the 5 letters on a line are read correctly, then the patient will be given credit for that line. For example, if the patient reads 20/25 +3, then 20/20 will be recorded,

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

A decrease in best-corrected visual acuity of 3 lines or more from the Screening visit should be reported as an adverse event. An adverse event of visual acuity will be counted from the following lines: 20/20 or better, 20/25, 20/30, 20/40, 20/50, 20/60, 20/70, 20/80, 20/100, 20/125, 20/150, and 20/200. If the acuity at screening is better than 20/20, then the decrease will be calculated from 20/20.

In the event of a decrease in visual acuity of 3 lines or more from screening, refraction should be rechecked.

#### Biomicroscopy

Slit-lamp biomicroscopy without dilation of the pupil will be performed a qualified practioner. Slit-lamp biomicroscopy should precede intraocular pressure (IOP) measurement and the administration of any pupil-dilating agent for ophthalmoscopy.

Any abnormalities of the lids, conjunctivae, cornea, anterior chamber, iris, or lens will be recorded at screening and any change from screening will be graded as mild, moderate, or severe. Aphakia or intraocular lens (anterior chamber intraocular lens, posterior chamber intraocular lens, or iris clip) and status of the posterior lens capsule (intact, open, or absent) should be specified. Cells and flare in the anterior chamber should be noted during the slit-lamp examination.

Table 7. Intraocular Inflammation Grading Scale for Biomicroscopy

| | Grade | | | | |
|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 |
| Grading of aqueous flare <sup>a</sup> | Completely<br>Absent | Barely<br>Detectable | Moderate (iris and<br>lens details clear) | Marked (ins<br>and lens details<br>hazy) | Intense<br>(formed fibrin<br>in aqueous) |
| Grading of cells in<br>the aqueous <sup>a,b</sup> | No cells | 1 to 5 cells | 6 to 10 cells | 11 to 20 cells | >20 cells |

- \* Evaluation of Anterior Chamber Inflammation:
  - Examination of the anterior chamber for cells must be performed before either dilation or applanation tonometry.
  - 2. The light intensity of the slit lamp is turned to the maximum tolerated by the patient.
  - 3. High magnification and 1 x 2 mm slit are used
  - 4. The ray of light as directed at an angle of approximately 45° to the plane of the iris.
- Modified from Hogan MJ, Kimura SJ, Thygeson P: Signs and symptoms of uveitis: I. Anterior uveitis. Am J Ophthalmol 1959:47:155-70.

#### Ophthalmoscopy

Ophthalmoscopy will be performed after pupillary dilation to examine the vitreous body, retina macular, retina non-macula (peripheral), and optic nerve head.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

For those patients who are selected for additional testing based on clinical judgment, the refractive error (sphere, cylinder, axis), pupillary size (millimeters), optical coherence tomographic central retinal subfield thickness (microns), and intraocular pressure (mm Hg) will be collected at screening and during the treatment period, and as clinically indicated.

#### 7.2. Pharmacokinetics Assessments

Since at the time of this protocol amendment the 11 patients on active treatment have received at least 5 treatment cycles, the PK activities required in the original Schedule of Activities (SOA) and in this section are no longer applicable. Based on that, the original Schedule of Activities has been replaced with a simplified one, no longer including the PK assessments.

Plasma samples will be obtained from all patients for PK analysis of axitinib and crizotinib (and its metabolite) depending on the treatment cohort that they belong to.

### 7.2.1. Blood Sample Collection for Pharmacokinetic Analysis

Where noted in the Schedule of Activities (SOA), blood samples will be collected at approximately the same time as other assessments wherever possible. Pharmacokinetic samples will be collected from all patients in the Dose Escalation Phase. In the Dose Expansion Phase, pharmacokinetic samples will be obtained from at least 8 evaluable patients in Cohort 1.

PK table indicates PK blood sampling time points for axitinib alone and axitinib in combination with crizotinib. On the days of sample collection, patients should be instructed to hold morning dosing until the pre dose sample has been drawn. Patients should have been taking axitinib uninterrupted for at least 3 days prior to each of the axitinib pharmacokinetic sample collection visits. For all collections, the time of dosing, as well as actual times of pharmacokinetic collections will be recorded in the source documents and CRF.

The pharmacokinetics of steady state axitinib alone will be evaluated on Lead-in Day 7. Pharmacokinetics of axitinib and crizotinib will be evaluated on Cycle 1 Day 15. The pharmacokinetics of crizotinib alone will be evaluated on Day 1 of Cycle 2, Cycle 3. Cycle 4 and Cycle 5.

Serial pharmacokinetic samples for axitinib will be collected on Lead-in Day 7 and Cycle 1 Day 15. Serial pharmacokinetic samples for crizotinib will be collected on Cycle 1 Day 15. On both days of serial pharmacokinetic sampling (Lead-in Day 7 and Cycle 1 Day 15), blood samples will be obtained at the following time points: predose, 1, 2, 3, 4, 6, and 8 hours after dosing. Additionally, predose samples for crizotinib will be collected on Day 1 of Cycle 2, Cycle 3, Cycle 4 and Cycle 5.

In addition to samples collected at the scheduled times, an additional blood sample should be collected from patients experiencing unexpected and/or SAE's and the date and time documented in the CRF.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

All efforts will be made to obtain the pharmacokinetic samples at the scheduled nominal time relative to dosing. If a scheduled blood sample collection cannot be completed for any reason, the missed sample time may be re scheduled with agreement of clinical Investigators, patient and Sponsor.

PK samples will be assayed for axitinib, crizotinib and related metabolites using validated analytical methods in compliance with Pfizer standard operating procedures. Additional details regarding the collection, processing, storage and shipping of the blood samples will be provided in the study manual.

### 7.2.2. Collection of Crizotinib PK Samples

At each time point for crizotinib, a 3 mL whole blood sample will be collected into an appropriately labeled K<sub>2</sub>EDTA tubes to provide a minimum of 1 mL plasma for pharmacokinetic analysis.

### 7.2.3. Collection of Axitinib PK Samples

At each time point for axitinib, a 3 mL whole blood sample will be collected into an appropriately labeled K<sub>3</sub>EDTA tubes to provide a minimum of 1 mL plasma for pharmacokinetic analysis.

#### 7,2.4. Processing, Storage and Shipment of Crizotinib and Axitinib PK Samples

The following special precautions should be taken to minimize the rapid degradation of axitinib and crizotinib in plasma when exposed to visible light:

- Following collection of blood samples, samples should be processed as soon as
  possible. Preferably, harvested plasma should be frozen within 1 hour of collection.
- The blood collection tube should be gently inverted (8-10 times) to thoroughly mix the blood with the anti-coagulant.
- Vacutainer tubes should be protected from light (covered completely in aluminum foil or in black protection tubes) and placed in an ice-bath while samples are waiting to be centrifuged to harvest plasma.
- Following centrifugation (for at least 10 minutes at 1700 g at 4°C or lower), plasma should be transferred rapidly to labeled amber cryovials and stored at -20°C or lower.
- All samples should be transferred to an opaque box to protect from light exposure during storage and shipment. If a sample is inadvertently exposed to light (for 5 minutes or more), the sponsor should be notified so that the sample can be flagged for possibly spurious results.
- Once frozen, samples should not be allowed to thaw, including during shipment.
AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Samples will be shipped with the completed sample inventory form and sufficient dry ice to last for at least two days. Detailed instructions on sample collection, preparation, storage, and shipping will also be provided in the Study Manual.

Axitinib and crizotinib pharmacokinetic samples will be analyzed using separate validated analytical methods for each drug in compliance with Pfizer Standard Operating Procedures to determine plasma concentrations for axitinib, crizotinib and their metabolites. As part of the understanding of the pharmacokinetics of the study drug, samples may be used for potential qualitative and/or quantitative metabolite analyses and/or evaluation of the bioanalytical methods for axitinib, crizotinib and their metabolites. The results of such analyses may be included in the clinical report.

### 7.3. Pharmacodynamic Assessments

A key objective of the biomarker analyses that will be performed in this study is to investigate candidate biomarkers that may have predictive value in identifying those patients who may benefit from treatment with crizotinib when used in combination with a VEGF inhibitor. In addition, analyses of sequentially obtained tissue and blood biomarkers will provide an opportunity to investigate potential mechanisms of resistance as well as pharmacodynamic markers that may further the understanding of the mechanistic effects of the drug combination being studied. As described in the Rationale for Protocol Amendment #3, enrollment in Expansion Phase Cohort 2 was challenging and afforded small patient numbers (7 patients overall), which led to a decision to discontinue further enrollment. For these reasons, biomarker analyses will be performed only on Cohort 1.

### 7.3.1. Archived Tumor Tissue and De Novo Tumor Biopsies

Tumor tissue from archived tissue samples and/or a de novo biopsy (see Section 6.1.1 and 6.1.2) will be used to analyze candidate DNA, RNA or protein markers for their ability to predict or identify those patients who are most likely to benefit from treatment with the study drugs. Markers that may be analyzed include, but may not be limited to, cMET gene mutation and gene amplification, PTEN mutation or deletion; c-MET, HGF, PBRM1 protein expression assessed by immunohistochemistry (IHC). Comparisons between de novo biopsies from RCC patients treated with one prior line of systemic therapy and archived tumor tissue obtained prior to the one line of systemic treatment will be made to investigate whether potential predictive markers represent intrinsic or acquired mechanisms of resistance. As described in the Rationale for Protocol Amendment #3, enrollment in Expansion Phase Cohort 2 was challenging and afforded small patient numbers (7 patients overall), which led to a decision to discontinue further enrollment. For these reasons, biomarker analyses will be performed only on Cohort 1.

### 7.3.2. Peripheral Blood

Blood samples for plasma and serum preparations will be obtained from all enrolled patients (in the Dose Escalation Phase and in the Dose Expansion Phase Cohort 1 and 2) to measure DNA, RNA or protein markers known or suspected to be of relevance to the mechanism of action, the development of resistance, or the identification of those patients who might benefit from treatment with axitinib and crizotinib combination. Markers that may be

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

analyzed include, but may not be limited to, the soluble c-MET ectodomain, HGF, Ang 2, and miRNA signature. Samples should be obtained pre-dose and at the same time as PK samples whenever possible (see Schedule of Activities). As described in the Rationale for Protocol Amendment #3, enrollment in Expansion Phase Cohort 2 was challenging and afforded small patient numbers (7 patients overall), which led to a decision to discontinue further enrollment. For these reasons, biomarker analyses will be performed only on Cohort 1.

### 7.4. Banked Biospecimens

### 7.4.1. Markers of Drug Response

Studying the variation in genetic markers and other biomarkers may help to explain some of the variability in response seen with some drugs among different individuals. This is referred to as pharmacogenomic/biomarker research. Comparing the DNA, RNA, protein, and metabolite variation patterns of patients who respond well and those who respond poorly to treatment may help to better define the most appropriate group of patients in which to target a given treatment. Collecting biospecimens for exploratory pharmacogenomic/biomarker analyses and retaining them in the Pfizer BioBank makes it possible to better understand the drug's mechanism of action and to seek explanations for differences in, for example, exposure, efficacy, tolerability, or safety not anticipated prior to the beginning of the study. Providing these biospecimens is a required study activity for study sites and patients, unless prohibited as such by local regulations or ethics committee decision.

To protect patients' confidentiality, the banked biospecimens and data generated from them will be coded with the patient's study identification (ID) number. Samples will be kept in a facility accessible only by swiping a badge. Data will be stored on password-protected computer systems. The key between the code and the patient's personal identifiers will be held at the study site; the researchers using the biospecimens and data generated from them will not have access to the key or any personally identifying information. Biospecimens will be used only for the purposes described here and in the informed consent document/patient information sheet; any other uses require additional ethical approval. Unless a time limitation is required by local regulations or ethical requirements, biospecimens will be stored indefinitely to allow for future research on the topics described here, including research conducted during the lengthy drug development process and also post-marketing research. Patients can withdraw their consent for the use of their biospecimens at any time by making a request to the Investigator, in which event any remaining biospecimen will be destroyed; data already generated from the biospecimens will continue to be stored to protect the integrity of existing analyses. It is very unlikely that results generated from the biospecimens will have any clinical, diagnostic, or therapeutic implications for the individual study participants. Patients are notified in the informed consent document/patient information sheet that their results will not be given to them, unless required by local laws or regulations, in which case results will be returned via the Investigator. Results will not be provided to family members or other physicians; nor will they be recorded in the patient's medical record. There is no intention to contact patients after completion of the clinical trial.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

A 4 mL blood biospecimen **Prep D1** (**K**<sub>2</sub> **EDTA whole blood collection optimized for DNA analysis**) will be collected at the Baseline visit to be retained for potential pharmacogenomic/biomarker analyses related to drug response, unless prohibited by local regulations or ethics committee decision. For example, putative safety biomarkers, drug metabolizing enzyme genes, drug transport protein genes, or genes thought to be related to the mechanism of drug action may be examined.

### 7.4.2. Additional Research

Unless prohibited by local regulations or ethics committee decision, patients will be asked to indicate on the consent form whether they will allow the Banked Biospecimens to also be used for the following research:

- . Investigations of the disease under study in the clinical trial, and related conditions.
- Biospecimens may be used as controls. This includes use in case-control studies of diseases for which Pfizer is researching drug therapies; use in characterizing the natural variation amongst people in genes, RNA, proteins, and metabolites; and use in developing new technologies related to Pharmacogenomics/biomarkers.

Patients need not provide additional biospecimens for the uses described in this section; the biospecimen specified in Markers of Drug Response Section will be used. Patients may still participate in the clinical trial if they elect not to allow their Banked Biospecimens to be used for the additional purposes described in this section.

## 7.5. Tumor Response Assessments

Tumor assessments will include all known or suspected disease sites. Imaging may include chest, abdomen and pelvis CT or magnetic resonance imaging (MRI) scans; brain CT or MRI scan for patients with suspected brain metastases. The CT scans should be performed with contrast agents unless contraindicated for medical reasons.

The same imaging technique used to characterize each identified and reported lesion at baseline will be employed in the following tumor assessments.

Antitumor activity will be assessed through radiological tumor assessments conducted at baseline, and then according to local clinical practice, but not less than every 12 weeks (±2 weeks), whenever disease progression is suspected (eg. symptomatic deterioration), and at the time of withdrawal from the treatment (if not done in the previous 12 weeks).

For patients with known or suspected bone metastases a bone scan (bone scintigraphy) or <sup>18</sup>F-FDG-PET/CT is required at screening. Repeat bone imaging is required every 16 weeks only if bone metastases are present at baseline. Otherwise bone imaging is required only if new bone metastases are suspected. Bone imaging is also required at the time of confirmation of response for patients who have bone metastases.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Measurable or evaluable lesions that have been previously irradiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.

Assessment of response will be made using RECIST version 1.1 (Appendix 2),

All patients' files and radiologic images must be available for source verification and for potential peer review.

### 8. ADVERSE EVENT REPORTING

#### 8.1. Requirements

The table below summarizes the requirements for recording safety events on the CRF and for reporting safety events on the Clinical Trial (CT) Serious Adverse Event (SAE) Report Form to Pfizer Safety. These requirements are delineated for 3 types of events: (1) SAEs; (2) non-serious adverse events (AEs); and (3) exposure to the investigational product under study during pregnancy or breastfeeding, and occupational exposure.

| Safety Event | Recorded on the CRF | Reported on the CT<br>SAE Report Form to<br>Pfizer Safety Within<br>24 Hours of Awareness |
|---|---|---|
| SAE | All | All |
| Non-serious AE | All | None |
| Exposure to the investigational product under study during pregnancy or breastfeeding, and occupational exposure | All (regardless of whether associated with an AE), except occupational exposure | Exposure during pregnancy, exposure via breastfeeding, occupational exposure (regardless of whether associated with an AE) |

All observed or volunteered AEs regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported as described in the following paragraphs.

Events listed in the table above that require reporting to Pfizer Safety on the CT SAE Report Form within 24 hours of awareness of the event by the investigator are to be reported regardless of whether the event is determined by the investigator to be related to an investigational product under study. In particular, if the SAE is fatal or life-threatening, notification to Pfizer Safety must be made immediately, irrespective of the extent of available event information. This time frame also applies to additional new (follow-up) information on previously forwarded reports. In the rare situation that the investigator does not become

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

immediately aware of the occurrence of an event, the investigator must report the event within 24 hours after learning of it and document the time of his/her first awareness of the event

For each event, the Investigator must pursue and obtain information adequate both to determine the outcome and to assess whether it meets the criteria for classification as an SAE (see the Serious Adverse Events section below). In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion. This information is more detailed than that recorded on the CRF. In general, this will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a patient death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety. Any pertinent additional information must be reported on the CT SAE Report Form; additional source documents (eg, medical records, CRF, laboratory data) are to be sent to Pfizer Safety ONLY upon request.

As part of ongoing safety reviews conducted by the Sponsor, any non-serious adverse event that is determined by the Sponsor to be serious will be reported by the Sponsor as an SAE. To assist in the determination of case seriousness further information may be requested from the Investigator to provide clarity and understanding of the event in the context of the clinical study.

### 8.1.1. Additional Details On Recording Adverse Events on the CRF

All events detailed in the table above will be recorded on the AE page(s) of the CRF. It should be noted that the CT SAE Report Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the CT SAE Report Form for reporting of SAE information.

## 8.1.2. Eliciting Adverse Event Information

The investigator is to record on the CRF all directly observed AEs and all AEs spontaneously reported by the study patient. In addition, each study patient will be questioned about the occurrence of AEs in a non-leading manner.

## 8.1.3. Withdrawal From the Study Due to Adverse Events (see also the Patient Withdrawal section)

Withdrawal due to AEs should be distinguished from withdrawal due to other causes, according to the definition of AE noted below, and recorded on the CRF.

When a patient withdraws from the study because of an SAE, the SAE must be recorded on the CRF and reported, as appropriate, on the CT SAE Report Form, in accordance with the Requirements section above.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 8.1.4. Time Period for Collecting AE/SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each patient begins from the time the patient provides informed consent, which is obtained before the patient's participation in the study (ie, before undergoing any study-related procedure and/or receiving investigational product), through and including a minimum of 28 calendar days after the last administration of the investigational product.

For patients who are screen failures, the active collection period ends when screen failure status is determined.

### 8.1.4.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a patient during the active collection period are reported to Pfizer Safety on the CT SAE Report Form.

SAEs occurring in a patient after the active collection period has ended are reported to Pfizer Safety if the investigator becomes aware of them; at a minimum, all SAEs that the investigator believes have at least a reasonable possibility of being related to investigational product must be reported to Pfizer Safety.

Follow up by the investigator continues throughout and after the active collection period and until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

If a patient begins a new anticancer therapy, SAEs occurring during the above-indicated active collection period must still be reported to Pfizer Safety irrespective of any intervening treatment.

### 8.1.4.2. Recording Non-serious AEs and SAEs on the CRF

During the active collection period, both non-serious AEs and SAEs are recorded on the CRF.

Follow-up by the investigator may be required until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

If a patient begins a new anticancer therapy, the recording period for non-serious AEs ends at the time the new treatment is started; however, SAEs must continue to be recorded on the CRF during the above-indicated active collection period.

#### 8.1.5. Causality Assessment

The investigator's assessment of causality must be provided for all AEs (serious and non-serious); the investigator must record the causal relationship on the CRF, and report such an assessment in accordance with the SAE reporting requirements, if applicable. An investigator's causality assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an AE; generally the facts (evidence) or arguments to suggest a causal relationship should be provided. If the

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

investigator does not know whether or not the investigational product caused the event, then the event will be handled as "related to investigational product" for reporting purposes, as defined by the sponsor. If the investigator's causality assessment is "unknown but not related" to investigational product, this should be clearly documented on study records.

In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the CT SAE Report Form and in accordance with the SAE reporting requirements.

### 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities

AE reporting, including suspected unexpected serious adverse reactions, will be carried out in accordance with applicable local regulations.

### 8.2. Definitions

#### 8.2.1. Adverse Events

An AE is any untoward medical occurrence in a study patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Examples of AEs include, but are not limited to:

- Abnormal test findings;
- Clinically significant symptoms and signs;
- Changes in physical examination findings;
- Hypersensitivity;
- Drug abuse;
- Drug dependency.

Additionally, they may include the signs or symptoms resulting from:

- Drug overdose;
- Drug withdrawal;
- Drug misuse;
- Drug interactions:
- Extravasation;
- · Exposure during pregnancy (EDP);

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- · Exposure via breastfeeding:
- Medication error;
- · Occupational exposure:

Worsening of signs and symptoms of the malignancy under study should be reported as AEs in the appropriate section of the CRF. Disease progression assessed by measurement of malignant lesions on radiographs or other methods should not be reported as AEs.

### 8.2.2. Abnormal Test Findings

Abnormal objective test finding should be recorded as AE when any of the following conditions are met:

- Test result is associated with accompanying symptoms; and/or
- Test result requires additional diagnostic testing or medical/surgical intervention; and/or
- Test result leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy; and/or
- Test result is considered to be an AE by the Investigator or Sponsor.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an AE. Any abnormal test result that is determined to be an error does not require reporting as an AE.

#### 8.2.3. Serious Adverse Events

A serious adverse event is any untoward medical occurrence at any dose that:

- Results in death:
- . Is life-threatening (immediate risk of death),
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions);
- · Results in congenital anomaly/birth defect;

Or that is considered to be:

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

An important medical event.

Medical and scientific judgment is exercised in determining whether an event is an important medical event. An important medical event may not be immediately life-threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the patient or may require intervention to prevent one of the other AE outcomes, the important medical event should be reported as serious.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

Progression of the malignancy under study (including signs and symptoms of progression) should not be reported as an SAE unless the outcome is fatal within the active collection period. Hospitalization due to signs and symptoms of disease progression should not be reported as an SAE. If the malignancy has a fatal outcome during the study or within the active collection period, then the event leading to death must be recorded as an AE on the CRF, and as an SAE with CTCAE Grade 5 (see the Severity Assessment section).

### 8.2.4. Hospitalization

Hospitalization is defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility, or any prolongation of an existing admission. Admission also includes transfer within the hospital to an acute/intensive care unit (eg. from the psychiatric wing to a medical floor, medical floor to a coronary care unit, or neurological floor to a tuberculosis unit). An emergency room visit does not necessarily constitute a hospitalization; however, the event leading to the emergency room visit is assessed for medical importance.

Hospitalization does not include the following:

- · Rehabilitation facilities;
- Hospice facilities;
- Respite care (eg, caregiver relief);
- Skilled nursing facilities;
- Nursing homes;
- Same-day surgeries (as outpatient/same-day/ambulatory procedures).

Hospitalization or prolongation of hospitalization in the absence of a precipitating clinical AE is not in itself an SAE. Examples include:

 Admission for treatment of a preexisting condition not associated with the development of a new AE or with a worsening of the preexisting condition (eg. for workup of a persistent pretreatment laboratory abnormality);

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Social admission (eg, patient has no place to sleep);
- Administrative admission (eg, for yearly physical examination);
- Protocol-specified admission during a study (eg, for a procedure required by the study protocol);
- Optional admission not associated with a precipitating clinical AE (eg, for elective cosmetic surgery);
- Hospitalization for observation without a medical AE;
- Preplanned treatments or surgical procedures. These should be noted in the baseline documentation for the entire protocol and/or for the individual patient;
- Admission exclusively for the administration of blood products.

Diagnostic and therapeutic noninvasive and invasive procedures, such as surgery, should not be reported as SAEs. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an SAE. For example, an acute appendicitis that begins during the reporting period should be reported if the SAE requirements are met, and the resulting appendectomy should be recorded as treatment of the AE.

### 8.3. Severity Assessment

| GRADE | Clinical Description of Severity |
|---|---|
| 0 | No change from normal or reference range (This grade is not included in the Version 4.03 CTCAE document but may be used in certain circumstances.) |
| 1 | MILD adverse event |
| 2 | MODERATE adverse event |
| 3 | SEVERE adverse event |
| 4. | LIFE-THREATENING consequences; urgent intervention indicated |
| 5 | DEATH RELATED TO adverse event |

Note the distinction between the severity and the seriousness of an AE. A severe event is not necessarily an SAE. For example, a headache may be severe (interferes significantly with the patient's usual function) but would not be classified as serious unless it met one of the criteria for SAEs, listed above.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 8.4. Special Situations

### 8.4.1. Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury, but adapt are termed "adaptors." In some patients, transaminase elevations are a harbinger of a more serious potential outcome. These patients fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as drug-induced liver injury (DILI). Patients who experience a transaminase elevation above 3 times the upper limit of normal (\* ULN) should be monitored more frequently to determine if they are an "adaptor" or are "susceptible."

In the majority of DILI cases, elevations in aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) precede total bilirubin (TBili) elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same lab sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the patient's individual baseline values and underlying conditions. Patients who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

- Patients with AST or ALT and total bilirubin baseline values within the normal range
  who subsequently present with AST OR ALT >3 x ULN AND a total bilirubin value
  >2 X ULN with no evidence of hemolysis and an alkaline phosphatase value <2 X
  ULN or not available.</li>
- For patients with preexisting ALT OR AST OR total bilirubin values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Pre-existing AST or ALT baseline values above the normal range; AST or ALT value >2 times the baseline values AND >3 X ULN, or >8 X ULN (whichever is smaller).
  - Pre-existing values of total bilirubin above the normal range: Total bilirubin level
    increased from baseline value by an amount of at least 1 x ULN or if the value
    reaches >3 x ULN (whichever is smaller).

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Rises in AST/ALT and total bilirubin separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The patient should return to the investigational site and be evaluated as soon as possible. preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history and physical assessment and for oncology studies, the possibility of hepatic neoplasia (primary or secondary) should be considered. In addition to repeating measurements of AST and ALT and total bilirubin, laboratory tests should include albumin, creatine kinase (CK), direct and indirect bilirubin, gamma-glutamyl transferase, prothrombin time (PT)/INR, total bile acids, alkaline phosphatase and acetaminophen drug and/or protein adduct levels. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection and liver imaging (eg, biliary tract) may be warranted.

All cases confirmed on repeat testing as meeting the laboratory criteria of AST/ALT and total bilirubin elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the LFT abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

## $\bf 8.4.2. \ Exposure \ to \ the \ Investigational \ Product \ During \ Pregnancy \ or \ Breastfeeding, and \ Occupational \ Exposure$

Exposure to the investigational product under study during pregnancy or breastfeeding and occupational exposure are reportable to Pfizer Safety within 24 hours of investigator awareness.

## 8.4.2.1. Exposure During Pregnancy

For both unapproved/unlicensed products and for marketed products, an exposure during pregnancy (EDP) occurs if:

 A female becomes, or is found to be, pregnant either while receiving or having been exposed (eg. because of treatment or environmental exposure) to the investigational product; or the female becomes or is found to be pregnant after discontinuing and/or being exposed to the investigational product;

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

An example of environmental exposure would be a case involving direct contact with a Pfizer product in a pregnant women (eg, a nurse reports that she is pregnant and has been exposed to chemotherapeutic products).

A male has been exposed (eg, because of treatment or environmental exposure) to the investigational product prior to or around the time of conception and/or is exposed during his partner's pregnancy.

If a patient or patient's partner becomes or is found to be pregnant during the patient's treatment with the investigational product, the Investigator must report this information to Pfizer Safety on the CT Serious Adverse Event Form and an EDP Supplemental Form, regardless of whether an SAE has occurred. In addition, the Investigator must submit information regarding environmental exposure to a Pfizer product in a pregnant woman (eg, a patient reports that she is pregnant and has been exposed to a cytotoxic product by inhalation or spillage) to Pfizer Safety using the EDP Supplemental Form. This must be done irrespective of whether an AE has occurred and within 24 hours of awareness of the exposure. The information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The Investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow up to the initial EDP Supplemental Form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the Investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- · Spontaneous abortion includes miscarriage and missed abortion.
- Neonatal deaths that occur within 1 month of birth should be reported, without regard
  to causality, as SAEs. In addition, infant deaths after 1 month should be reported as
  serious adverse events when the Investigator assesses the infant death as related or
  possibly related to exposure to the investigational product.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the Investigator will provide the study patient with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the patient was given the Pregnant Partner Release of Information Form to provide to his partner.

#### 8.4.2.2. Exposure During Breastfeeding

Scenarios of exposure during breastfeeding must be reported, irrespective of the presence of an associated SAE, to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form. An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg. vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug's administration, the SAE is reported together with the exposure during breastfeeding.

### 8.4.2.3. Occupational Exposure

An occupational exposure occurs when, during the performance of job duties, a person (whether a healthcare professional or otherwise) gets in unplanned direct contact with the product, which may or may not lead to the occurrence of an AE.

An occupational exposure is reported to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form, regardless of whether there is an associated SAE. Since the information does not pertain to a patient enrolled in the study, the information is not reported on a CRF; however, a copy of the completed CT SAE Report Form is maintained in the investigator site file.

## 8.4.3. Medication Errors

Other exposures to the investigational product under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the CT<br>SAE Report Form to<br>Pfizer Safety Within<br>24 Hours of Awareness |
|---|---|---|
| Medication errors | All (regardless of whether<br>associated with an AE) | Only if associated with an SAE |

### 8.4.3.1. Medication Errors

Medication errors may result from the administration or consumption of the investigational product by the wrong patient, or at the wrong time, or at the wrong dosage strength.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### Medication errors include:

- Medication errors involving patient exposure to the investigational product;
- Potential medication errors or uses outside of what is foreseen in the protocol that do
  or do not involve the participating patient.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of medication dosing error, the sponsor should be notified immediately.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and non-serious, are recorded on an AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a CT SAE Report Form only when associated with an SAE.

### 9. DATA ANALYSIS/STATISTICAL METHODS

Detailed methodology for summary and statistical analyses of the data collected in this trial will be documented in a Statistical Analysis Plan (SAP), which will be maintained by Pfizer. This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoint and/or its analysis will also be reflected in a protocol amendment.

## 9.1. Analysis sets

The following patient sets will be assessed.

Safety analysis set.

The safety analysis set includes all enrolled patients who receive at least one dose of axitinib or crizotinib.

Per protocol analysis set (evaluable for DLT).

All enrolled patients who are eligible, receive at least one dose of axitinib and crizotinib, and who either experience DLT during the first cycle, or complete the 1st cycle observation period. Patients who are lost to follow-up before receiving at least 75% of the planned first-cycle dose due to reasons unrelated to treatment related adverse events are not evaluable for DLT.

· Response evaluable analysis set.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

All patients who start Cycle 1 with an adequate baseline tumor assessment and at least 1 follow up tumor assessment will be considered evaluable for anti-tumor efficacy using standard RECIST 1.1 criteria. Patients who are treated and removed from study prior to on-study tumor assessment because of disease progression will be considered evaluable for efficacy and counted as failures.

#### PK analysis set.

The PK concentration population is defined as all treated patients who have at least 1 concentration of any of the study drugs.

The PK parameter analysis population is defined as all treated patients who have at least 1 of the PK parameters of interest of any of the study drugs.

### Biomarker analysis set.

As described in the Rationale for Protocol Amendment #3, enrollment in Expansion Phase Cohort 2 was challenging and afforded small patient numbers (7 patients overall), which led to a decision to discontinue further enrollment. For these reasons, biomarker analyses will be performed only on Cohort 1.

The biomarker analysis set is defined as all treated patients who have at least one screening biomarker assessment, and have received at least one dose of any study drug. Analysis sets will be defined separately for blood-based and tumor tissue-based biomarkers.

If mutational profiling is performed on samples derived from the biomarker analysis set, the analysis may be limited to screening samples only.

### 9.2. Statistical Methods and Properties

### 9.2.1. Statistical Methods for Dose Escalation/De-Escalation: mTPI

Many alternative designs have been proposed to the standard 3+3 design for Phase 1 dose escalation trials that improve accuracy, efficiency and statistical validity.

The modified toxicity probability interval (mTPI) design <sup>38</sup> uses a Bayesian statistics framework and a beta/binomial hierarchical model to compute the posterior probability of three dosing intervals that reflect the relative difference between the toxicity rate of each dose level to the target rate (pT = 0.30). If the toxicity rate of the currently used dose level is far smaller than pT, the mTPI will recommend escalating the dose level; if it is close to pT, the mTPI will recommend continuing at the current dose; if it is far greater than pT, the mTPI will recommend de-escalating the dose level. These rules are conceptually similar to those used by the 3+3 design, except the decisions of an mTPI design are based on posterior probabilities calculated under a coherent probability model.

Being a model-based design, mTPI automatically and appropriately tailors dose-escalation and de-escalation decisions for different trials with different toxicity parameters. More importantly, all the dose-escalation decisions for a given trial can be pre-calculated under the mTPI design and presented in a two-way table (Appendix 5). Thus, compared to other

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

advanced model-based designs published in the literature, the mTPI design is logistically less complicated and easier to implement. Recently, a Phase I trial based on the mTPI design has been published.<sup>39</sup>

Decision rules are based on calculating unit probability mass (UPM) of three dosing intervals corresponding to under, proper, and over dosing in terms of toxicity. Specifically, the underdosing interval is defined as  $(0; pT-e_1)$ , the over-dosing interval  $(pT+e_2)$ , and the proper-dosing interval  $(pT-e_1, pT+e_2)$ , where  $e_1$  and  $e_2$  are small fractions. Based on the safety profile of axitinib and crizotinib,  $e_1$  is selected as 0.05, and  $e_2$  is selected as 0.00. Therefore, the target dosing interval for the DLT rate is (0.25, 0.30).

The three dosing intervals are associated with three different dose-escalation decisions. The under-dosing interval corresponds to a dose escalation (E), over-dosing corresponds to a dose de-escalation (D), and proper-dosing corresponds to remaining at the current dose (S). Given a dosing interval and a probability distribution, the unit probability mass (UPM) of that dosing interval is defined as the probability of a subject belonging to that dosing interval divided by the length of the dosing interval. The mTPI design calculates the UPMs for the three dosing intervals, and the one with the largest UPM informs the corresponding dose-finding decision, which is the dose level to be used for future patients. For example, if the under-dosing interval has the largest UPM, the decision will be to escalate, and the next cohort of patients will be treated at the next higher dose level. Ji and collaborators have demonstrated that the decision based on UPM is optimal in that it minimizes a posterior expected loss (ie, minimizes the chance of making a wrong dosing decision).

The dose-finding component of the trial is terminated when either approximately 25 DLT evaluable patients have been enrolled or when at least 10 evaluable patients have been treated at the highest dose with DLT rate <0.33, whichever comes first.

## 9.2.2. Statistical Method for Estimating the MTD

As described in Section 3.1.3, the estimated MTD will be the highest tested dose level with a DLT rate <0.33 in at least 10 DLT evaluable patients. We assume that higher doses of either axitinib or crizotinib result in higher toxicity rates. But, due to the relatively low number of patients that may be potentially allocated to any dose combination, this assumption may be violated.

For example, at the end of the study, the dose combination (crizotinib 250 mg BID) axitinib 3 mg BID) may have a higher proportion of observed toxicities than, say, (crizotinib 250 mg BID), axitinib 5 mg BID), and this variability may be simply related to small cohort size alone. To overcome this potential problem, we use a bivariate isotonic regression to smooth the resulting toxicity surface to a monotonically increasing one. The determination of the MTD contour is accomplished using the Dykstra-Roberston algorithm. Once a monotonically increasing toxicity surface is obtained (either observed or smoothed according to the bivariate isotonic regression algorithm), the MTD combinations closest to the targeted DLT rate of 0.3 but still <0.33 are calculated. Clinical judgment will be exercised in taking forward combinations to the Expansion Phase cohort(s), in case no clear choice exists between more than 1 competing MTD combination. While the limited sample size may result in up to 2 dose combinations of equal potential anti-tumor activity, under the circumstances of this trial, likely only one will be chosen for the expansion cohort. This

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

decision will be based upon the combination of data related to safety, anti-tumor activity, and clinical judgment of the Investigators and the Sponsor.

#### 9.3. Sample Size Determination

The sample sizes planned for the study arise from logistic feasibility and past experience with Phase 1b studies in oncology and are not entirely driven by statistical considerations. It is expected that approximately 65 patients will be required to achieve all study objectives.

Due to the dynamic nature of the Bayesian allocation procedure, the sample size of the Up-and-Down matrix design using the mTPI approach cannot be determined in advance. It is estimated 25 DLT evaluable patients will be enrolled in the dose escalation stage in order to have a reliable and accurate estimate of the MTD. In addition, there will be Dose Expansion Phase cohorts to characterize safety, biomarkers, and efficacy in terms of probability (p) of achieving an event of interest including, but not limited to, objective response (OR). The goal will be to estimate proportions of such patients with the standard error (SE) of not greater than 0.12, ie, by definition,

$$SE = \sqrt{\frac{p(1-p)}{n}} \le \frac{1}{2\sqrt{n}}$$

Therefore, a sample of twenty patients (n-20) per Dose Expansion Phase cohort will allow estimation of the probability of achieving an event of interest with the standard error <0.12.

## 9.4. Efficacy Analysis

In this study anti-tumor activity is a secondary objective. Efficacy analyses will be presented in the form of statistical summaries and data listing for the Dose Expansion Phase cohorts. For the Dose Escalation cohorts only data listings will be presented.

## 9.4.1. Analysis of Efficacy Endpoints (Dose Expansion Phase Cohorts)

Objective response rate (ORR) is defined as the proportion of patients with a confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1 definitions, relative to the response evaluable population as well as the safety population. Confirmed responses are those that persist on repeat tumor assessments for at least 4 weeks after initial documentation or response. Otherwise, the patient will be counted as a non-responder in the assessment of ORR.

Duration of Response (DR) is defined as the time from the first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.

Progression Free Survival (PFS) is defined as the time from the first dose to the first progression of disease (PD) or death for any reason in the absence of documented PD. PFS will be summarized in the safety analysis set. PFS data will be censored on the date of the last tumor assessment on study for patients who do not have objective tumor progression and

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

who do not die while on study. Patients lacking an evaluation of tumor response after enrollment will have their PFS time censored on the date of first dose with a duration of 1 day. Patients who are treated and removed from study prior to on-study tumor assessment because of disease progression will be considered evaluable for efficacy and counted as an event at the time of progression. Additionally, patients who start a new anti-cancer therapy prior to documented PD will be censored at the date of the last tumor assessment prior to the start of the new therapy.

Summaries will include: ORR, DR and 6-month PFS probabilities. Time-to event endpoints (PFS and DR) will be analysed with Kaplan-Meier method. Point estimates will be presented with their 95% confidence intervals. In addition, progression date, death date, date of first response and last tumor assessment date will be listed, together with best overall response (BOR), DR and PFS.

### 9.5. Analysis of Other Endpoints

#### 9.5.1. Analysis of Pharmacokinetics

### 9.5.1.1. Pharmacokinetic Analysis of Crizotinib and Axitinib

All patients who complete at least one day of PK blood sampling will be included in the PK analyses. Standard plasma PK parameters for axitinib and crizotinib (and metabolite) will be estimated using non-compartmental analysis. For crizotinib, standard PK parameters will include the maximum plasma concentration ( $C_{max}$ ), minimum plasma concentration ( $T_{max}$ ), time to maximum plasma concentration ( $T_{max}$ ), area under the plasma concentration versus time curve to the time of the last measurable concentration ( $AUC_{0-last}$ ), area under the plasma concentration versus time curve to 12 hours ( $AUC_{0-l2}$ ), and oral plasma clearance (CL/F). For axitinib, standard PK parameters will include  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-last}$ ,  $AUC_{0-l2}$ , CL/F, apparent volume of distribution ( $V_2/F$ ) and plasma elimination half life ( $t^1/2$ ). Descriptive statistics for the PK parameters for each drug will be provided by day of assessment in tabular form.

All plasma concentrations will be summarized descriptively (n, mean, SD, CV, median, minimum, maximum, geometric mean, its associated CV, and 95% confidence interval) by dose, cycle, day and nominal time. Individual patient and median profiles of the concentration-time data will be plotted by dose, cycle and day (single dose and steady-state) using nominal times. Median profiles will be presented on both linear-linear and log-linear scales.

Trough concentrations for crizotinib will be plotted for each dose using a box-whisker plot by cycle and day within cycle in order to assess the attainment of steady-state.

In addition, Non-linear Mixed Effects Modeling (NONMEM) approaches will be explored to further describe the pharmacokinetic profile and assess potential drug interaction.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 9.5.1.2. Effect of Crizotinib on Axitinib Pharmacokinetics

The effect of repeated crizotinib dosing on axitinib PK will be evaluated using AUC<sub>0-12</sub> of axitinib on Lead-in Day 7 and Cycle 1 Day 15, respectively, as the primary pharmacokinetic parameter. Ninety-percent confidence interval for the ratio of geometric means of AUC<sub>0-12</sub> (axitinib in presence of crizotinib/axitinib alone) will be computed to assess the magnitude of the effect.

### 9.5.1.3. Population Pharmacokinetic Analysis or PK/PD Modeling

Mechanism-based or semi-mechanistic sequential pharmacokinetic-pharmacodynamic models may be developed using NONMEM® to explore any relationships between plasma drug concentrations and selected safety, biomarker, and efficacy endpoints.

The results of these analyses, if performed, will be reported separately.

## 9.5.1.4. Statistical Analysis of Biomarker Endpoints

Biomarkers will be assessed separately for blood and tumor tissue samples. In each case, summaries of baseline levels and changes from baseline will be reported. Summary statistics may include the mean and standard deviation, median, and minimum/maximum levels of biomarker measures or frequency statistics, as appropriate.

Data from biomarker assays will be analyzed using graphical methods and descriptive statistics such as linear regression, t-test, and analysis of variance (ANOVA). The statistical approach may examine correlations of biomarker results with pharmacokinetic parameters and measures of anti-tumor efficacy.

Due to the exploratory nature of the proposed biomarkers, the data analysis will be conducted with the goal of identifying biomarkers with the strongest concordance to clinical outcome, encompassing both safety and efficacy. Candidate biomarkers will be validated in subsequent trials.

### 9.6. Safety Analysis

Summaries and analyses of the primary safety endpoint will be based on the per protocol analysis set. All other summaries and analyses of safety parameters will include all patients in the Safety Analysis Set. Safety data will be summarized by each cohort for all treated patients using appropriate tabulations and descriptive statistics. Safety data collected during the lead-in PK period will be reported separately. The analysis of safety will extend through 28 days after the last administration of study drug.

### 9.6.1. Analysis of Primary Safety Endpoint

Dose Limiting Toxicity (DLTs) is the primary endpoint of the Dose Escalation Phase of the study. The occurrence of DLTs observed in the Dose Escalation Cohorts is used to estimate the MTD (if reached) as described in Section 3.1.3. Adverse Events constituting DLTs will be listed per cohort.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 9.6.2. Analysis of Secondary Safety Endpoints

### 9.6.2.1. Adverse Events

Adverse Events (AEs) will be graded by the Investigator according to the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA). The focus of AE summaries will be on Treatment Emergent Adverse Events, those with initial onset or increasing in severity after the first dose of study medication. The number and percentage of patients who experienced any AE, serious AE (SAE), treatment related AE, and treatment related SAE will be summarized according to worst toxicity grades. The summaries will present AEs both on the entire study period and by cycle (Cycle 1 and Cycles beyond 1).

### 9.6.2.2. Laboratory Tests Abnormalities

The number and percentage of patients who experienced laboratory test abnormalities will be summarized according to worst toxicity grade observed for each lab assay. The analyses will summarize laboratory tests both on the entire study period and by cycle (Cycle 1 and Cycles beyond 1). Shift tables will be provided to examine the distribution of laboratory toxicities.

For laboratory tests without NCI CTCAE grade definitions, results will be categorized as normal, abnormal or not done.

### 9.6.2.3. ECG

All ECGs obtained during the study will be evaluated for safety. The triplicate ECG data will be averaged. All summary statistics and data presentations will use the triplicate averaged data. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Any data obtained from hand-reading of abnormal ECGs by a cardiologist (reported as unplanned ECGs in CRF) will be averaged separately and reported in summary tables, although both cardiologist manual overreads and machine-calculated values for the same time points will be provided in data listings. QT measurements corrected by heart rate (QTc) using Bazett's (QTcB) and Fridericia's (QTcF) methods will be used for the data analysis and interpretation.

### 9.6.3. Concomitant Medications/Follow-up Systemic Therapy

All medications received during the treatment period will be considered as concomitant medications and will be coded by WHO medical dictionary. Patients who received concomitant medications will be listed. Follow-up systemic therapy for the primary diagnosis will be summarized by categories of follow-up therapy and will be listed for each patient as appropriate.

### 9.6.4. Ophthalmologic Data

Best corrected visual acuity (Snellen fraction), biomicroscopic, and ophthalmoscopic findings will be recorded at baseline and any change from baseline will be summarized/listed for all patients who receive a dose of study treatment, with a baseline assessment and at least one post-baseline assessment.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

For those patients who are selected for additional testing based on clinical judgment, the refractive error (sphere, cylinder, axis), pupillary size (millimeters), optical coherence tomographic central retinal subfield thickness (microns), and intraocular pressure (mm Hg) at screening and their changes from screening will be quantitatively summarized/listed. The qualitative findings of fundus photography and optical coherence tomography at screening and their changes from screening will also be summarized/listed.

For the baseline screening results, percentages of patients falling into each category of the examination status (normal, mild, moderate, or severe) will be summarized/listed for each structure by eye. For post-baseline results, percentages of patients falling into each category of the examination status (new findings/worsening of finding, no change, improvement of finding, etc.) will be summarized/listed for each eye structure.

Additional summaries of ophthalmologic data will be considered as appropriate and described in the SAP.

#### 9.7. Data Monitoring Committee

An external Data Safety Monitoring Committee will not be established for the study. For the purpose of this protocol, Pfizer procedures for periodic safety review will be applied by an internal safety review team with medical and statistical capabilities to review individual and summary data collected in the safety and clinical databases. Procedures include:

- Surveillance for SAEs according to regulatory guidelines.
- Discussions between the Investigators and the Sponsor of AEs, laboratory tests
  abnormalities, vital signs and ECGs findings observed at each dose level in an
  ongoing manner at regular teleconferences and/or meetings to determine the safety
  profile and make risk/benefit assessment and decide if further enrollment is
  appropriate. During the Dose Escalation Phase, in particular, monitoring and safety
  findings satisfying the DLT criteria will be discussed in an on-going manner.
- Findings having immediate implication for the management of patients on study will be communicated to all Principal Investigators in the timeframe associated with unexpected and drug-related SAEs.

### 10. QUALITY CONTROL AND QUALITY ASSURANCE

Pfizer or its agent will conduct periodic monitoring visits during study conduct to ensure that the protocol and Good Clinical Practices (GCPs) are being followed. The monitors may review source documents to confirm that the data recorded on CRFs is accurate. The Investigator and institution will allow Pfizer monitors/auditors or its agents and appropriate regulatory authorities direct access to source documents to perform this verification. This verification may also occur after study completion.

During study conduct and/or after study completion, the investigator site may be subject to review by the Institutional Review Board (IRB)/Ethics Committee (EC), and/or to quality assurance audits performed by Pfizer, or companies working with or on behalf of Pfizer, and/or to inspection by appropriate regulatory authorities.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

The investigator(s) will notify Pfizer or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with Pfizer or its agents to prepare the investigator site for the inspection and will allow Pfizer or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the patient's medical records. The investigator will promptly provide copies of the inspection findings to Pfizer or its agent. Before response submission to the regulatory authorities, the investigator will provide Pfizer or its agents with an opportunity to review and comment on responses to any such findings.

It is important that the Investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

#### 11. DATA HANDLING AND RECORD KEEPING

### 11.1. Case Report Forms/Electronic Data Record

As used in this protocol, the term CRF should be understood to refer to either a paper form or an electronic data record or both, depending on the data collection method used in this study.

A CRF is required and should be completed for each included patient. The completed original CRFs are the sole property of Pfizer and should not be made available in any form to third parties, except for authorized representatives of Pfizer or appropriate regulatory authorities, without written permission from Pfizer.

The Investigator has ultimate responsibility for the collection and reporting of all clinical, safety and laboratory data entered on the CRFs and any other data collection forms (source documents) and ensuring that they are accurate, authentic / original, attributable, complete, consistent, legible, timely (contemporaneous), enduring and available when required. The CRFs must be signed by the Investigator or by an authorized staff member to attest that the data contained on the CRFs is true. Any corrections to entries made in the CRFs, source documents must be dated, initialed and explained (if necessary) and should not obscure the original entry.

In most cases, the source documents are the hospital's or the physician's patient chart. In these cases data collected on the CRFs must match the data in those charts.

In some cases, the CRF, or part of the CRF, may also serve as source documents. In these cases, a document should be available at the Investigator's site as well as at Pfizer and clearly identify those data that will be recorded in the CRF, and for which the CRF will stand as the source document.

### 11.2. Record Retention

To enable evaluations and/or inspections/audits from regulatory authorities or Pfizer, the Investigator agrees to keep records, including the identity of all participating patients (sufficient information to link records, eg. CRFs and hospital records), all original signed informed consent documents, copies of all CRFs, safety reporting forms, source documents,

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

and detailed records of treatment disposition, and adequate documentation of relevant correspondence (eg. letters, meeting minutes, telephone calls reports). The records should be retained by the Investigator according to International Conference on Harmonisation (ICH), guidelines, according to local regulations, or as specified in the Clinical Study Agreement (CSA), whichever is longer.

If the Investigator becomes unable for any reason to continue to retain study records for the required period (eg, retirement, relocation), Pfizer should be prospectively notified. The study records must be transferred to a designee acceptable to Pfizer, such as another Investigator, another institution, or to an independent third party arranged by Pfizer. Investigator records must be kept for a minimum of 15 years after completion or discontinuation of the study or for longer if required by applicable local regulations.

The Investigator must obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

### 12. ETHICS

#### 12.1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

It is the responsibility of the Investigator to have prospective approval of the study protocol, protocol amendments, informed consent documents, and other relevant documents, eg, recruitment advertisements, if applicable, from the IRB/IEC. All correspondence with the IRB/IEC should be retained in the Investigator File. Copies of IRB/IEC approvals should be forwarded to Pfizer.

The only circumstance in which an amendment may be initiated prior to IRB/IEC approval is where the change is necessary to eliminate apparent immediate hazards to the patients. In that event, the Investigator must notify the IRB/IEC and Pfizer in writing immediately after the implementation.

#### 12.2. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects (Council for International Organizations of Medical Sciences 2002), Guidelines for GCP (ICH 1996), and the Declaration of Helsinki (World Medical Association 1996 & 2008).

In addition, the study will be conducted in accordance with the protocol, the ICH guideline on GCP, and applicable local regulatory requirements and laws.

#### 12.3. Patient Information and Consent

All parties will ensure protection of patient personal data and will not include patient names other identifiable data in any reports, publications, or other disclosures, except where required by laws.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

When study data are compiled for transfer to Pfizer and other authorized parties, patient names, addresses, and other identifiable data will be replaced by numerical codes based on a numbering system provided by Pfizer in order to de-identify study patients. The investigator site will maintain a confidential list of patients who participated in the study, linking each patient's numerical code to his or her actual identity. In case of data transfer, Pfizer will maintain high standards of confidentiality and protection of patients' personal data consistent with applicable privacy laws.

The informed consent documents and any patient recruitment materials must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws.

The informed consent document(s) used during the informed consent process and any patient recruitment materials must be reviewed and approved by Pfizer, approved by the IRB/EC before use, and available for inspection.

The Investigator must ensure that each study patient is fully informed about the nature and objectives of the study and possible risks associated with participation.

The Investigator, or a person designated by the Investigator, will obtain written informed consent from each patient before any study-specific activity is performed. The Investigator will retain the original of each patient's signed consent document.

### 12.4. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the Investigator is aware of any new information that might influence the evaluation of the benefits and risks of the investigational product, Pfizer should be informed immediately.

In addition, the Investigator will inform Pfizer immediately of any urgent safety measures taken by the Investigator to protect the study patients against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the Investigator becomes aware of.

### 13. DEFINITION OF END OF TRIAL

#### 13.1. End of Trial in a Member State

End of Trial in a Member State of the European Union is defined as the time at which it is deemed that sufficient patients have been recruited and completed the study as stated in the regulatory application (ie, Clinical Trial Application (CTA)) and ethics application in the Member State. Poor recruitment (recruiting less than the anticipated number in the CTA) by a Member State is not a reason for premature termination but is considered a normal conclusion to the study in that Member State.

## 13.2. End of Trial in all other Participating Countries

End of Trial in all other participating countries is defined as Last Subject Last Visit.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### 14. SPONSOR DISCONTINUATION CRITERIA

Premature termination of this study may occur because of a regulatory authority decision, change in opinion of the IRB/IEC, or investigational product safety problems, or at the discretion of Pfizer. In addition, Pfizer retains the right to discontinue development of axitinib or crizotinib at any time.

If a study is prematurely terminated or discontinued, Pfizer will promptly notify the Investigator. After notification, the Investigator must contact all participating patients and the hospital pharmacy (if applicable) within 1 month. As directed by Pfizer, all study materials must be collected and all CRFs completed to the greatest extent possible.

### 15. PUBLICATION OF STUDY RESULTS

### 15.1. Communication of Results by Pfizer

Pfizer fulfills its commitment to publicly disclose clinical trial results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the European Clinical Trials Database (EudraCT), and or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

### www.elinicaltrials.gov

Pfizer posts clinical trial US Basic Results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a Pfizer product, regardless of the geographical location in which the study is conducted. US Basic Results are submitted for posting within 1 year of the primary completion date for studies in adult populations or within 6 months of the primary completion date for studies in pediatric populations.

Primary Completion Date is defined as the date that the final patient was examined or received an intervention for the purposes of final collection of data for the primary outcome, whether the clinical trial concluded according to the pre-specified protocol or was terminated.

## **EudraCT**

Pfizer posts European (EU) Basic Results on EudraCT for all Pfizer-sponsored interventional studies that are in scope of EU requirements. EU Basic Results are submitted for posting within 1 year of the primary completion date for studies in adult populations or within 6 months of the primary completion date for studies in pediatric populations.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### www.pfizer.com

Pfizer posts Public Disclosure Synopses (clinical study report synopses in which any data that could be used to identify individual patients has been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the US Basic Results document is posted to www.clinicaltrials.gov.

#### 15.2. Publications by Investigators

Pfizer supports the exercise of academic freedom and has no objection to publication by principal investigator of the results of the study based on information collected or generated by principal investigator, whether or not the results are favorable to the Pfizer product. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Investigator will provide Pfizer an opportunity to review any proposed publication or other type of disclosure of the results of the study (collectively, "Publication") before it is submitted or otherwise disclosed.

Investigator will provide any publication to Pfizer at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

Investigator will, on request, remove any previously undisclosed Confidential Information before disclosure, except for any study- or Pfizer product-related information necessary to the appropriate scientific presentation or understanding of the study results.

If the Study is part of a multi-centre study, Investigator agrees that the first publication is to be a joint publication covering all study sites, and that any subsequent publications by the principal investigator will reference that primary publication. However, if a joint manuscript has not been submitted for publication within 12 months of completion or termination of the Study at all participating sites, Investigator is free to publish separately, patient to the other requirements of this Section.

For all publications relating to the Study, Institution will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

Publication of study results is also provided for in the Clinical Study Agreement between Pfizer and the institution. In this section entitled Publications by Investigators, the defined terms shall have the meanings given to them in the Clinical Study Agreement.

If there is any conflict between the CSA and any Attachments to it, the terms of the CSA control. If there is any conflict between this protocol and the CSA, this protocol will control as to any issue regarding treatment of study patients, and the CSA will control as to all other issues.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

#### 16. REFERENCES

- Ferrar N. Kerbel R. S. 2005 Angogenesis as a therapeutic target. Nature 438:967.
- Ellis L.M. Hicklin D.J. 2008 VEGF-targeted therapy: Mechanisms of anti-tumor activity. Nat. Rev. Cancer 8:579.
- American Cancer Society, Cancer Facts & Figures 2013, Atlanta: American Cancer Society; 2013.
- Choueiri T.K., Vaishampayan U., Rosenberg J.E., et al 2013 Phase II and Biomarker Study of the Dual MET/VEGFR2 Inhibitor Foretinib in Patients with Papillary Renal Cell Carcinoma J. Clin. Oncol. 31:181-186.
- Finley D.S., Pantuck A.J., Belldegrun A.S. 2011 Tumor Biology and Prognostic Factors in Renal Cell Carcinoma. The Oncologist, 16:4.
- NCCN Clinical Practice Guidelines in Oncology: Kidney Cancer. Version 2,2017.
- Gross-Goupil M., Massard C., Rayaud A. 2012 Targeted Therapies in Metastatic Renal Cell Carcinoma: Overview of the Past Year Curr. Urol. Rep. 13:16-23.
- Mihaly Z., Sztupinszki Z., Surowiak P., and Gyorffy B. 2012 A Comprehensive Overview of Targeted Therapy in Metastatic Renal Cell Carcinoma Current Cancer Drug Targets 12:857-872.
- Escudier B., Albiges L., and Sonpavde G. 2013 Optimal Management of Metastatic Renal Cell Carcinoma: Current Status Drugs 73:427-38.
- Grepin R., and Pages G. 2010 Molecular Mechanisms of Resistance to Tumour Anti-Angiogenic Strategies., *Journal of Oncology* 2010:1.
- Bergers, G. & Hanahan, D. 2008 Modes of resistance to anti-angiogenic therapy. Nature. Rev. Cancer 8:592.
- Paez-Ribes M., Allen E., Hudock J., et al. 2009, Antiangiogenic Therapy Elicits Malignant Progression of Tumors to Increased Local Invasion and Distant Metastasis. Cancer Cell 15:220.
- Ebos J.M.L., Lee C.R., Kerbel R.S. et al., 2009 Tumor and Host-Mediated Pathways of Resistance and Disease Progression to Antiangiogenic Therapy. Clin Cancer Res; 5020:15(16).
- Ebos J.M.L., Lee C.R., Cruz-Munoz W., et al., 2009 Accelerated Metastasis after Short-Term Treatment with a Potent Inhibitor of Tumor Angiogenesis. Cancer Cell 15.
- Martin T.A., Jiang W.G., 2010 Hepatocyte Growth Factor and Its receptor Singalling Complex as Targets in Cancer Therapy. Anti-cancer agents in medicinal chemistry 10:2.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Trusolino L., Bertotti A., Comoglio P., 2010 MET signalling: principles and functions in development, organ regeneration and cancer. *Nature*, 11:834.
- Jahangiri A., De Lay M., Miller L.M. et al 2013 Gene Expression Profile Identifies
  Tyrosine Kinase c-Met as a Targetable Mediator of Antiangiogenic Therapy Resistance
  Clin. Cancer Res. 19:1773-83.
- Semino B, and McDonald D.M. 2012 Controlling escape from angiogenesis inhibitors Nature Reviews/ CANCER 12:699-709.
- Shojaei F., Lee J.H., Simmons B.H., et al., 2010 HGF/c-Met Acts as an Alternative Angiogenic Pathway in Sunitinib-Resistant Tumors. Cancer Res, 70:10090.
- Shojaci F., Simmons B.H., Lee J.H., et al 2012 HGF/c-Met pathway is one of the mediators of sunitinib-induced tumor cell type-dependent metastasis Cancer Letters 320: 48-55.
- Sennino B., Ishiguro-Oonuma T., Wei Y. et al 2012 Suppression of Tumor Invasion and Metastasis by Concurrent Inhibition of c-Met and VEGF Signaling in Pancreatic Neuroendocrine Tumors Cancer Discovery 2:270-87.
- You W-K, Sennino B., Williamson C.W., et al 2011 VEGF and c-Met Blockade Amplify Angiogenesis Inhibition in Pancreatic Islet Cancer Canc. Res. 71:4758-68.
- Ciamporcero E.S., Kiersten M.M., Adelaiye R. et al 2013 Combination of axitinib and crizotinib in renal cell carcinoma models AACR Annual meeting Abstract Number 1618.
- Vaishampayan U. 2013 Cabozantinib as a Novel Therapy for Renal Cell Carcinoma Curr Onco. Rep. 15:76-82.
- Smith D.C., Smith MR., Sweeney C. et al 2013 Cabozantinib in Patients with Advanced Prostate Cancer: Results of Phase II Randomized Discontinuation Trial J. Clin. Oncol. 31:412-419.
- Choueiri T.K., Pal S.K., McDermott D.F. et al 2012 Efficacy of cabozantinib (XL184) in patients (pts) with metastatic, refractory renal cell carcinoma (RCC) J.Clin. Oncol. vol. 30, No 15 suppl (May 20 Supplement) 2012: 4504.
- Ou S-H.I., Huang Bartlett, C. Mino-Kenudson M., et al 2012 Crizotinib for the Treatment of ALK-Rearranged Non-Small Cell Lung Cancer: A Success Story to Usher in the Second Decade of Molecular Targeted Therapy in Oncology *The Oncologist* 17:1351-1375.
- Robinson K.W., and Sandler A.B. The Role of MET Receptor Tyrosine Kinase in Non-Small Cell Lung Cancer and Clinical Development of Targeted anti-MET agents 2013 The Oncologist 18:115-122.
- 29. Investigator's Brochure of Crizotinib (PF-02341066), dated December 2016.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- Schoffski P., Garcia J.A., Stadler W.M., et al., 2010 A phase II study of the efficacy and safety of AMG 102 in patients with metastatic renal cell carcinoma. BJU International 2010 1.
- Lennerz J.K., Kwak E.L., Ackerman A., et al. 2011 MET amplification identifies a small and aggressive subgroup of esophagogastric adenocarcinoma with evidence of responsiveness to crizotinib. J.Clin Oncol 29: 4803-10.
- Ou S-H.L. Kwak E.L. Stwak-Tapp C. et al. 2011 Activity of crizotinib (PF2341066), a
  dual mesenchymal-epithelial transition (MET) and anaplastic lymphoma kinase (ALK)
  inhibitor, in a non-small cell lung cancer patient with De Novo MET amplification. J.
  Thoracic Oncol. 6: 942-6.
- Chi A.S., Batchelor T.T., Kwak E.L., et al. 2012 Rapid radiographic and clinical improvement after treatment of a MET-amplified recurrent glioblastoma with a mesenchymal-epithelial transition inhibitor J. Clin Oncol 30:e30-e33.
- 34. United States Package Insert for Xalkori®, dated April 2017.
- 35. Investigator's Brochure of AG-013736, dated July 2016.
- 36. United States Package Insert for Inlyta®, dated August 2014.
- Larochelle P., Kollmannsberger C., Feldman R.D., et al. 2012 Hypertension management in patients with renal cell cancer treated with anti-angiogenic agents. Curr. Oncol 19:202-208.
- Ji Y et al. A modified toxicity probability interval method for dose-finding trials. Clinical Trials 2010; 7:653 663.
- Fanale M et al. Phase I study of bortezomib plus ICE (BICE) for the treatment of relapsed/refractory Hodgkin lymphoma. British Journal of Haematology, 154:284 286, 2011.
- Dykstra R, Robertson T. An algorithm for isotonic regression for two or more independent variables. Ann Stat. 1982;10:708-716.
- 2006. Update of Recommendations for the Use of White Blood Cell Growth Factors: An Evidence-Based Clinical Practice Guideline. J. Clin Oncol Jul 1:3187-3205.
- T.K. Choueiri, B. Escudier, T. Powles, et al. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. The New England Journal of Medicine 2015 (DOI: 10.1056/NEJMoa1510016).
- B.I. Rini, B. Escudier, P. Tomczak, et al. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomized phase 3 trial. The Lancet, 378:1931-1939, 2011.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

## Appendix 1. ECOG Performance Status

| Score | Definition |
|---|---|
| 0 | Fully active, able to carry on all pre-disease activities without restriction |
| £ | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work or office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair |
| 5 | Dead |

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### Appendix 2. RECIST 1.1

The determination of antitumor efficacy during this study will be based on objective tumor assessments made according to the RECIST system of unidimensional evaluation.

### Measurability of Tumor Lesions

At baseline, individual tumor lesions will be categorized by the Investigator as either measurable or non-measurable by the RECIST criteria as described below.

### Measurable:

<u>Tumor lesion</u>: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

- 10 mm by CT scan (CT scan slice thickness no greater than 5 mm);
- 10 mm caliper measurement by clinical exam (lesions which cannot be accurately
  measured with calipers should be recorded as non-measurable).

Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

Non-Measurable: All other lesions, including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 mm to <15 mm short axis) as well as truly non-measurable lesions. Lesions considered truly non-measurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

NOTE: If measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.

### **Recording Tumor Measurements**

All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total representative of all involved organs should be identified as **target lesions** and measured and recorded at baseline and at the stipulated intervals during treatment. Target lesions should be selected on the basis of their size (lesion with the longest diameters) and their suitability for accurate repetitive measurements (either by imaging techniques or clinically).

The longest diameter will be recorded for each target lesion. The sum of the longest diameter for all target lesions will be calculated and recorded as the baseline sum longest diameter to be used as reference to further characterize the objective tumor response of the measurable dimension of the disease during treatment. All measurements should be performed using a caliper or ruler and should be recorded in metric notation in centimeters.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

All other lesions (or sites of disease) should be identified as **non-target lesions** and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present" or "absent."

### **Techniques for Assessing Measurable Disease**

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at screening and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical (physical) examination when both methods have been used to assess the antitumor effect of a treatment.

### **Definitions of Tumor Response**

## **Target Lesions**

Complete response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

Partial response (PR) is defined as a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.

Progressive disease (PD) is defined as a  $\geq 20\%$  increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as a reference the smallest sum of the longest dimensions since the treatment started.

### Non-Target Lesions

Complete response (CR) is defined as the disappearance of all non-target lesions. All lymph nodes must be non-pathological in size (<10 mm short axis).

Non-CR/Non-PD is defined as a persistence of ≥1 non-target lesions.

Progressive disease (PD) is defined as unequivocal progression of existing non-target lesions, or the appearance of ≥1 new lesion.

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease and progressive disease.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### Confirmation of Tumor Response

To be assigned a status of PR or CR, changes in tumor measurements in patients with responding tumors must be confirmed by repeat studies that should be performed ≥4 weeks after the criteria for response are first met. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 8 weeks.

### Determination of Tumor Response by the RECIST Criteria

When both target and non-target lesions are present, individual assessments will be recorded separately. Determination of tumor response at each assessment is summarized in the following table.

### Response Evaluation Criteria in Solid Tumors

| Target Lesions1 | Non-Target Lesions <sup>2</sup> | New Lesions | Tumor Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR. | Not evaluated | No | PR |
| PR. | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| PD | Any response | Yes or No | PD |
| Any response | PD | Yes or No | PD |
| Any response | Any response | Yes | PD |

<sup>&</sup>lt;sup>1</sup> Measurable lesions only

### **Determination of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). For CR and PR, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 8 weeks.

NOTE: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment. It should also be noted that a tumor marker increase does not constitute adequate objective evidence of tumor progression. However, such a tumor marker increase should prompt a repeat radiographic evaluation to document whether or not objective tumor progression has occurred.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of complete response depends upon this determination, it is recommended that the residual lesion be investigated by fine needle aspirate or biopsy before confirming the complete response status.

<sup>&</sup>lt;sup>2</sup> May include measurable lesions not followed as target lesions or non-measurable lesions.

Measurable or non-measurable lesions.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

Appendix 3. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)

The NCI CTCAE (version 4.03, dated 14 June 2010) has been placed in the Study Reference Binder for this protocol. Alternatively, the NCI CTCAE may be reviewed online at the following NCI website:

http://ctep.cancer.gov/reporting/ctc.html

AG-013736, PF-02341066

A4061068

Final Protocol Amendment 3, 09 June 2017

## Appendix 4. Abbreviations and Definitions of Term

AE Adverse Event

AHFS American Hospital Formulary Service AIDS Acquired Immune Deficiency Syndrome

ALK Anaplastic Lymphoma Kinase
ALT Alanine aminotransferase
ANC Absolute Neutrophil Count
ATP Adenosine TriPhosphate

ASHP American Society of Hospital Pharmacists

AST Aspartate aminotransferase
AUC Area Under the Curve
BAL BronchoAlveolar Lavage
BCVA Best Corrected Visual Acuity

BHD Birt-Hogg-Dubé BID Twice/day

BNP B-type Natriuretic Peptide

BP Blood Pressure
BUN Blood Urea Nitrogen
CDS Core Data Sheet

CHF Congestive Heart Failure
CI Confidence Interval

CI. Clearance

Cmax Maximum plasma Concentration
Cmin Minimum plasma Concentration

CR Complete Response CRF Case Report Form

CRPC Castration-Resistant Prostate Cancer

CSA Clinical Study Agreement CT Computerized Tomography

CTCAE Common Terminology Criteria for Adverse Events (US-NCI)

CTM Clinical Trial Material

CYP1A2 Cytochrome P450 enzyme-1A2 CYP3A4/5 Cytochrome P450 enzyme-3A4/5

DLT Dose Limiting Toxicity
DR Duration of Response
EC Ethics Committee
ECG Electrocardiogram

ECOG Easter Cooperative Oncology Group

EDP Exposure During Pregnancy

EIU Exposure in Utero

EU Europe

FDA Food and Drug Administration

<sup>18</sup>F FDG PET/CT 2-[18F]-Iluoro-2-deoxy-d-glucose Positron emission tomography/

computed tomography

FFPE Formalin Fixed, Paraffin Embedded

AG-013736, PF-02341066

A4061068

Final Protocol Amendment 3, 09 June 2017

| FH | Fumarate Hydratase |
|---|---|
| FSH | Follicle-Stimulating Hormone |
| GCP | Good Clinical Practice |
| GGT | Gamma-Glutamyl Transferase |
| HDPE | High Density PolyEthylene |
| HGF | Hepatocyte Growth Factor |
| HIF | Hypoxia-Inducable transcription Factor |
| HIV | Human Immunodeficiency Virus |
| ICH | International Committee Harmonization |
| ID | Identification |
| IFN | Interferon alpha |
| IL-2 | Interleukin-2 |
| IHC | ImmunoHistoChemistry |
| IND | Investigational New Drug |
| INR | International Normalized Ratio |
| IOP | IntraOcular Pressure |
| IRB | Institutional Review Board |
| | and the state of t |
| IUD | Intra Uterine Device |
| LFT | Liver Function Test |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MET | Mesenchymal Epithelial Transition factor |
| MRI | Magnetic Resonance Imaging |
| MTD | Maximum Tolerated Dose |
| mTOR | Mammalian Target Of Rapamycin |
| mTPI | Modified Toxicity Probability Interval |
| NCI | National Cancer Institute |
| NONMEM | Non linear Mixed Effects Modeling |
| NSCLC | Non-Small Cell Lung Cancer |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PD | Pharmacodynamic |
| PD | Progressive Disease |
| PDGF | Platelet-Derived Growth Factor |
| PDGFR | Platelet-Derived Growth Factor Receptor |
| PD-1 | Programmed Death-1 |
| PFS | Progression Free Survival |
| PK | Pharmacokinetics |
| PO | Per Os (by mouth) |
| PR | Partial Response |
| PS | Performance Status |
| PT | Prothrombin Time |
| QD | Every Day |
| QTe | Corrected Q-T interval |
| RCC | Renal Cell Cancer |
| RECIST | Response Evaluation Criteria in Solid Tumor |
| RP2D | Recommended Phase 2 Dose |
| KI ZD | Recommended Phase 2 Dose |

AG-013736, PF-02341066 A4061068

Final Protocol Amendment 3, 09 June 2017

SAE Serious Adverse Event
SD Stable Disease
SD Standard Deviation
SOA Schedule of Activities
SRSD Single Reference Safety Document
1½ Plasma elimination half life
TK1 Tyrosine Kinase Inhibitor

Tmax Time to maximum plasma concentration

TSH Thyroid Stimulating Hormone ULN Upper Limit of Normal

US United States

USPI United States Package Insert VEGF Vascular Endothelial Growth Factor

VEGFR Vascular Endothelial Growth Factor Receptor

VHL Hippel Lindau tumor suppressor gene

WBC White Blood Cell

WHO World Health Organization

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

### Appendix 5. Detailed Dose Escalation/De-Escalation Scheme

#### Number of patients treated at current dose 1 2 3 4 5 6 7 8 9 10 11 12 13 14 15 16 17 18 OEE E E E E E E E E E E E E E E 1DSSSSSEEEEEEEEEEEE SSS S S S S E E E DU DU D D S S S S S S S S S S E DU DU DU D D S S S S S S S S S S 5 DU DU DU DU DU D S S S S S SS 6 DU DU DU DU DU DU D D S Number of toxicities 7 DU DU DU DU DU DU DU D 8 DU D 9 DU 10 DU 11 DU 12 DU 13 14 DU DU DU DU DU 15 DU DU DU DU 16 DU DU DU 17 DU DU 18 DU

E = Escalate to the next higher dose
S = Stay at the current dose
D = De-escalate to the next lower dose
U = The current dose is unacceptably toxic
MTD = 30%

## Escalation/De-escalation algorithms for total number of patients treated at the current dose level (current and previous cohorts)

- With 3 patients treated at current dose level:
  - 0 DLT → escalate;
  - 1 DLT → remain at the same dose;
  - $2 DLTs \rightarrow de\text{-escalate};$
  - 3 DLTs → de-escalate and consider current dose as intolerable.
- With 4 patients treated at current dose level:
  - 0 DLT → escalate;
  - 1 DLTs → remain at the same dose;

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- 2 DLTs → de-escalate;
- 3-4 DLTs → de-escalate and consider current dose as intolerable.
- With 5 patients treated at current dose level:
  - 0 DLT → escalate;
  - 1-2 DLTs → remain at the same dose;
  - 3 DLTs → de-escalate;
    - 4-5 DLTs → de-escalate and consider current dose as intolerable.
- With 6 patients treated at current dose level:
  - 0 DLT → escalate:
  - 1-2 DLTs → remain at the same dose;
    - 3 DLTs → de-escalate;
      - 4-6 DLTs → de-escalate and consider current dose as intolerable.
- With 7 patients treated at current dose level:
  - 0-1 DLT → escalate;
  - 2-3 DLTs → remain at the same dose;
  - 4 DLTs → de-escalate;
  - 5-7 DLTs → de-escalate and consider current dose as intolerable.
- With 8 patients treated at current dose level:
  - 0-1 DLT → escalate;
  - 2-3 DLTs → remain at the same dose;
  - 4 DLTs → de-escalate;
  - 5-8 DLTs → de-escalate and consider currentdose as intolerable.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- With 9 patients treated at current dose level:
  - 0-1 DLT → escalate;
  - 2-4 DLTs → remain at the same dose;
    - 5-9 DLTs → de-escalate and consider currentdose as intolerable.
- · With 10 patients treated at current dose level:
  - 0-1 DLT → escalate;
    - 2-4 DLTs → remain at the same dose;
    - 5 DLTs → de-escalate;
    - 6-10 DLTs → de-escalate and consider currentdose as intolerable.
- · With 11 patients treated at current dose level:
  - 0-1 DLT → escalate;
  - 2-5 DLTs → remain at the same dose;
    - 6-11 DLTs → de-escalate and consider currentdose as intolerable.
- With 12 patients treated at current dose level:
  - 0-2 DLTs → escalate;
  - 3-5 DLTs → remain at the same dose;
  - 6 DLTs → de-escalate;
  - 7-12 DLTs → de-escalate and consider current dose as intolerable.
- With 13 patients treated at current dose level:
  - 0-2 DLTs → escalate;
  - 3-5 DLTs → remain at the same dose;
  - 6 DLTs → de-escalate;
  - 7-13 DLTs → de-escalate and consider current dose as intolerable.

AG-013736, PF-02341066 A4061068 Final Protocol Amendment 3, 09 June 2017

- With 14 patients treated at current dose level:
  - 0-2 DLTs → escalate;
  - 3-6 DLTs → remain at the same dose;
    - 7 DLTs → de-escalate;
    - 8-14 DLTs → de-escalate and consider current dose as intolerable.
- With 15 patients treated at current dose level:
  - 0-2 DLTs → escalate;
  - 3-6 DLTs → remain at the same dose;
    - 7 DLTs → de-escalate;
    - 8-15 DLTs → de-escalate and consider current dose as intolerable.
- With 16 patients treated at current dose level:
  - 0-2 DLTs → escalate;
  - 3-7 DLTs → remain at the same dose;
  - 8-16 DLTs → de-escalate and consider current dose as intolerable.
- With 17 patients treated at current dose level:
  - 0-2 DLTs → escalate;
    - 3-7 DLTs → remain at the same dose;
    - 8 DLTs → de-escalate;
    - 9-17 DLTs → de-escalate and consider current dose as intolerable.
- With 18 patients treated at current dose level:
  - 0-3 DLTs → escalate;
  - 4-7 DLTs → remain at the same dose;
  - 8 DLTs → de-escalate;
  - 9-18 DLTs → de-escalate and consider current dose as intolerable.

## **Document Approval Record**

**Document Name:** A4061008 Protocol Amendment 7, 08 November 2018

**Document Title:** A4061008 Protocol Amendment 7, 08 November 2018

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 26-Nov-2018 20:58:12 | Final Approval |
| | 27-Nov-2018 16:21:50 | Final Approval |